**Version Date:** 4/29/2025

**Abbreviated Title:** Pomalidomide for cGvHD

NIH Protocol #: 12C0197 NCT #: NCT01688466 Version Date: 4/29/2025

Title: A Randomized Phase 2 Single-Center Study of Pomalidomide for Chronic GVHD

NCI Principal Investigator: Najla El Jurdi, MD

Immune Deficiency Cellular Therapy Program (IDCTP)

Center for Cancer Research (CCR) National Cancer Institute (NCI) National Institutes of Health (NIH) 10 Center Drive, RM 8D44C

9000 Rockville Pike Bethesda, MD 20892 Phone: 240-858-3287

Email: najla.eljurdi@nih.gov

| Drug Name: | ame: Pomalidomide |
|---|---|
| IND Number: | 115336 |
| Sponsor: Center for Cancer Research | |
| Manufacturer: Celgene | |
| | Protocol tracking number: PO-GvHD-NCI-0046 |


## **PRÉCIS**

## **Background:**

- Chronic graft-versus-host disease (cGvHD) is the leading cause of non-relapse morbidity and mortality in persons after allogeneic hematopoietic cell transplants.
- About 50% of persons with cGvHD have disease refractory to systemic corticosteroids and there is no standard second-line therapy.
- Thalidomide, a drug with immune-modulating effects, was active in advanced cGvHD but was difficult to use at appropriate doses.
- Pomalidomide is related to thalidomide but with higher potency and more favorable toxicity profile. It is active in multiple myeloma and myeloproliferative neoplasm—associated myelofibrosis. Preliminary data in humans with cGvHD are encouraging but data are limited.

## **Objective:**

• Primary: Determine whether pomalidomide is effective in persons with moderate or severe cGvHD not controlled by corticosteroids.

## **Eligibility:**

- Inclusion Criteria
  - o Moderate or severe cGvHD per NIH criteria
  - o Age 18 to 75 years old
  - o Karnofsky performance score ≥60%
  - o Has cGvHD that did not respond to high-dose corticosteroids (average 0.5 mg/kg/d prednisone for ≥8 weeks) or second-line therapy
  - o Receiving stable or tapering doses of systemic therapy in the preceding 4 weeks
  - o Agree to adhere to methods of contraception and other fertility control measures as prescribed by the protocol
- Exclusion Criteria
  - o Acute GvHD (classic and late per NIH criteria)
  - O Absolute neutrophils <1.0x10<sup>9</sup>/L, platelets <75x10<sup>9</sup>/L, estimated creatinine clearance <50 mL/min/1.73m<sup>2</sup>
  - o NIH lung score 3
  - o Pregnant or lactating
  - Uncontrolled infection

## Design:

Randomized phase 2 trial with the single stage selection design. Patients will receive either a constant low dose of pomalidomide (0.5 mg/day) for six months or a strategy of increasing dose of pomalidomide from 0.5 mg/d up through each individual patients' maximum tolerated dose, with escalations by 0.5 mg/d every 2 weeks to a maximum of 2.0 mg/d. As an early stopping rule for futility, if after 7 patients have enrolled on either arm, 0 have responded, then no further patients will be accrued to that arm as soon as this can be determined. To protect patient safety, an early stopping rule will be implemented. With two arms, each of which has a maximal accrual of 16 patients, up to 32 evaluable patients will be randomized. Response assessments will occur


every 3 months with primary efficacy endpoint evaluated at 6 months. Patients with responding disease will continue therapy for another 6 months.

## TABLE OF CONTENTS

| P. | RÉCIS | S | 2 |
|---|---|---|---|
| T. | ABLE | OF CONTENTS | 4 |
| S | TATE: | MENT OF COMPLIANCE | 7 |
| 1 | IN | TRODUCTION | 7 |
| | 1.1 | Study Objectives | 7 |
| | 1.2 | Background and Rationale | 7 |
| | 1.3 | Pomalidomide | 12 |
| | 1.3.3. | 1 Pharmacokinetics and Product Metabolism in Humans | 14 |
| | 1.4 | Study Design and Rationale | 21 |
| 2 | EL | IGIBILITY ASSESSMENT AND ENROLLMENT | 22 |
| | 2.1 | Eligibility Criteria | 22 |
| | 2.2 | Required Testing and Counseling for FCBP and Partners of FCBP | 24 |
| | 2.3 | Screening Evaluation | 24 |
| | 2.4 | Registration Procedures | 25 |
| | 2.5 | Treatment Assignment and Randomization procedures | 25 |
| | 2.6 | Baseline Evaluation | 26 |
| 3 | ST | UDY IMPLEMENTATION | 26 |
| | 3.1 | Study Design | 26 |
| | 3.2 | Drug Administration | 28 |
| | 3.3 | Dose Modifications | 29 |
| | 3.4 | Questionnaires | 31 |
| | 3.5 | Study Calendar | 32 |
| | 3.6 | Criteria for Removal from Protocol Therapy and Off Study Criteria | 37 |
| 4 | CO | NCOMITANT MEDICATIONS/MEASURES | 37 |
| | 4.1 | Concomitant Corticosteroid Therapy and Tapering Guideline | 37 |
| | 4.2 | Other Treatments for cGvHD | 38 |
| | 4.3 | Venous Thromboembolism Prophylaxis | 38 |
| | 4.4 | Other Allowed Concomitant Therapy | 38 |
| | 4.5 | Prohibited Concomitant Therapy | 39 |
| 5 | BIG | OSPECIMEN COLLECTION | 39 |
| | 5.1 | Correlative Studies for Research | 39 |

| | 5.2 | Sample Storage, Tracking and Disposition | 40 |
|---|---|---|---|
| 6 | Г | DATA COLLECTION AND EVALUATION | 41 |
| | 6.1 | Data Collection | 41 |
| | 6.2 | Response Criteria | 43 |
| | 6.3 | Toxicity Criteria | 46 |
| 7 | N | NIH REPORTING REQUIREMENTS/DATA AND SAFETY MONITORING PLAN | 46 |
| | 7.1 | Definitions | 46 |
| | 7.2 | OHSRP Office of Compliance and Training / IRB Reporting | 47 |
| | 7.3 | NCI Clinical Director Reporting | 47 |
| | 7.4 | NIH Required Data and Safety Monitoring Plan | 47 |
| 8 | S | PONSOR PROTOCOL/SAFETY REPORTING | 48 |
| | 8.1 | Definitions | 48 |
| | 8.2 | Assessment of Safety Events | 49 |
| | 8.3 | Reporting of Serious Adverse Events | 49 |
| | 8.4 | Safety Reporting Criteria to the Pharmaceutical Collaborators | 50 |
| | 8.5 | Reporting Pregnancy | 50 |
| | 8.6 | Regulatory Reporting for Studies Conducted Under CCR-Sponsored IND | 50 |
| | 8.7 | Sponsor Protocol Deviation Reporting | 51 |
| 9 | C | CLINICAL MONITORING | 51 |
| 1( | ) | STATISTICAL CONSIDERATIONS | 51 |
| 1 | 1 | COLLABORATIVE AGREEMENTS | 52 |
| | 11.1 | Cooperative Research and Development Agreement (CRADA) | 52 |
| 12 | 2 | HUMAN SUBJECTS PROTECTIONS | 53 |
| | 12.1 | 1 Rationale For Subject Selection | 53 |
| | 12.2 | Participation of Children | 53 |
| | 12.3 | Participation of NIH Subjects Unable to Give Consent | 53 |
| | 12.4 | Evaluation of Benefits and Risks/Discomforts | 53 |
| | 12.5 | 5 Risks/Benefits Analysis | 54 |
| | 12.6 | 6 Consent Process and Documentation | 54 |
| 1. | 3 | REGULATORY AND OPERATIONAL CONSIDERATIONS | 55 |
| | 13.1 | 1 Study Discontinuation and Closure | 55 |
| | 13.2 | 2 Quality Assurance and Quality Control | 55 |

| 13.3 | Conflict of Interest Policy | 56 |
|---|---|---|
| 13.4 | Confidentiality and Privacy | 56 |
| 14 P | HARMACEUTICAL INFORMATION | 57 |
| 14.1 | Pomalidomide | 57 |
| 15 R | EFERENCES | 60 |
| 16 A | PPENDICES | 66 |
| 16.1 | APPENDIX A: Performance Status Criteria | 66 |
| 16.2 | APPENDIX B: Measurement of Pomalidomide Serum Levels | 67 |
| 16.3 | APPENDIX C: Diagnostic Criteria of Chronic GVHD | 68 |
| 16.4 | APPENDIX D: Clinical Differentiation of Acute and Chronic GVHD | 72 |
| 16.5 | APPENDIX E: Organ Specific and Global Scoring of Chronic GVHD | 73 |
| 16.6 | APPENDIX F: Global Scoring of cGvHD | 76 |
| 16.7 | APPENDIX G: Chronic GVHD Assessment (Clinician) Form | 77 |
| 16.8 | APPENDIX H: Calculations for Partial Response in Chronic GVHD | 81 |
| 16.9 | APPENDIX I: Calculations for Progression in Chronic GVHD | 82 |
| 16.10 | APPENDIX J: Chronic GVHD Cutaneous Assessment Worksheet (Adult) | 83 |
| 16.11 | APPENDIX K: Lee Symptom Scale | 85 |
| 16.12 | Appendix L: Pomalidomide Pregnancy Prevention Risk Management Plans | 87 |
| 16.13<br>and A | Appendix M: Pomalidomide Risks of Fetal Exposure, Pregnancy Testing Guidecceptable Birth Control Methods | |
| 16.14 | Appendix N: Pomalidomide Information Sheet | 92 |
| 16.15 | Appendix O: Medication Diary | 94 |
| 16.16 | Appendix P: Data Collection Elements Required By Protocol | 97 |
| 16.17 | Appendix Q:Chronic GVHD Composite Assessment Scale – Evaluation Tools | 99 |
| 16.18<br>SCOF | Appendix R: Chronic GVHD Composite Assessment Scale BARTHEL INDEX 132 | X |
| 16.19 | Appendix S: Chronic GVHD Composite Assessment Scale Frenchay activities 134 | Index |
| 16.20<br>yearly | | |


#### STATEMENT OF COMPLIANCE

The trial will be carried out in accordance with International Council for Harmonisation Good Clinical Practice (ICH GCP) and the following:

• United States (US) Code of Federal Regulations (CFR) applicable to clinical studies (45 CFR Part 46, 21 CFR Part 50, 21 CFR Part 56, 21 CFR Part 312, and/or 21 CFR Part 812)

National Institutes of Health (NIH)-funded investigators and clinical trial site staff who are responsible for the conduct, management, or oversight of NIH-funded clinical trials have completed Human Subjects Protection and ICH GCP Training.

The protocol, informed consent form(s), recruitment materials, and all participant materials will be submitted to the Institutional Review Board (IRB) for review and approval. Approval of both the protocol and the consent form must be obtained before any participant is enrolled. Any amendment to the protocol will require review and approval by the IRB before the changes are implemented to the study. In addition, all changes to the consent form will be IRB-approved; an IRB determination will be made regarding whether a new consent needs to be obtained from participants who provided consent, using a previously approved consent form.

## 1 INTRODUCTION

#### 1.1 STUDY OBJECTIVES

- 1.1.1 Primary Objective:
- 1.1.2 Determine whether pomalidomide is effective in persons with moderate or severe chronic graft-versus-host disease (cGvHD) not controlled by corticosteroids.
- 1.1.3 Secondary Objectives:
- 1.1.3.1 Determine whether pomalidomide is safe in persons with moderate or severe cGvHD not controlled by corticosteroids.
- 1.1.3.2 Determine the immune-modulatory effects of pomalidomide in persons with moderate or severe cGvHD.
- 1.1.3.3 Determine limited pharmacokinetics after oral administration of pomalidomide.

#### 1.2 BACKGROUND AND RATIONALE

## 1.2.1 Chronic Graft-Versus-Host Disease

cGvHD is an important late complication of allogeneic hematopoietic cell transplantation. It is a leading cause of mortality in persons more than 2 years post transplant. Symptoms of cGvHD usually appear within 2 years post transplant. Incidences range from 6%-80% depending on recipient age, donor type (related or unrelated, HLA matched or mismatched), graft type (blood, bone marrow or umbilical cord), graft manipulation or donor lymphocyte infusions. Chronic GvHD is strongly associated with prior acute GvHD (aGvHD). Traditionally the cutoff point between aGvHD and cGvHD was day 100 post transplant. In 2005 an NIH consensus project proposed two main GVHD categories, each with two subcategories: (1) "classic" aGvHD occurring within 100 days post transplant and (2) "persistent, recurrent or late" aGvHD. The broad


category of cGvHD includes: (1) "classic" cGvHD (without features or characteristics of aGvHD) and (2) an "overlap syndrome" with concordant features of cGvHD and aGvHD.<sup>3</sup> cGvHD is a multi-organ alloimmune and autoimmune disorder characterized by immune dysregulation, immunodeficiency, impaired organ function and decreased survival. It requires prolonged ongoing immunosuppression and inter-disciplinary management.

## 1.2.1.1 Pathophysiology

The pathophysiology of cGvHD is poorly understood. T- (both Th1 and Th2) and B-cells play a role in the pathogenesis of cGvHD, suggesting a general loss of tolerance, including abnormalities in the function of regulatory T-cells (Tregs). Natural Tregs (CD4+,CD25+,FoxP3+) maintain self-tolerance.<sup>6</sup> Studies in mice indicate Tregs can suppress GvHD and that a deficiency of Tregs worsens GHD.<sup>7</sup> There are conflicting data in humans concerning role of Tregs in the development of cGvHD.<sup>8</sup> A recent study suggested *in vivo* administration of low-dose IL-2 as a potential Tregmediated therapeutic approach for severe cGvHD.<sup>9</sup>

Several studies suggested that aGvHD is associated with predominant Th1-type immune response and cGvHD with Th2-type immune response. Th1 cells produce interferon-  $\gamma$  (IFN- $\gamma$ ) that mediates cell immunity, and Th2 cells produce interleukin (IL)-4, IL-5 and IL-13, which mediate humoral immunity. Following T-cell dysregulation, there is consequently cytokine dysregulation. In persons with cGvHD, higher levels of tumor necrosis factor- $\alpha$ , IL- 6, transforming growth factor- $\beta$ , IL-1 $\beta$  and lower levels of INF- $\gamma$  and IL-10 are reported.<sup>1,10-13</sup>

Autoimmunity and autoreactive T-cells have an important role in cGvHD. Some studies have shown that host thymus is not required for induction of cGvHD and that quiescent autoreactive T-and B-cells in transplants from non-autoimmune donors may be activated and expanded to cause cGvHD.<sup>14</sup> In contrast, involvement of thymus-dependent pathways in cGvHD development begins with injury to the thymus from a chemotherapy-conditioning regimen or aGvHD, leading to loss of B-cells with their ability to produce antibodies and to present antigen, which may enhance development of cGvHD. Autoantibodies like anti-nuclear, anti-mitochondrial, anti-parietal, anti-smooth muscle and anti-parotid are present in persons with cGvHD.<sup>15,16</sup> Also, persons with autoantibodies had more cGvHD-associated symptoms than persons without autoantibodies.<sup>15</sup> Autoantibodies against platelet-derived growth factor receptor (PDGFR) may play a role in cGvHD.<sup>17</sup> These PDGFR-α autoantibodies stimulate thyrosine phosphorylation in a cascade of events contributing inflammation and fibrosis.

The studies report elevated levels of BAFF (B-cell activating factor of the TNF family), which is produced by T-cells and granulocytes. BAFF supports differentiation and survival of normal B-cells in persons with cGvHD and autoimmune diseases.<sup>7,18</sup> Fuji et al. showed that in early-onset cGvHD, there are elevated sBAFF, sIL-2Rα, sCD13, and anti-dsDNA levels. In late-onset cGvHD, sBAFF, anti-dsDNA and ANA are higher, suggesting that the B-cell activation is predominant.<sup>19</sup> These observations create rationale for treatments with anti-CD20 antibodies in cGvHD.<sup>20</sup>All of these pathways are potential targets for cGvHD therapy. However, to date no laboratory parameter is considered a reliable biomarker for the diagnosis, measurement of severity, prognosis or therapeutic effect in cGvHD.

## 1.2.1.2 Clinical Manifestations

The usually affected organs in cGvHD are the skin, eyes, mouth, gut, liver, lungs, joints and genitourinary tract. Examples of diagnostic skin manifestations are sclerotic features and


poikiloderma, lichen-type and hyperkeratotic plaques in the mouth or bronchiolitis obliterans in lung biopsy.<sup>3</sup> The clinical manifestations of the disease are reminiscent of the autoimmune diseases such as systemic sclerosis, systemic lupus erythematosus or Sjögren syndrome.<sup>3</sup> According to the NIH consensus global scoring system, cGvHD is categorized as mild, moderate or severe. Systemic immune-suppressive therapy is usually indicated in persons with cGvHD involving 3 or more organs or with a severity score of 2 or higher in any organ. Systemic therapy is also to be considered in persons with thrombocytopenia (platelets <100x10<sup>9</sup>/L) or progressive onset during prednisone treatment.<sup>4</sup> cGvHD eventually leads to impaired functional performance, deteriorating quality of life, increased risk of infections and death.<sup>21-25</sup>

## 1.2.1.3 Treatment

Initial therapy for cGvHD is well established consisting of prednisone with or without a calcineurin inhibitor. However, only about 50% of persons have a durable response.<sup>6</sup> There are no standard recommendations for second-line treatment of cGvHD and there is no FDA approved agent. Recommendations for therapy are based on a long list of poorly standardized phase 2 trials or retrospective case analyses.<sup>26</sup> Diverse drugs (about 40 are described) are used, including sirolimus, tacrolimus, mycophenolate, methotrexate, extracorporeal photopheresis, monoclonal antibodies, pentostatin, imatinib and others. Choice between drugs is based on logistics, cost, failed prior treatments, toxicity profile and subject or clinician preferences.

For many years cGvHD has been difficult to address because of the lack of standardized criteria for diagnosis, staging and response to therapy. Recently, as an effort of the NIH-sponsored Consensus Development Project, a new series of guidelines have been published addressing diagnosis and staging, histopathology, biomarkers, assessment of response to therapy, ancillary therapy, supportive care and the design of clinical trials. <sup>22,27-31</sup> Typically, cGvHD usually lasts 2 to 5 years, and approximately 85% of survivors are able to discontinue systemic immune suppression. Five-year survival rates for persons who develop cGvHD range from 30% to 40% for high-risk persons and persons with cGvHD resistant to steroid therapy to 70% for standard-risk cGvHD persons. Treatment goals in management of cGvHD include both alleviation of symptoms and the control and reversion of the destructive immunological process. Therapy for cGvHD is largely unsatisfactory and persons should be treated on investigational clinical protocols whenever possible. <sup>23</sup>

## 1.2.2 Thalidomide in cGvHD

Thalidomide is effective in modulating cGvHD in rodents and has been tried for the prophylaxis and treatment of cGvHD in humans.<sup>32</sup> Thalidomide was found to have immune modulating effects from reduced production of TNF-α, costimulation of T-cells to produce IL-2 and IFNγ, inhibition of other cytokines such as IL-1β, IL-6 and IL-12 and down-regulation of cell surface adhesion molecules involved in leukocyte migration.<sup>26,33</sup> It also has anti-angiogenic properties.<sup>34</sup> Since the report by Vogelsang et al. in 1992 presenting thalidomide as a safe and effective treatment for severe cGvHD, several other phase 2 studies in children and adults reproduced these findings in salvage treatment of cGvHD. Historically, thalidomide is the third most commonly tested drug in trials of cGvHD second-line therapy.<sup>35</sup> Vogelsang et al. treated 44 persons with cGvHD who were high risk at diagnosis (21) or refractory (23) to conventional treatment with thalidomide for 3 months after a complete response (CR) and for 6 months after a partial response (PR). High-risk cGvHD was defined as having 2 out of following 3 characteristics: evolving from aGvHD, lichenoid skin or mucous-membrane changes and hepatic dysfunction. Absolute survival was 64%,


78% among persons receiving salvage therapy and 48% among those with high-risk cGvHD. Complete CR was achieved in 14 persons (7 high risk, 7 salvage), PR in 12 (1 high risk, 11 salvage) and no response in 18 (13 high risk, 5 salvage). The main side effects were sedation, neuropathy and constipation.<sup>36</sup> In the United States, thalidomide is FDA approved for erythema nodosum leprosum and in combination with dexamethasone for newly diagnosed multiple myeloma.<sup>37</sup>

Six other phase 2 studies have suggested efficacy of thalidomide in high-risk or refractory cGvHD (Table 1). Most trials were small but 3 had more than 30 subjects. Complete and partial remissions (variously defined) were reported with overall response rates of 20% to 86%. Heney et al.<sup>38</sup> reported responses in 5 of 6 persons, best in cutaneous involvement; 2 persons developed peripheral neuropathy. In a study in children by Rovelli et al., 10 subjects responded (6 CR, 4 PR).<sup>39</sup> Forsyth reported a thalidomide-responsive case of pulmonary cGvHD (brochiolitis obliterans). 40 Staumont-Salle reported a response in lichenoid vulvar lesions. 41 In study by Browne et al., 42 38% of subjects with cGvHD responded (46% children, 25% adults). In a 1995 study by Parker et al., 20% of subjects had sustained responses, and 36% discontinued because of side effects, including sedation, constipation, neuritis, neutropenia and rash. In a phase 2 study by Cole et al., 5 children received doses 100 to 800 mg—1 CR and 4 PRs were reported. Side effects were minimal, and there was no neuropathy. 43 Kulkarni et al. reported 13 CRs and 8 PRs in 59 subjects with cGvHD at thalidomide doses of 600 to 1200 mg/d. Two subjects had polyneuropathy, 2 had deep vein thrombosis (DVT) and 1 had thrombocytopenia. Mehta treated 6 children with cGvHD.<sup>44</sup> One child had a CR and one a PR. One child had a rash, eosinophilia and pancreatitis shortly after starting thalidomide, which resolved only after discontinuing thalidomide.

Two randomized trials (with approximately 50 subjects each) using thalidomide as part of the front-line therapy in cGvHD are reported. In one open-label, add-on to steroids and cyclosporine study, comparable response rates were seen in the thalidomide and control cohorts. The second study was a placebo-controlled trial using initial doses of 200 to 800 mg/d. Thalidomide had to be discontinued in 92% of persons in contrast to 65% in the placebo group due to intolerance, mostly neutropenia, sedation and neuropathy. A third randomized trial of thalidomide in cGvHD was performed by Chao et al. for cGvHD prevention. This study showed increased incidence of cGvHD and inferior survival in the thalidomide arm with such strategy. Collectively, these data suggest efficacy of thalidomide as salvage therapy for cGvHD but not for prevention or as front-line therapy.

In summary, several phase 2 trials report response rates of 20% to 83% with thalidomide doses of 100 to 1600mg/d.<sup>26,34</sup> Thalidomide doses higher than 200 mg/d are poorly tolerated. Phase 3 trials show, however, no benefit of thalidomide for front-line therapy and detrimental effect in cGvHD prevention. These data suggest that although thalidomide may be active at high doses in rodents, these doses cannot be reliably and safely achieved in humans. Developing pomalidomide, which has similar immune-modulating effects as thalidomide but less toxicity, is of considerable interest in cGvHD.

Table 1. Studies of Thalidomide in cGvHD

| Reference | Dose<br>(mg/day) | No. of Persons | Toxicities | Response Rate |
|---|---|---|---|---|
| Phase 2 salvage therapy | | | | |
| Heney et a | 1.38 100-200 | 6 | 2 PNS not stopped | 2 CR, 3 PR |
| 1991 | | | | |

| Reference | Dose | No. of | Toxicities | Response Rate |
|---|---|---|---|---|
| Reference | (mg/day) | Persons | TOXICITIES | Response Rate |
| Vogelsang et al. <sup>36</sup><br>1992, steroid<br>refractory or high-<br>risk cGvHD | 800-1600 | 44 | 4 PNS, 91% sedation<br>during first week, 24,<br>at least single episode<br>of constipation | 14 CR, 12 PR |
| Cole et al. <sup>43</sup> 1994 | 100-800 | 5 | 1 constipation | 1 CR, 4PR |
| Parker et al. <sup>48</sup> 1995 | 400-1200 | 80 | 3 PNS, 7 somnolence,<br>3 constipation, 6 skin<br>rash, 10 neutropenia | 9 CR, 7 PR |
| Rovelli et al. <sup>39</sup> | 100-800 | 14 | 0 | 6 CR, 4 PR |
| Browne et al. <sup>42</sup> 2000 | 200-800 | 37 | 1 constipation, 2 somnolence, 1 mild PNS, 2 severe whole-body erythema, one recovered, one died (toxic epidermal necrolysis) | 1 CR, 13 PR |
| Kulkarni S. <sup>49</sup> 2003 (thalidomide in combination with CSP, prednisone and azathioprine) | 600-1200 | 59 | 2 PNS, 2 DVT, 1 thrombocytopenia | 13 CR, 8 PR |
| Phase 3 front-line | therapy | | | |
| Koc et al. 46 2000 thalidomide versus placebo, given in combination with CSP (or tacrolimus) and prednisone | 200-800 | 52 (26<br>thalidomide,<br>26 placebo) | 14 neutropenia (stopped), 11 neurologic symptoms (stopped), 17 sedation, 10 constipation | Treatment with<br>the<br>study drug was<br>discontinued<br>before resolution<br>of cGvHD in 23<br>(92%) of persons |
| Arora et al. <sup>45</sup> 2001 CSP and prednisone versus CSP, prednisone, and thalidomide Phase 3 prevention | 200-800<br>(adults)<br>0.75-3 mg/kg<br>(children) | 54 (27 in each arm) | 17 sleepiness, 1 seizures, 14 constipation, 13 PNS, 2 TTP/HUS | CR+PR similar response in both groups at 2, 6 months and 1 year; no clinical benefit when included in initial therapy |


| Reference | Dose | No. of | Toxicities | Response Rate |
|---|---|---|---|---|
| | (mg/day) | Persons | | |
| Chao et al <sup>47</sup> 1996, | 200 mg BID | 59 subjects | | Increased |
| randomized at day | | randomized, | | incidence of |
| 80 after transplant | | 54 evaluable | | cGvHD and |
| | | (26 placebo, | | inferior survival |
| | | 28 | | in thalidomide |
| | | thalidomide) | | arm |

Abbreviations: PNS, polyneuropathy symptoms; CR, complete response; PR, partial response; DVT, deep venous thrombosis; CSP, cyclosporine; TTP/HUS, thrombotic thrombocytopenic purpura/hemolytic uremic syndrome.

## 1.3 POMALIDOMIDE

Pomalidomide is a novel immune-modulatory drug, a thalidomide analogue with 4,000-fold greater inhibition of TNF-α production relative to thalidomide (Celgene Corp data on file<sup>50</sup>). The pharmacodynamic (PD) properties of pomalidomide are of potential therapeutic benefit in the treatment of various hematologic malignancies (such as multiple myeloma and myeloproliferative neoplasm [MPN]–associated myelofibrosis and other hematologic disorders (like β-thalassemia and sickle cell disease) as well as solid cancers (prostate, thyroid and lung cancer). In addition, several features of pomalidomide suggest it may be useful in treating cGvHD, including: (1) in vitro suppression of TNF-α (human monocytes);<sup>51</sup> (2) increasing Th1 (mouse cancer vaccine, human CD4+ T-cells in vitro);<sup>52,53</sup> (3) suppression of Th2 (mouse cancer vaccine);<sup>52</sup> and (4) stimulation of IL-12 and sIL-2Rα (humans).<sup>54</sup> However, other effects of pomalidomide may have potential adverse effects in cGvHD, including: (1) increased CD45RO+ (memory) CD4 and CD8 T-cells (humans);<sup>54</sup> (2) decreased Tregs;<sup>55</sup> (3) increased Th2 (polarized human CD4+ T-cells in vitro);<sup>53</sup> and (4) increased B-cells (in vitro human CD19+ cells).<sup>56</sup> Because the precise pathogenesis of cGvHD is unknown (and may be different in different persons), it is impossible to predict the effect of therapy with pomalidomide outside of the context of a clinical trial.

## 1.3.1 Preclinical Studies

In a series of in vitro studies, pomalidomide exhibited several immune-modulating properties such as potent inhibition of TNF- $\alpha$  activity, IL-1 $\beta$ , IL-6, IL-12, monocyte chemoattractant protein (MCP)-1 and macrophage inflammatory protein, and production and inhibition of cellular cyclooxygenase-2, as well as modulation of angiogenesis. Pomalidomide also augmented the activity of natural killer (NK) cells and enhanced antibody-dependent cell-mediated cytotoxicity of targeted tumor cells in combination with therapeutic antibodies to tumor-specific surface antigens. Pomalidomide enhances T-cell stimulation by augmenting T-cell proliferation, increasing production of IL-2, IFN- $\gamma$  and RANTES, and decreasing IL-10 production. Furthermore, pomalidomide is a potent inhibitor of the proliferation of multiple myeloma cell lines in vitro and has been shown to be active in subjects with relapsed or refractory myeloma. <sup>54,57</sup> Based on its numerous mechanisms of carcinoma growth inhibition, pomalidomide is being tested as part of induction chemotherapy regimens and as post-induction maintenance therapy for solid cancers.

More information emerged recently about the specific mode of pomalidomide action as cereblon (*CRBN*), the primary target for thalidomide teratogenicity<sup>58</sup>, is now identified also as an essential


target for pomalidomide anti-myeloma activity.<sup>59</sup> The immediate result of this binding is interferon regulatory factor 4 (IRF4) down-regulation, which is also essential for Th-17 cell development.<sup>60,61</sup>

## 1.3.2 Animal Models

Oral pomalidomide is rapidly absorbed in rats and monkeys and the bioavailability is dose dependent, at high doses 100mg/kg, the bioavailability was low (15%) however at 2mg/kg the bioavailability was 100%. Following intravenous (IV) administration to rats and monkeys, pomalidomide exhibited low clearance (240 to 286 mL/h/kg), a moderate volume of distribution (2.2 to 2.5 L/kg), and a moderately long terminal half-life (approximately 6 hours). Renal excretion of metabolites was the predominant route of clearance in animal models. The toxicity of pomalidomide after oral and IV dosing was studied in rats and mice. There were no deaths and no significant clinical observations in rodents given a single dose of pomalidomide at 2000 mg/kg orally or up to 50 mg/kg IV. No treatment-related macroscopic changes were observed. In rats administered a single dose of 10, 25 and 50 mg/kg pomalidomide by IV injection, the high dose produced piloerection, hunching, and tachypnea. Palpebral closure was observed at doses of 25 and 50 mg/kg, and hyperpnea at 50 mg/kg. The severity and persistence of clinical observations increased with increased dose. Pomalidomide at oral doses of 100, 500 or 1500 mg/kg was well tolerated when given once daily to male and female rats for 90 consecutive days. Therefore, the no-observable-adverse-effect level (NOAEL) under the conditions of this study was 1500 mg/kg.

A 13-week study evaluated the toxicity and toxicokinetics of pomalidomide in male and female cynomolgus monkeys after oral doses of 0.05, 0.2, 2 or 10 mg/kg. Lesions in the bone marrow, spleen, and thymus were observed in animals dosed at 2 and 10 mg/kg. Based on the results from this study, the NOAEL was 0.2 mg/kg/day; the maximum plasma concentration (Cmax) and the area under the plasma concentration-time curve (AUC) values at this dosage were approximately 150 ng/mL and 600 ngh/mL, respectively. Since the monkey was identified as the most sensitive species in the toxicology program, the NOAEL of 0.2 mg/kg/day was used to calculate the human equivalent dose of 0.06 mg/kg or 3.8 mg for a 60 kg person. External and cardiac malformations were observed in fetuses of pregnant rabbits that were administered pomalidomide orally at 10, 100 and 250 mg/kg/day. A relationship was noted between increasing pomalidomide dose and the number of fetuses affected, as well as the frequency of occurrence of each type of malformation. Based on these data, it was concluded that pomalidomide causes fetal malformations in rabbits. A nonclinical safety PD study demonstrated no major safety concerns with cardiac and respiratory functions in dogs, rats or monkeys. In rats and monkeys pomalidomide administrated orally was absorbed fairly rapidly (T<sub>max</sub> of 2 to 4 hours) and had low oral bioavailability (13%-15%). Renal excretion was the predominant route of clearance in animal models.

In the mouse model of bleomycin-induced skin fibrosis, pomalidomide exerted potent anti-fibrotic effects and not only prevented progression of experimental fibrosis, but also induced regression of established fibrosis. In this model, pomalidomide reduced dermal thickening and reduced the numbers of myofibroblasts in the skin, whether it was administered prophylactically or therapeutically. These results show that pomalidomide exerts potent anti-fibrotic effects and not only prevents the progression, but also induces a regression of established fibrosis in a nonclinical model of skin fibrosis (Celgene, unpublished).

In multiple myeloma, pomalidomide induces growth arrest and/or apoptosis of multiple myeloma cells (via caspase-8 death receptor pathway), and it also reduces stromal cell expression of vascular


endothelial growth factor (VEGF) and basic fibroblast growth factor (bFGF), which decreases angiogenesis. <sup>62</sup> One characteristic of immune-modulatory drugs is their potency to act as a costimulus of T-cell receptor ligation, leading to increased production of IL-2 and INF-γ, indicative of a Th1 phenotype. <sup>63</sup> Pomalidomide promotes T-cell differentiation via the augmentation of T-bet, which leads to upregulation of INF-γ. <sup>63</sup> It also increases antibody-dependent cell cytotoxicity.

## 1.3.3 Experience in Humans

Pomalidomide is active in multiple myeloma and MPN-associated myelofibrosis. It has been also used to treat cGvHD. Given at doses up to 3 mg/day is usually well tolerated and main toxicities are neutropenia and thrombocytopenia, there have been no drug-related deaths in clinical trials with pomalidomide (summarized in Table 2).

## 1.3.3.1 Pharmacokinetics and Product Metabolism in Humans

A phase-1, single-center, single-blind, placebo-controlled, ascending single oral dose study (CC-4047 1398/132) was conducted to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of pomalidomide in 30 healthy male subjects, aged 19 to 55 years. Pomalidomide was administered orally in capsule form at 5 dose levels comprised of 1, 5, 10, 25, and 50 mg, and corresponding to 0.01, 0.07, 0.13, 0.30, and 0.59 mg/kg, respectively, when adjusted for group mean body weight. At each dose level, 4 subjects received pomalidomide and 2 subjects received placebo in a fasted state. A total of 20 subjects each received a single oral dose of pomalidomide in doses ranging from 1 mg to 50 mg, and 10 received placebo. Following each dose level of pomalidomide, the absorption of pomalidomide was moderately rapid. The maximum plasma concentration ( $C_{max}$ ) occurred at a median  $t_{max}$  of 2.5 to 6 hours postdose. The systemic exposure of pomalidomide as determined from the area under the plasma concentrationtime curve  $[AUC_{(0-tz)}]$  and  $AUC_{(0-\infty)}$  increased in an approximately dose-proportional manner, whereas  $C_{max}$  increased in a subproportional manner. After reaching  $C_{max}$ , plasma concentrations of pomalidomide declined in an apparent biphasic manner. The geometric mean terminal elimination half-life ( $t_{1/2}$ ) ranged from 8.2 to 10.8 hours, with no apparent dose-related trend. Less than 3% of the administered dose was excreted in urine as unchanged pomalidomide across all dose levels.

A phase-1b, single-center, ascending dose, open-label study (CDC-407-00-001) was conducted to identify the MTD and evaluate the safety and efficacy of pomalidomide in male and female subjects with relapsed or refractory Multiple Myeloma (MM). Pomalidomide was administered orally in capsule form at doses of 1, 2, 5, and 10 mg in either once daily dosing (Cohort 1) or alternate day dosing (Cohort 2) for 4 weeks. The study design did not allow for a precise calculation of subject numbers, as the number of subjects per dose group was dependent on the frequency of DLT. Subjects were enrolled in groups of 3 per dose group beginning with the 1-mg dose group. If no DLT were experienced (in one dose group) at a given dose level, the subsequent group of 3 subjects were to receive the next highest dose. If 1 of the 3 subjects in a dose group experienced a DLT, that cohort would then be expanded to 6 subjects. If 2 or more subjects in a cohort of up to 6 subjects experienced a DLT, no additional escalation of dose would occur. Escalations would occur until an MTD was established or the maximum dose of 10 mg/day was reached. A DLT was defined as a Grade 3 or higher non-hematologic toxicity or a Grade 4 or higher hematologic toxicity using the NCI CTC. A total of 45 subjects were enrolled in the study; 24 subjects in Cohort 1 and 21 subjects in Cohort 2. Blood samples for the


analysis of pomalidomide were collected from 28 subjects and included in the pharmacokinetic analysis. Dose levels of pomalidomide evaluated in the pharmacokinetic assessment were 1, 2, 5, and 10 mg once daily and 5 mg on alternate days. Blood and urine samples for analysis of plasma and urinary pomalidomide concentrations were collected for up to 24 hours after dosing on Day 1 and Week 4 (Day 29). Plasma concentrations (Geometric means and coefficient of variation percent [CV%]) of pomalidomide in subjects with MM on Day 1 and Week 4 are summarized in Figure 1 and Figure 2.

**Figure 1:** Plasma Concentrations of Pomalidomide on Day 1



OD = once daily; QOD = every other day.


Figure 2: Plasma Concentrations of Pomalidomide on Week 4



OD =once daily; QOD =every other day.

Following administration of pomalidomide at dose levels of 1, 2, 5, and 10 mg once daily and 5 mg every other day to subjects with MM, absorption of pomalidomide was steady with median  $t_{max}$  ranging from 1.5 to 4.0 hours postdose on Day 1 and Week 4. The mean  $t_{1/2}$  of pomalidomide was similar across dose levels and dosing days being approximately 7 to 8 hours.

At the 1 and 2 mg daily dose levels, there was slightly greater accumulation of pomalidomide in plasma upon multiple dosing than predicted. However, at the 5 mg daily and 5 mg alternate day dose levels, there was little or no accumulation of pomalidomide upon multiple dosing.

There was a less than dose proportional increase in  $AUC_{(0-\infty)}$  and  $C_{max}$  for pomalidomide over the 1 to 10 mg dose range on Day 1, with a more pronounced sub-proportional increase in both parameters on Week 4 over the 1 to 5 mg dose range.

The fraction of the dose excreted in the urine as unchanged drug was low for all dosing regimens, with a maximum of 4.5% being eliminated up to 24 hours after dosing on Day 1 and Week 4 for individual subjects.

#### 1.3.3.2 Clinical studies with Pomalidomide

In a phase 1 single-center, single-blind, placebo-controlled, ascending single-dose study, pharmacokinetics (PK), PD and safety of pomalidomide were studied in 30 healthy male subjects. The results demonstrated that pomalidomide administered at a dose of 1 to 50 mg has an acceptable safety profile. Adverse events (AEs) reported in the study were mild or moderate in nature and no clinically significant changes in any laboratory or other parameters, except a dose-related decrease in the CD4+ cell count, were observed.

A phase 1b study was conducted to identify the maximum tolerated dose (MTD) and evaluate safety and efficacy of pomalidomide in persons with relapsed or refractory multiple myeloma. A


total of 24 persons were treated with the dose-escalating regimen (1, 2, 5 and 10 mg). The MTD was 2 mg. Pomalidomide was well tolerated with no serious nonhematological AEs and excellent disease responses. Fifty-eight percent of persons developed grade 3/4 neutropenia and 16% of persons developed DVT. <sup>64</sup> In this study, the cytokines were measured and it was noticed that the serum IL-12 and sIL-2 levels increased during the first 4 weeks of treatment. IL-12 is derived from monocytes and macrophages and has a key role in amplifying a Th1-type response. <sup>65</sup> No significant changes and no correlation was found between IL-6, TNF-α, IL-10, VEGF and bFGF levels and paraprotein response.

A standard dose escalation phase 1 study was conducted to determine the MTD of pomalidomide at 1 mg, 2 mg, 5 mg, and 10 mg on alternate days in persons with relapsed myeloma. Patients were evaluated prior to study enrolment and weekly for the first month and monthly thereafter. The overall response rate (>50% reduction in paraprotein) to pomalidomide monotherapy was 50%. Hematological monitoring over 4 weeks showed significant decline in hemoglobin, white blood cells, and neutrophils. Platelets decreased but without statistical significance. Significant decrease was noticed in the B-cell percentage (P=0.002) and absolute B-cell number. The CD3+ percentage and CD8+ percentage increased (P=0.003, P=0.007). The CD4+ percentage and absolute as well as NK cell percentage were increased but without statistical significance. There was a significant negative association between B-cell percentage or absolute B-cell count at 4 weeks and maximal percentage change in paraprotein (P=0.05, P=0.03).

Tefferi et al. published a phase 2 randomized, multicenter, double-blind study of pomalidomide in MPN-associated myelofibrosis. Four arms were studied pomalidomide (2 mg) plus placebo, pomalidomide (2 mg) plus prednisone, pomalidomide (0.5 mg) plus placebo and pomalidomide (0.5 mg) plus prednisone. Pomalidomide was well tolerated. Anemia response rate was up to 40%. There was relatively low incidence of grade ≥3 neutropenia and thrombocytopenia. How pomalidomide works in MPN-associated myelofibrosis is unclear, but it is known that TNF-α directly inhibits erythropoiesis in vitro. In this study it was also described that overall bone marrow cellularity, degree of fibrosis, or cytogenetic findings did not change (bone marrow examination was done in 4 responders who completed 1 year treatment with pomalidomide with or without prednisone.

A multicenter, randomized, phase 2 study of pomalidomide in combination with low-dose dexamethasone was conducted in patients with relapsed/refractory myeloma who received prior therapy (lenalidomide or bortezomib). Pomalidomide 2 mg po daily was given on days 1 through 28 of a 28-day cycle. Dexamethasone 40 mg daily was given on days 1, 8, 15 and 22 of each cycle. Thirty-eight patients achieved objective response (63%), including CR in 5%, very good PR in 28% and PR in 30%. Responses were seen in 40% of lenalidomide-refractory persons, 37% thalidomide-refractory and 60% of bortezomib-refractory persons. Toxicity was primary myelosuppression. Grade 3 or 4 hematologic toxicity consisted of anemia (5%), thrombocytopenia (3%) and neutropenia (32%). Among those that developed grade 3/4 neutropenia, all first experienced the neutropenia in cycle 1-3; no new patients experienced grade 3/4 neutropenia in cycle 4 or later. One patient experienced thromboembolic event. The most common nonhematologic grade 3 or 4 toxicities consisted of fatigue (17%) and pneumonia (8%); less than 5% of patients experienced neuropathy, diarrhea, constipation or hyperglycemia. One patient (1.6%) had a thromboembolic event of DVT.

In a phase 1/2 study in MPN-associated myelofibrosis with 19 patients, 3 mg was determined to be the MTD, but no efficacy was observed at that dose. Two of three patients in the 3.5 mg cohort


had dose-limiting myelosuppression. Overall, 7 subjects had an anemia response and 2 a spleen response.

In another trial of pomalidomide in MPN-associated myelofibrosis, low-dose pomalidomide (0.5 mg/day) was given to 58 persons. Anemia response was documented only in persons with JAK2V617F (24 vs 0%; P=0.03). Nine of the 10 anemia responders became red blood cell–transfusion independent. Fourteen of 24 persons with platelets ≤100x10e9 /L had a greater than 50% increase in platelets. Grade 3 or 4 thrombocytopenia/neutropenia occurred rarely. This study established low-dose pomalidomide as effective and safe in MPN-associated myelofibrosis with anemia.

#### 1.3.3.1 Pomalidomide in cGvHD

Pusic et al. reported results of a phase 2 study of pomalidomide in patients with cGvHD not controlled by corticosteroids.<sup>67</sup> Eight subjects received 3 mg/day with dose reductions to 2 mg, 1 mg and 0.5 mg. Seven subjects required dose reduction because of muscle cramps, tremor and fatigue. Five subjects discontinued therapy for worsening of cGvHD of the skin and mouth (N=1), pain (N=1) and no response (N=3). No bone marrow suppression, somnolence, constipation or DVT were observed. Three persons reached the primary evaluation endpoint at 6 months at the 2 mg dose (N=2) or 1 mg dose (N=1). The 3 patients had global PRs per NIH criteria (skin erythema, GI) and <PR ongoing improvements in the skin, mouth and eyes. This study established feasibility of giving pomalidomide to humans with cGvHD and the absence of serious side effects at doses less than 2 mg/day.


**Table 2. Clinical Studies of Pomalidomide** 

| Reference | Setting | Study<br>Design | Study<br>Duration | Dose | N | MTD | Toxicities | Response Rate |
|---|---|---|---|---|---|---|---|---|
| Phase 1 | | | • | | | | | |
| Celgene,<br>not<br>published | Healthy<br>volunteers | Single-blind,<br>placebo-<br>controlled,<br>ascending<br>single dose | | 1, 5, 10, 25, 50 mg | 30, 10 received placebo | N/A | Mild or moderate<br>AEs; no clinically<br>significant changes<br>in any laboratory<br>parameter tested | N/A |
| Streetly et al.,2008 <sup>64</sup> | Relapsed<br>MM | Standard<br>dose<br>escalation | 4 weeks | 1, 2, 5, 10<br>mg | 20 | 5 mg | 10 mg, grade 4<br>neutropenia in 3/3<br>pts, DVT 0% | 10% CR and >50% reduction in paraprotein in 50% |
| Schey et al., 2004 <sup>65</sup> | Relapsed or refractory MM | Dose<br>escalating<br>regimen | 4 weeks | 1, 2, 5, 10<br>mg | 24 | 2 mg | Grade 3/4<br>neutropenia in<br>58% pts and DVT<br>in 16% | 17% CR, >25% reduction in paraprotein in 67%, >50% reduction in paraprotein in 54% |
| Phase 2 | | | • | | | | | |
| Tefferi et al. 2009 <sup>37</sup> | Anemia<br>associated<br>with<br>myelofibrosis | Randomized,<br>double-<br>blind,<br>multicenter | Up to 12<br>28-day<br>treatment<br>cycles | 4 arms (2 mg+ placebo, 2 mg + prednisone, 0.5 mg + prednisone, and prednisone + placebo | 84 | 2 mg | Relatively low incidence of grade ≥3 neutropenia and thrombo-cytopenia | Response in anemia 20 pts (40%) 23%, 2 mg/d + placebo; 16%, 2 mg/d + prednisone; 36%, 0.5 mg/d + prednisone; 19%, prednisone + placebo |


| Mesa et al., 2009 <sup>68</sup> | Myelofibrosis | Phase 1/2,<br>multicenter<br>dose<br>escalation | 28 days | 2.5, 3.0 and<br>3.5 mg/day;<br>no efficacy<br>at 3 mg,<br>dose<br>reduction to<br><b>0.5 mg</b> | 19 | 3 mg | DLT myelosuppression in 2/3 pts in 3.5 mg cohort | 7 pts anemia response, 2 spleen response |
|---|---|---|---|---|---|---|---|---|
| Lacy et al., 2009 <sup>69</sup> | Relapsed<br>MM | Multicenter | 2 mg/d<br>on days<br>1-28 of a<br>28-day<br>cycle,<br>dexame-<br>thasone<br>40 mg<br>on days<br>1, 8, 15,<br>22 | 2mg/day | 60 | | Primarily myelosuppression. Grade 3 or 4 hemato-logic toxicity consisted of anemia (5%), thrombo-cytopenia (3%) and neutropenia (32%) | Objective response in 63%, including CR in 5%, very good PR in 28% and PR in 30% |
| Begna et al., 2011 <sup>70</sup> | Myelofibrosis<br>(JAK2V617F<br>positive) | Single-<br>center | 28-day<br>cycles:<br>84% pts<br>had ≥3<br>cycles | 0.5 mg/day,<br>after 6<br>cycles<br>2 mg/day | 58 | 2 mg | No AE reason for<br>stopping therapy. 1<br>pt neuropathy, 1 pt<br>grade3/4 thrombo-<br>cytopenia | 10 (17%) anemia response, 20% anemia RR in pts who received ≥3 cycles |
| Pusic et al., 2010 <sup>67</sup> | cGvHD | Multicenter, response evaluated every 3 months | | 3 mg/day<br>with dose<br>reductions<br>to 2, 1 and<br>0.5 mg/day | 8 | 3 mg | Muscle cramps,<br>tremor and fatigue | 2 CRs, 1 PR<br>(3 pts reached<br>6 months) |


## 1.4 STUDY DESIGN AND RATIONALE

Better therapies for cGvHD are needed. In about 50% of persons with cGvHD, the disease does not respond to corticosteroids, and there is no standard second-line therapy or FDA-approved drug for cGvHD. Thalidomide is an immune-modulating drug effective in a rodent model of cGvHD and in humans for salvage therapy after failure of steroids, but at doses expected to be effective it is associated with troublesome side effects including somnolence, neuropathy and constipation, which precluded wider use in this population. Pomalidomide is a new immune-modulating drug that is more potent than thalidomide and has been shown in early trials in cancer and cGvHD to be without the toxicities that limited the use of thalidomide. Several biological features of pomalidomide suggest that this drug may be useful in treating cGvHD. Since the precise pathogenesis of cGvHD is unknown, the most compelling evidence for testing pomalidomide in a clinical trial is the encouraging efficacy data with thalidomide. Preliminary studies of pomalidomide in persons with cGvHD suggest absence of typical thalidomide-related side effects or significant myelosuppression and a preliminary suggestion of efficacy if doses of less than 3 mg/day could be given for at least 6 months (the typical primary response evaluation time point in cGvHD trials).

The use of the NIH Consensus Diagnosis, Staging Criteria now provides an updated, standardized assessment of persons with cGvHD for inclusion in clinical trials.<sup>71,72</sup> Although NIH Consensus Response Criteria are not yet validated in large clinical trials there are preliminary data on validity and reproducibility that provide guidance for further use and testing.<sup>73</sup>

At the intramural NCI there is a well-established clinical research infrastructure, the "NIH Chronic GVHD Study Group," that is uniquely qualified to conduct drug development studies and cGvHD assessments in a multi-disciplinary specialty setting. This environment is also uniquely conducive for further studies of cGvHD biology and in vivo pomalidomide effects by using the ETIB immunology pre-clinical core and the established cGvHD murine models expertise. The proposed study is not only expected to address a specific clinical therapeutic question related to pomalidomide in cGvHD but also allows establishment of experience with this important group of agents in general in patients after allogeneic hematopoietic stem cell transplantation.

The proposed study is a randomized phase 2 trial with the single stage selection design Patients will receive either a constant low dose of pomalidomide (0.5 mg/day) for six months or a strategy of increasing dose of pomalidomide from 0.5 mg/d up through each individual patients' maximum tolerated dose, with escalations by 0.5 mg/d every 2 weeks to a maximum of 2.0 mg/d. To protect patient safety, an early stopping rule will be implemented as outlined in section 8. With two arms, each of which has a maximal accrual of 16 patients, up to 32 evaluable patients will be randomized. Response assessments will occur every 3 months with primary efficacy endpoint evaluated at 6 months. Patients with responding disease will continue therapy for another 6 months.


#### 2 ELIGIBILITY ASSESSMENT AND ENROLLMENT

#### 2.1 ELIGIBILITY CRITERIA

#### 2.1.1 Inclusion Criteria

- 2.1.1.1 Moderate or severe cGvHD diagnosed and staged per NIH criteria (Filipovich et al 2005)<sup>22</sup>, Appendix C, Appendix D, Appendix E and Appendix F..
- 2.1.1.2 ≥18-75 years of age, because no dosing or adverse event data are currently available on the use of pomalidomide in persons <18 years of age
- 2.1.1.3 Has cGvHD that did not respond to high-dose corticosteroids (average 0.5 mg/kg/d prednisone for ≥8 weeks) or second-line systemic therapy
- 2.1.1.4 If taking systemic therapy for cGvHD at the time of enrollment, must be on a stable or tapering schedule in the preceding 4 weeks (extracorporeal photopheresis has to be stopped at least by 4 weeks before enrollment)
- 2.1.1.5 Karnofsky performance score ≥60% (Appendix A)
- 2.1.1.6 Life expectancy > 3 months
- 2.1.1.7 Stable primary malignancy for previous 3 months
- 2.1.1.8 Agree to adhere to methods of contraception and other fertility control measures as prescribed by the protocol
  - Agents of this class are known to be teratogenic, women of child-bearing potential and
    men must agree to use effective forms of contraception (hormonal or barrier method of
    birth control; abstinence) prior to study entry and for the duration of study participation.
    Should a woman become pregnant or suspect she is pregnant while she or her partner
    is participating in this study, she should inform her treating physician immediately.
  - Female Subjects
    - o Females of childbearing potential (FCBP)<sup>†</sup> must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10 − 14 days prior to and again within 24 hours of starting pomalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, one highly effective method and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking pomalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a vasectomy. All patients must be counseled every 28 days about pregnancy precautions and risks of fetal exposure through the POMALYST REMS™ program. See Appendix M: Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods.

## Male Subjects

 Must agree to use a latex condom during sexual contact with females of childbearing potential while participating in the study and for at least 28 days

<sup>&</sup>lt;sup>†</sup> A female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).


- following discontinuation of study drug even if he has undergone a successful vasectomy
- Will be warned that sharing study drug is prohibited and will be counseled about pregnancy precautions and potential risks of fetal exposure
- o Must agree to abstain from donating blood, semen, or sperm during study participation and for at least 28 days after discontinuation of study drug.
- Must agree that if a pregnancy or a positive pregnancy test does occur in a study subject or the partner of a male study subject during study participation, study drug must be immediately discontinued.
- Patients must agree to not share study drug with anyone during participation in the study.
- 2.1.1.9 Ability of subject to understand and the willingness to sign a written informed consent document.
- 2.1.1.10 All study participants must be registered into the mandatory POMALYST REMS<sup>TM</sup> program, and be willing and able to comply with the requirements of the POMALYST REMS<sup>TM</sup> program.

## 2.1.2 Exclusion Criteria

- 2.1.2.1 Acute GvHD, classic (\( \leq \text{day } 100 \)) or late-onset (\( \leq \text{day } 100 \)) Appendix D
- 2.1.2.2 Systemic immune suppression or systemic therapy for cGvHD started within preceding 4 weeks including extracorporeal photopheresis
- 2.1.2.3 Hypersensitivity to thalidomide, lenalidomide or pomalidomide
- 2.1.2.4 Any serious medical condition which places the subject at an unacceptable risk if he or she were to participate in the study or confounds the ability to interpret data from the study, including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
- 2.1.2.5 Neutrophil <1.0x10<sup>9</sup>/L, platelets <75x10<sup>9</sup>/L, estimated creatinine clearance <50 mL/min/1.73m<sup>2</sup> (Cockroft-Gault formula) total bilirubin >3 mg/dL, transaminase >3xUNL
- 2.1.2.6 Uncontrolled infection
- 2.1.2.7 Active HIV-1, HBV and/or HCV infection
- 2.1.2.8 Uncontrolled arrhythmias or symptomatic heart disease or LVEF <45%
- 2.1.2.9 Other cancer except that for which the transplant was done <2 years before study entry, except non-melanoma skin cancer or carcinoma in situ of the uterine cervix or breast
- 2.1.2.10 Taking other investigational drugs
- 2.1.2.11 NIH lung score 3 (Appendix E)
- 2.1.2.12 Pregnant women are excluded from this study because pomalidomide has potential for teratogenic effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with pomalidomide, breastfeeding must be discontinued while the mother is taking study drug and for at least 28 days after discontinuation of study drug. These potential risks may also apply to other agents used in this study.


#### 2.1.3 Recruitment

Subjects will be recruited from NIH Clinical Center hematopoietic stem cell transplant clinics but could be referred from the outside institutions. Study participants will be primarily recruited from the 04-C-0281 cGvHD natural history study protocol, which currently has more than 260 persons registered and enrolls approximately 3 persons per month, most of them with moderate or severe cGvHD. Referrals will be also accepted from the other NIH protocols or from the extramural community. Every effort will be made to screen potential candidates through the existing 04-C-0281 natural history protocol, which is a non-therapeutic study as part of pre-enrollment evaluations. The patient population enrolled on this study is expected to be representative of the population of persons receiving allogeneic hematopoietic stem cell transplantation at the NIH and nationwide.

## 2.2 REQUIRED TESTING AND COUNSELING FOR FCBP AND PARTNERS OF FCBP

## 2.2.1 During study participation and for 28 days following discontinuation of study drug:

- Pregnancy tests for females of childbearing potential. A female of childbearing potential (FCBP) is a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
- Pregnancy tests must occur 10 14 days and again within 24 hours prior to initiation of pomalidomide. FCBP with regular or no menstruation must have a pregnancy test weekly for the first 4 weeks and then every 28 days while on therapy (including breaks in therapy); at discontinuation of pomalidomide and at Day 28 post the last dose of pomalidomide. Females with irregular menstruation must have a pregnancy test weekly for the first 4 weeks and then every 14 days while on therapy (including breaks in therapy), at discontinuation of pomalidomide and at Day 14 and Day 28 post the last dose of pomalidomide (see <a href="Appendix M">Appendix M</a>: Pomalidomide Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods).
- All patients must be counseled about pregnancy precautions, risks of fetal exposure and other risks. The counseling must be done every 28 days and at drug discontinuation through the POMALYST REMS<sup>TM</sup> program. See <u>Appendix M</u>: Pomalidomide Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods.

## 2.3 SCREENING EVALUATION

Screening procedures may be performed on a CCR screening protocol, most commonly on 04-C-0281 "Natural History of Chronic GVHD." All studies must be completed within 8 weeks prior to enrollment:

- History and physical exam, Karnofsky performance score
- Documentation of cGvHD diagnosis, NIH organ and global severity stage
- CBC, platelets, differential, PT/PTT, serum chemistries (including sodium, potassium, chloride, CO<sub>2</sub>, calcium, magnesium, phosphorus, blood urea nitrogen [BUN], creatinine, glucose, albumin, total protein, alkaline phosphatase, total bilirubin, AST [SGOT], ALT


[SGPT], lactate dehydrogenase [LDH], and uric acid), urinalysis, urine pregnancy testing, TSH

- Infectious serology markers (HIV-1, HBV, HCV)
- Determination of estimated creatinine clearance
- Pulmonary function testing, CT of the chest (BOS sequence), cardiac ECHO, ECG
- Social work screening consult

For baseline evaluations, please see Section 2.6.

## 2.4 REGISTRATION PROCEDURES

Authorized staff must register an eligible candidate with NCI Central Registration Office (CRO) within 24 hours of signing consent. A registration Eligibility Checklist from the web site (<a href="http://home.ccr.cancer.gov/intra/eligibility/welcome.htm">http://home.ccr.cancer.gov/intra/eligibility/welcome.htm</a>) must be completed and sent via encrypted email to: NCI Central Registration Office (HOIS) <ncicentralregistration-l@mail.nih.gov. After confirmation of eligibility at Central Registration Office, CRO staff will call pharmacy to advise them of the acceptance of the patient on the protocol prior to the release of any investigational agents. Verification of Registration will be forwarded electronically via email to the research team. A recorder is available during non-working hours.

## 2.5 TREATMENT ASSIGNMENT AND RANDOMIZATION PROCEDURES

#### **Cohorts**

| Number | Name | Description |
|---|---|---|
| 1 | cGvHD Patients | Patients with moderate or severe cGvHD as per NIH criteria that has not responded to high-dose corticosteroids or second-line therapy. |

#### Arms

| Number | Name | Description |
|---|---|---|
| 1 | Experimental 1 | 0.5 mg/day without Dose Escalation |
| 2 | Experimental 2 | 0.5 mg/day with Dose Escalation by 0.5 mg/day increments every 2 weeks to a maximum of 2.0 mg/day |

## Randomization and Arm Assignment

Randomization will be done at the time of enrollment by the Central Registration Office, which will perform the randomization using randomization assignments determined by the study statistician. Subjects will be randomized to one of two treatment arms: low dose (0.5 mg/d) and high dose (0.5, escalating every two weeks to 1.0. 1.5 or 2.0 mg/d) pomalidomide. If one of the arms closes due to futility, toxicity or completion, enrollment will continue to the remaining arm.


#### 2.6 BASELINE EVALUATION

Following studies will be performed at the baseline before/after the enrollment and within four weeks prior to starting taking the study drug unless otherwise indicated below:

- History and physical exam, Karnofsky performance score
- CBC, platelets, differential, PT/PTT, serum chemistries (including sodium, potassium, chloride, CO<sub>2</sub>, calcium, magnesium, phosphorus, blood urea nitrogen [BUN], creatinine, glucose, albumin, total protein, alkaline phosphatase, total bilirubin, AST [SGOT], ALT [SGPT], lactate dehydrogenase [LDH], and uric acid), CRP, total complement and C3 and C4, urine pregnancy testing (once within 10-14 days prior to the start of study drug and again within 24 hours prior to the start of study drug), immunoglobulin levels, TBNK, blood CMV PCR, drug levels if pertinent (e.g., cyclosporine, tacrolimus, sirolimus)
- MRI of the involved extremity if clinically indicated (acceptable if done within 8 weeks)
- Documentation of cGvHD per NIH criteria (diagnostic, distinct, other and common manifestations), NIH organ and global stage, baseline assessments (form A and form B) per NIH response criteria, date of cGvHD diagnosis, prior and current treatments, prednisone or other steroids oral dose, and other patient, donor and transplant characteristics per Appendix Q.
- Specialty evaluations of cGvHD: dermatology, ophthalmology, dental, rehabilitation and occupational therapy, gynecology if applicable (can be done up to two weeks after starting study drug, except for dermatology and dental evaluations which must be done prior to starting study drug)
- Diagnostic and research biopsies of the skin and mouth (all persons), and other organs (only if clinically indicated)
- ECG
- Research laboratory (blood, saliva, urine)
- Study drug dispensation
- Subject diary review
- Documentation of concurrent medications

## 3 STUDY IMPLEMENTATION

## 3.1 STUDY DESIGN

The study is a randomized phase 2 trial with the single stage selection design. It is known from prior trials that the maximum tolerated dose of pomalidomide is about 3 mg/d in persons with bone marrow disorders receiving prior therapies for cancer, in cGvHD doses <3 mg/d have been well tolerated. This study will explore clinical toxicity of gradual escalation of pomalidomide doses <3 mg/d in subjects with cGvHD. Patients will receive either a constant low dose of pomalidomide (0.5 mg/day) for six months or a strategy of increasing dose of pomalidomide from 0.5 mg/d up through each individual patients' maximum tolerated dose, with escalations by 0.5 mg/d every 2 weeks to a maximum of 2.0 mg/d. In each of the two arms, the trial will use a single stage design.


As an early stopping rule for futility as outlined in section **8**, if after 7 patients have enrolled on either arm, 0 have responded, then no further patients will be accrued to that arm as soon as this can be determined. To protect patient safety, an early stopping rule will be implemented. With two arms, each of which has a maximal accrual of 16 patients, up to 32 evaluable patients will be randomized. Safety assessments and pregnancy testing for FCBP will be performed at scheduled intervals as described in the Study Calendar.

Response will be assessed every 3 months while taking pomalidomide following the criteria in Section 6.2. The primary efficacy endpoint will be evaluated at 6 months. Efficacy outcome is defined as clinical response (CR or PR) in subjects who enter the study with stable cGvHD or stable disease for ≥3 mo for subjects with progressive cGvHD at study-entry. (Stability will be assessed by the clinician and by the clinical exam at the screening evaluation based on the clinician estimate of the disease trajectory during the 3 months pre-randomization). Subjects who meet the response criteria at 6 months will continue therapy for another 6 months. If in the subject's best interest, efforts will be made to provide access to study drug on compassionate basis beyond the 12-month study endpoint.

Patients who discontinue therapy for any reason will be followed for up to 24 months after starting pomalidomide as described in Section **6.1.3**.

Concurrent topical and ancillary treatments for cGvHD are allowed per standards of care and will be recorded (see Section 4).<sup>27</sup> Other systemic immune suppression must stay stable or be tapered (systemic immunosuppression taper should be attempted no earlier than after 4-6 weeks on study), throughout the treatment with pomalidomide (with up to 2 steroid pulses allowed for disease stabilization per Section 4.1).

## **Study Schema**



treatment (primary endpoint at 6 months)

## 3.1.1 Dose-Limiting Toxicity

DLT will be defined as any grade ≥3 adverse event which is thought to be probably or definitively related to the investigational drug administration (notable exceptions where grades 2 or lower can be considered as DLTs are indicated in Table 4 below in Section 3.3). In addition, any persons who are unable to tolerate the dose to which they are assigned will be counted as a DLT at the maximum dose explored for that patient. The time frame for evaluation in which toxicity will count towards a DLT will be up to 28 days after therapy received at a given dose


level. In addition, a grade  $\geq$  3 AE will not be considered as DLT if the adverse event is attributed to a GVHD flare and responds to steroid pulse therapy as outlined in section 4.1. Whether treated on either arm, if there are 2 patients in the first 6 who experience a DLT from a given dose level, then no further patients will be treated at that dose level on the trial, regardless of arm. Furthermore, when more than 6 patients have received a given dose level, if at any time 33% or more patients experience a DLT when treated at that dose level, then no further patients will be treated at that dose level. Data from all subjects who receive  $\geq$ 1 dose of pomalidomide will be include in the safety analysis.

## 3.1.2 Dose Escalation

All subjects, independently of the randomization arm, will start pomalidomide at 0.5 mg/d. Those randomized to the high-dose arm will escalate to the target dose level by increasing the pomalidomide dose in 0.5 mg increments (**Table 3**) every 2 weeks to the next level. If the escalation is not tolerated, the patient will be treated on the next lower dose level. MTD designation will be given to the highest dose in which no more than 1 DLT occurred per cohort.

| | 1 ( 0 ) |
|--------------------------------|----------------------------|
| Dose Level | Dose |
| <b>Starting Dose (level 1)</b> | 0.5 mg daily on Days 1-14 |
| Dose Level 2 | 1.0 mg daily on Days 15-28 |
| Dose Level 3 | 1.5 mg daily on Days 29-42 |
| Dose Level 4 | 2.0 mg daily on Days 43-56 |

Table 3. Pomalidomide Dose Escalation Steps (high-dose arm)

#### 3.2 DRUG ADMINISTRATION

Pomalidomide will be given as 0.5 mg, 1.0 mg, or 2.0 mg capsules to be taken orally once a day on days 1–28 of a 28-day cycle. Each daily dose of pomalidomide should be taken at approximately the same time of day. Patients will be asked to complete a medication diary (Appendix P).

Pomalidomide capsules should be swallowed whole, and should not be broken, chewed or opened.

If a dose of pomalidomide is missed, it should be taken as soon as possible on the same day. If it is missed for the entire day, it should not be made up.

Patients who take more than the prescribed dose of pomalidomide should be instructed to seek emergency medical care if needed and contact study staff immediately.

Patients are instructed to fast (water or clear fluids only) for at least 2 hours prior to taking a dose to at least 1 hour post dosing. Pomalidomide should not be swallowed concurrently with other allowed medications while on-study.

## 3.2.1 Drug Dispensing

Pomalidomide (POMALYST®) will be provided to research subjects for the duration of their participation in this trial at no charge to them or their insurance providers. Pomalidomide will be provided in accordance with the Celgene Corporation's POMALYST REMS<sup>TM</sup> program. Per the standard POMALYST REMS<sup>TM</sup> program requirements, all physicians who prescribe pomalidomide for research subjects enrolled into this trial, and all research subjects enrolled into


this trial, must be registered in and must comply with all requirements of the POMALYST REMS<sup>TM</sup> program.

Drug will be shipped on a per patient basis by the contract pharmacy to the NIH pharmacy for IND studies. Only enough pomalidomide for one cycle of therapy will be supplied to the patient each cycle. This is in accordance with the POMALYST REMS<sup>TM</sup> program.

## Only enough pomalidomide capsules for 1 cycle of therapy may be provided to the patient each cycle.

Patients will be asked to maintain a dairy and bring to the next appointment all remaining capsules.

#### 3.3 DOSE MODIFICATIONS

Patients requiring dose reduction will be reassigned to one of the lower dose cohorts being evaluated: 0.5, 1.0 or 1.5 mg. Patients may be dose reduced to the lowest possible dose, i.e. 0.5 mg. For any dose reductions or if study drug needs to be held greater than 35 days, the Principal Investigator (PI) or Lead Associate Investigator (LAI) must be contacted. Once a dose has been reduced, it cannot be re-escalated. At the discretion of the PI, the use of granulocyte colony-stimulating factor (G-CSF) will be permitted to manage neutropenic fever or a Grade 4 neutropenia. Given the potentially long treatments delays, patients must have received 75% of the doses prescribed to be considered evaluable for the primary study endpoint.

**Table 4. Dose Modifications** 

| Common<br>Terminology<br>Criteria (CTCAE)<br>Version 4.0 | Adverse Event | Dose Change for Pomalidomide |
|---|---|---|
| Allergy/ Immunology | Allergic reaction/ hypersensitivity (including drug fever) - Grade 2 | Hold study drug until resolved to < Grade 1; Decrease dose by 1 dose level |
| Allergy/Immunology | Allergic reaction/ hypersensitivity (including drug fever) - Grade 3 or 4 | Discontinue Study Drug |
| Blood/Bone Marrow | Neutropenia (ANC) - Grade 3 with fever or Grade 4 | Hold study drug until < Grade 2;<br>Decrease dose by 1 dose level |
| Blood/Bone Marrow | Thrombocytopenia - Grade 3 or 4 | Hold study drug until <grade 2;<br="">Decrease dose by 1 dose level</grade> |
| Blood/Bone Marrow | Anemia - Grade 3 or 4 | Hold study drug and treat anemia as needed until Hgb within 0.5 g/dL of lower limit of normal; Decrease dose by 1 dose level |

| Common<br>Terminology<br>Criteria (CTCAE)<br>Version 4.0 | Adverse Event | Dose Change for Pomalidomide |
|---|---|---|
| Cardiac Arrhythmia | Grade 2 | Hold study drug until resolved to < Grade 1; Decrease dose by 1 dose level |
| Cardiac Arrhythmia | Grade 3 or 4 | Discontinue study drug |
| Prolonged QTs<br>Interval | Grade 3 (>0.50 second) | Hold study drug; decrease dose by 1 dose level and restart when resolved to < Grade 2 |
| Prolonged QTs<br>Interval | Grade 4 (>0.50 second, life threatening symptoms) | Discontinue study drug |
| Vascular | Thrombosis/embolism - Grade 2, 3 or 4 | Discontinue study drug |
| Dermatology/ Skin | Rash non-desquamation - Grade 3 | Hold study drug until resolved to < Grade 1. Decrease dose by 1 dose level |
| Dermatology/ Skin | Rash non-desquamation - Grade 4 | Discontinue study drug |
| Dermatology/ Skin | Rash / desquamation - Grade 3, 4 | Discontinue study drug |
| | Rash / desquamation - Grade 2 | The dose may be modified or discontinued at the investigators discretion. |
| Dermatology/ Skin | Rash Erythema multiforme | Discontinue study drug |
| Endocrine | Elevated or Reduced Thyroid<br>Function Test results without<br>symptoms of hyper- or hypo-<br>thyroidism | Confirm test results and if significant, refer for therapy; Do not alter study drug regimen |


| Common<br>Terminology<br>Criteria (CTCAE)<br>Version 4.0 | Adverse Event | Dose Change for Pomalidomide |
|---|---|---|
| Endocrine | Elevated or Reduced Thyroid<br>Function Test results with<br>symptoms of hyper- or hypo-<br>thyroidism | Hold study drug; Evaluate etiology and refer for appropriate therapy; Restart at the prior dose once symptoms have resolved and thyroid function has been stabilized with medical and/or surgical intervention |
| Neurology | Neuropathy cranial/motor/ sensory - Grade 2 | Hold study drug; Restart at same or 1 dose level lower once event has resolved to < Grade 1 |
| Neurology | Neuropathy cranial/motor/ sensory<br>Grade 3 or recurrence of Grade 2 | Hold study drug until resolved to < Grade 1; Decrease dose by 1 dose level |
| Neurology | Neuropathy cranial/motor/ sensory - Grade 4 | Discontinue study drug |
| Other pomalidomide related toxicity | Grade 3 or Grade 4 | Hold pomalidomide therapy;<br>Decrease dose by 1 dose level and<br>restart when resolved to < Grade 2 |

## 3.4 QUESTIONNAIRES

Patient self-report questionnaires administered in this study are part of the standard NIH chronic consensus recommended criteria for the evaluation of cGvHD in clinical trials.<sup>29</sup> These standardized assessments are designed to evaluate patient quality of life (SF-36, FACT-BMT), functional performance (HAP) and symptoms (Lee symptom scale, symptom intensity scale). The purpose of these evaluations is to assess the potential benefit of the administered therapy as compared to the baseline. These forms have been extensively used, published and validated. These forms are also standard part of many NCI CCR cGvHD protocols (Appendix G). In a recent study median time for persons to complete these forms was 15 minutes (range 8-22 minutes).<sup>73</sup>


## 3.5 STUDY CALENDAR

| Assessments | Screening | BL | | | | | | 3 | | 6 | | 9 | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | mos | | mos | | mos | | |
| | | BL/<br>C1<br>D1 | C1<br>D15<br>(+/-2<br>days) | C2<br>D1<br>(+/-2<br>days) | C2<br>D15<br>(+/-2<br>days) | C3<br>D1<br>(+/-2<br>days) | C3<br>D15<br>(+/-2<br>days) | C4<br>D1<br>(+/-3<br>days) | C5,6<br>D1<br>(+/-2<br>days) | C7<br>D1<br>(+/-3<br>days) | C8,9<br>D1<br>(+/-2<br>days) | C10<br>D1<br>(+/-3<br>days) | C11,<br>12<br>D1<br>(+/-2<br>days) | C12<br>D28<br>(+/-3<br>days) |
| Informed Consent | X | | | | | | | | | | | | <b>.</b> | |
| Randomization | X | | | | | | | | | | | | | |
| Pomalidomide po qd <sup>2</sup> | | X | X | X | X | X | X | X | X | $X^2$ | $X^2$ | $X^2$ | $X^2$ | $X^2$ |
| History and Physical<br>Exam | X | X | X | X | X | X | X | X | X | X | X | X | | X |
| Confirmation of cGvHD <sup>3</sup> | X | | | | | | | | | | | | | |
| Body Photography | | X | | | | | | | | X | | | | |
| cGVHD 3 Month<br>Trajectory (stable vs.<br>progressive) | | X | | | | | | | | | | | | |
| Pulmonary Function<br>Testing | X | | | | | | | X | | X | | X | | X |
| Diagnostic Imaging <sup>4</sup> | X | | | | | | | X | | X | | X | | |
| Pregnancy Test <sup>5</sup> | X | X | X | X | | X | | X | X | X | X | X | X | |
| POMALYST REMS <sup>TM</sup> program <sup>6</sup> | X | X | | X | | X | | X | X | X | X | X | X | X |
| cGvHD Therapies<br>Recording | X | Thro | oughout | the stu | dy | | | | | | | | | |


| Assessments | Screening | BL | | | | | | 3 | | 6 | | 9 | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | mos | | mos | | mos | | |
| | | BL/<br>C1<br>D1 | C1<br>D15<br>(+/-2<br>days) | C2<br>D1<br>(+/-2<br>days) | C2<br>D15<br>(+/-2<br>days) | C3<br>D1<br>(+/-2<br>days) | C3<br>D15<br>(+/-2<br>days) | C4<br>D1<br>(+/-3<br>days) | C5,6<br>D1<br>(+/-2<br>days) | C7<br>D1<br>(+/-3<br>days) | C8,9<br>D1<br>(+/-2<br>days) | C10<br>D1<br>(+/-3<br>days) | C11,<br>12<br>D1<br>(+/-2<br>days) | C12<br>D28<br>(+/-3<br>days) |
| Vital Signs | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Height | X | | | | | | | | | | | | | |
| Weight | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| ЕСНО | X | | | | | | | | | | | | | |
| ECG <sup>7</sup> | X | X | | X | | X | | X | | X | | | | |
| Gynecological Exam | | X <sup>14</sup> | | | | | | | | X | | | | |
| Karnofsky Performance<br>Status | X | | | | | | | X | | X | | X | | |
| CBC w/ differential, platelets <sup>8</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Serum Chemistry <sup>8</sup> | | X | X | X | X | X | X | X | X | X | X | X | X | X |
| CRP, total complement, C3, C4 | | X | | X | | X | | X | | X | | X | | X |
| Urinalysis | X | | | | | | | X | | X | | X | | |
| TSH, free T4 | X | | | | | | | X | | X | | X | | |
| cGvHD Assessment and<br>Response Calculation <sup>9</sup> | X | | | | | | | X | | X | | X | | |
| AE Monitoring | | Throughout the study | | | | | | | | | | | | |
| Concurrent Drugs | X | Thro | Throughout the study | | | | | | | | | | | |


| Assessments | Screening | BL | | | | | | 3<br>mos | | 6 | | 9<br>mos | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | mos | | | | |
| | | BL/<br>C1<br>D1 | C1<br>D15<br>(+/-2<br>days) | C2<br>D1<br>(+/-2<br>days) | C2<br>D15<br>(+/-2<br>days) | C3<br>D1<br>(+/-2<br>days) | C3<br>D15<br>(+/-2<br>days) | C4<br>D1<br>(+/-3<br>days) | C5,6<br>D1<br>(+/-2<br>days) | C7<br>D1<br>(+/-3<br>days) | C8,9<br>D1<br>(+/-2<br>days) | C10<br>D1<br>(+/-3<br>days) | C11,<br>12<br>D1<br>(+/-2<br>days) | C12<br>D28<br>(+/-3<br>days) |
| Skin and Oral Biopsies, saliva collection <sup>10</sup> | | X | | | | | | | | X | | | uaysj | |
| TBNK | | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Blood and urine for Immunologic Studies <sup>11</sup> | | X | | | | | | X | | X | | X | | X |
| Blood for PK Studies <sup>12</sup> | | X | X | X | X | X | X | X | X | X | | | | |
| Study drug<br>dispensation/<br>return/accountability | | | X | X | X | X | X | X | X | X | X | X | X | X |
| Rehabilitation medicine | | X <sup>14</sup> | | | | | | | | X | | | | |
| Occupational therapy<br>Consults | | X <sup>14</sup> | | | | | | X | | X | | X | | |
| Dermatology | | X | | | | | | | | X | | | | |
| Ophthalmology | | X <sup>14</sup> | | | | | | | | X | | | | |
| Schirmer's without anesthesia | | X | | | | | | X | | X | | X | | |
| NIH Advanced<br>Directives form <sup>15</sup> | | X | | | | | | | | | | | | |

<sup>&</sup>lt;sup>1</sup> Clinic visits can occur ± 3 days. All procedures at protocol-driven time points are performed at the NIH Clinical Center, but if circumstances make this impossible, these data points will be collected in collaboration with referring physicians.


<sup>2</sup> Pomalidomide at assigned doses for 6 months; another 6-month course of treatment will be allowed for patients with response (see Section 3.1.1). Only patients who continue therapy beyond 6 months will be required to have clinical monitoring tests during cycles 7 through 12.

- <sup>3</sup> Use NIH diagnostic criteria for cGvHD (<u>Appendix C</u>). In addition, use <u>Appendix D</u> for clinical differentiation of acute versus cGvHD.
- <sup>4</sup> MRI if indicated and chest CT at baseline and if indicated, at response assessments.
- <sup>5</sup> Pregnancy tests for females of childbearing potential must follow pregnancy testing requirements as outlined in the POMALYST REMS<sup>TM</sup> program. A female of childbearing potential (FCBP) is a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).

Pregnancy tests must occur 10–14 days and again within 24 hours prior to initiation of pomalidomide. FCBP with regular or no menstruation must have a pregnancy test weekly for the first 4 weeks and then every 28 days while on therapy (including breaks in therapy); at discontinuation of pomalidomide and at Day 28 post the last dose of pomalidomide. Females with irregular menstruation must have a pregnancy test weekly for the first 4 weeks and then every 14 days while on therapy (including breaks in therapy), at discontinuation of pomalidomide and at Day 14 and Day 28 post the last dose of pomalidomide (see <u>Appendix M</u>).

- <sup>6</sup> All patients must be counseled about pregnancy precautions, risks of fetal exposure and other risks through the POMALYST REMS<sup>TM</sup> program. The counseling must be done on at a minimum of every 28 days and at drug discontinuation. See <u>Appendix M</u>.
- <sup>7</sup> ECG at indicated intervals baseline, at C2D1, C3D1, C4D1, C7D1 and as clinically indicated. Prolongation of QTc > 0.5 s or QTc interval increases from baseline > 0.06 s is considered as a safety concern.
- <sup>8</sup> CBC with differential and platelets, serum chemistries (including sodium, potassium, chloride, CO<sub>2</sub>, calcium, magnesium, phosphorus, blood urea nitrogen [BUN], creatinine, glucose, albumin, total protein, alkaline phosphatase, total bilirubin, AST [SGOT], ALT [SGPT], lactate dehydrogenase [LDH], and uric acid) at least every other week the first 3 months, then monthly until 9 months, then on day 28 of cycle 12. Platelets should be repeated when clinically indicated (e.g., suspected thromboembolic events).
- <sup>9</sup> Includes primary and secondary measurement of response, performance scale, global rating, and Lee Symptom Scale (<u>Appendix G</u> through <u>Appendix K</u>).
- <sup>10</sup>Skin and oral biopsies and saliva collection will be performed before treatment and after 6 months of pomalidomide, with intent to sample as close to the same area as possible (Section **5.1.1**)


<sup>11</sup>Blood for Immunologic studies will be collected (Section **5.1.2**). A larger 100ml blood (12 R&G CPT) plus a 3ml theophylline citrate blood (for TGFb) will be collected only at baseline, at 3 months (beginning of cycle 4) and the 6 months evaluation (at the end of cycle 6)

<sup>12</sup>For determining serum pomalidomide levels, a 3-mL blood sample will be collected 2 hours (± 15 minutes) after initial oral administration and repeated every 2 weeks (20-24 hours after the last oral dose and 2 hours after the dose) until the 3-month evaluation, point then monthly until the 6-month evaluation (Section **5.1.3**). Pre- dosing PK can be done 18-30 hours post last dose of pomalidomide.

<sup>13</sup> Patients who discontinue study drug for any reason will be followed for survival and cGvHD course and therapy for up to 2 years from the start of study drug (see Section **6.1.3**).

<sup>14</sup>Can be done up to two weeks after starting study drug

<sup>15</sup> As indicated in section **10.3**, all subjects will be offered the opportunity to complete an NIH advanced directives form. This should be done preferably at baseline but can be done at any time during the study as long as the capacity to do so is retained. The completion of the form is strongly recommended, but is not required.

Patients may undergo additional subspecialty evaluations by Gynecology, Dermatology, Opthalmology, Dentistry, Physical Medicine and Rehabilitation and Occupational Medicine at any additional time points as indicated clinically or during the off study visit per investigator discretion.

#### 3.6 CRITERIA FOR REMOVAL FROM PROTOCOL THERAPY AND OFF STUDY CRITERIA

Prior to removal from study, effort must be made to have all subjects complete a safety visit approximately 30 days following the last dose of study therapy.

## 3.6.1 Criteria for removal from protocol therapy

- Completion of 6- or 12-month course of protocol therapy (depending on the level of response)
- Progressive cGvHD or malignancy requiring new line of systemic therapy
- Participant requests to be withdrawn from active therapy
- Unacceptable toxicity as defined in Section 3.3
- Dose interruption longer than 35 days
- Positive pregnancy test
- Investigator discretion

The PI is to be notified of all discontinuations from study drug. The reason for dose modification/discontinuation should be recorded in the CRF and in the patient's medical records.

## 3.6.2 Off-Study Criteria

- Completed 2-year follow-up period
- Subject withdrawal from follow-up period
- Patient lost for follow-up
- Death
- PI decision to end this study

## 3.6.3 Off Protocol Therapy and OffStudy Procedure

Authorized staff must notify Central Registration Office (CRO) when a subject is taken off-protocol therapy and when a subject is taken off study. A Participant Status Update Form from the web site (<a href="http://home.ccr.cancer.gov/intra/eligibility/welcome.htm">http://home.ccr.cancer.gov/intra/eligibility/welcome.htm</a>) main page must be completed and sent via encrypted email to: NCI Central Registration Office (HOIS) <a href="mailto:ncicentralregistration-l@mail.nih.gov">ncicentralregistration-l@mail.nih.gov</a>.

### 4 CONCOMITANT MEDICATIONS/MEASURES

All medications (prescription and non-prescription), treatments and therapies taken throughout the study must be recorded on the appropriate page of the CRF. Patients will be advised to contact the study team before starting any new medications.

### 4.1 CONCOMITANT CORTICOSTEROID THERAPY AND TAPERING GUIDELINE

During the study, persons may remain on corticosteroids with intent to taper it. A steroid taper will be allowed to begin earliest at 4-6 weeks after starting on protocol, with a 10% (of starting


dose) decrease per week. The study allows maximum two total pulses of steroids with subsequent rapid taper, one at the beginning of pomalidomide therapy in case of GvHD flares associated with the study drug initiation and/or another one later for any flares or worsening of cGvHD symptoms during steroid or other immunosuppression taper. Typical corticosteroid pulse is defined as up to 2 mg/kg/day prednisone or equivalent tapered to the pre-pulse baseline within 3 weeks. Steroid pulses require the PI's approval. If the patient has a GVHD flare and no other reasons to hold the drug for an AE the patient would continue pomalidomide administration concomitantly with steroid pulse. Administration steroid pulses will be carefully recorded in the protocol case report forms.

### 4.2 OTHER TREATMENTS FOR CGVHD

Patients who are taking concomitant systemic agents for control of cGvHD, such as calcineurin inhibitors (e.g., tacrolimus or cyclosporine) or other immunosuppressants (e.g., mycophenolate or sirolimus) must be on a stable dose in the preceding 4 weeks with an intent to stop if possible after corticosteroids are at stable or supplementation doses (maximum 7.5 mg prednisone/day) or discontinued. Patient should not receive any investigational drugs or initiate any systemic therapy for cGvHD once started on pomalidomide. Patient should not be undergoing extracorporeal photopheresis (ECP) concomitantly with study drug, and if they had ECP in the past, a minimum of 4 weeks should have passed since its discontinuation.

#### 4.3 VENOUS THROMBOEMBOLISM PROPHYLAXIS

Pomalidomide may increase the risk of thrombotic events in persons who are at high risk or with a history of thrombosis, in particular when combined with other drugs known to cause thrombosis. When pomalidomide is combined with other agents such as steroids (e.g., dexamethasone, prednisone), anthracyclines (doxorubicin) and erythropoietin, the risk of thrombosis may be increased. All persons if receiving study treatment in addition to any of these other agents must also agree to take venous thromboembolism (e.g., at minimum aspirin 325 mg/day) or some other form of prophylaxis as deemed appropriate by the PI, such as low molecular weight or unfractionated heparin.<sup>74</sup> Patients should continue to receive anti-thrombotic therapy for the duration of pomalidomide therapy and 5 days after pomalidomide is discontinued.

Because of the increased risk of venous thromboembolism in patients taking pomalidomide and dexamethasone, combined oral contraceptive pills are not recommended. If a patient is currently using combined oral contraception the patient should switch to another one of the effective methods listed above. The risk of venous thromboembolism continues for 4–6 weeks after discontinuing combined oral contraception. The efficacy of contraceptive steroids may be reduced during co-treatment with dexamethasone.

#### 4.4 OTHER ALLOWED CONCOMITANT THERAPY

Ancillary therapy and supportive care considered necessary for the patient's wellbeing may be administered at the discretion of the PI and will follow the NIH Blood and Marrow Transplant Consortium guidelines for supportive care: <a href="http://intranet.cc.nih.gov/bmt/clinicalcare/guidelines.shtml">http://intranet.cc.nih.gov/bmt/clinicalcare/guidelines.shtml</a>. Any ancillary or supportive care which may have some effect on efficacy analysis will be carefully recorded in the CRF. Patients are allowed to take topical steroids at a maximum of 1% hydrocortisone concentration potency equivalence.


#### 4.5 PROHIBITED CONCOMITANT THERAPY

Radiation therapy, cancer chemotherapy, biologic or immunotherapy is prohibited during participation in this study. Concomitant use of other investigational agents is not permitted while persons are receiving study drug.

## 5 BIOSPECIMEN COLLECTION

#### 5.1 CORRELATIVE STUDIES FOR RESEARCH

Note: All samples will be sent for storage until analysis as detailed in Section 5.2 under appropriate storage conditions.

## 5.1.1 Skin Biopsy and Oral Biopsy

Skin and oral research biopsies will be performed before treatment and after 6 months of pomalidomide treatment (with intent to sample as close to the same area as possible) for assessment of sclerotic or lichen-planus like disease by H&E and pathologist evaluation. Immunohistochemistry methods will be applied to look for myofibroblast markers and pSMAD in the sclerotic skin, for T-cell infiltrates, and IFN-induced factors in the oral mucosa and erythematous skin. The advantage of histology is the greater amount of information on cell populations and functional changes in situ of the disease. These biopsies will be obtained by one of the study investigators and processed, stored and analyzed. A biopsy sample will be also sent to the NCI pathology laboratory. Patients will have an option to decline such research biopsy and this will not be considered as protocol deviation. Biopsy samples collected on the 04-C-0281 cGvHD natural history study can be also used for these studies if obtained in the timeframe as part of the screening evaluations for this study.

## 5.1.2 Immunologic Analyses Using Plasma and PBMCs

- 1. <u>Blood</u>: Blood will be collected, and PBMC and plasma will be cryopreserved for later batch analyses of markers relevant to cGvHD activity. Plasma will be collected with theophylline-citrate anticoagulant (to prevent platelet breakdown) for assessment of TGFb and PDGF, which may be relevant to fibrosis. Heparinized plasma will be assayed for markers of cGvHD activity (including but not limited to BAFF, and IFN-induced chemokines). PBMC will be cryopreserved for subsequent flow cytometry of cell populations and sorting of monocytes for transcriptional analysis of genes upregulated in active cGvHD. The primary collection of blood for these analyses of pomalidomide effect on cGvHD will be at baseline and at 3 and 6 month evaluation time point. At these three timepoints one theophylline citrate plasma tube (for TGFb) and 12 red and green topped heparin CPT tubes (total of 100 cc) will be collected; a final collection will be done on patients continuing treatment until 12 months.
- 2. <u>Plasma</u> will be assayed for BAFF, IFN-induced chemokines and MCP-1. Separate collection of theophylline-citrate blood (different anticoagulant to prevent platelet breakdown) will be performed for assessment of TGFb and PDGF.
- 3. Monocyte transcriptome: Monocytes will be sorted from PBMC for Nanostring evaluation of the monocyte transcriptome. This would be done on cryopreserved cells at the end of the study. Monocytes circulate throughout the body, are responsive to a variety of cytokines


in tissues affected by cGvHD and maybe therefore serve as a reporter for changes in cGvHD-affected tissues.

4. Lymphocyte populations. Changes in circulating populations of lymphocytes will be assessed by flow cytometry on whole blood to determine changes in CD3, CD4, CD8, B and NK populations. At baseline, at the start of each cycle up to the 3 month time point and at 6 and 12 months, one 3ml lavender (EDTA) tube will be drawn and lymphophenotyping will be performed using Clinical center's CLIA certified Immunophenotyping panel and reported in the CRIS. Further research assessments of the percentages of regulatory T cells, of naïve, memory and effector T cells and of B cell transitional, naïve and memory populations will be done in the ETIB Preclinical Core (Fran Hakim) on the baseline and at 3 month evaluation time points until 12 months post enrollment. Active cGvHD has been associated with decreases in Treg populations, reduced thymopoiesis (fewer naïve T cells) and increases in CD21- transitional B cell populations. Urine will be collected at 3 month intervals for assessment of biomarkers in urine as compared with blood.

The assays indicated are designed to assess the alterations in skin, oral mucosa and in circulating lymphocytes and plasma that may result from pomalidomide. If there is a decline in TGFb production or response, then this may be evident in TGFb levels in the plasma and in degree of fibrosis (by pathologist evaluation) and extent of pSMAD2/3 in sclerotic skin. If there is an increase in Th1 cells or a shift in Treg populations, this may be reflected in circulating T cell populations, plasma cytokines and tissue infiltrates.

#### 5.1.3 Measurement of Pomalidomide Serum Levels

The objective of measuring pomalidomide serum levels is for the documentation of systemic absorption. A 6-mL blood sample will be collected 2 hours (+/- 20 minutes, exact time elapsed post-dosing will be recorded on PK sheets) after initial oral administration and repeated peak and trough every 2 weeks (20-28 hours after the last oral dose and 2 hours post-dose) until the 3-month evaluation, then monthly until the 6-month evaluation. Pre- dosing PK can be done 18-30 hours post last dose of pomalidomide. Actual dosing dates and times will be recorded. Detailed instruction for sample collection, processing, storage, and handling can be found in Appendix B. These sample collections will occur at the protocol scheduled evaluation visits at the NIH Clinical Center.

The determination of pomalidomide concentrations in plasma samples, as well as the pharmacokinetic data analysis, will be performed by the Clinical Pharmacology Program. Samples will be analyzed using a validated LC-MS/MS method.

## 5.2 SAMPLE STORAGE, TRACKING AND DISPOSITION

Samples will be ordered in CRIS and tracked through a Clinical Trial Data Management system. Should a CRIS screen not be available, the CRIS downtime procedures will be followed. Samples will not be sent outside NIH without appropriate approvals and/or agreements, if required.


### 5.2.1 Sample Procedures

Blood and tissue samples, collected for the purpose of research under IRB-approved protocols of the Experimental Transplantation and Immunology Branch (ETIB)/Immune Deficiency Cellular Therapy Program (IDCTP) will be stored and may be archived by the Biospecimen Processing Core (BPC), with the exception of blood samples for pomalidomide analysis, which will be stored separately by the Clinical Pharmacology Program (CPP) until analysis. These will be barcoded, with data entered and stored in the Labmatrix utilized by the BPC. This is a secure program, with access to Labmatrix limited to defined Figg lab personnel, who are issued individual user accounts. Installation of Labmatrix is limited to computers specified by Dr. Figg. These computers all have a password restricted login screen.

Labmatrix creates a unique barcode ID for every sample and sample box, which cannot be traced back to patients without Labmatrix access. The data recorded for each sample includes the patient ID, name, trial name/protocol number, time drawn, cycle time point, dose, material type, as well as box and freezer location. Patient demographics associated with the clinical center patient number are provided in the system. For each sample, there are notes associated with the processing method (delay in sample processing, storage conditions on the ward, etc.).

Barcoded samples are stored in locked freezers at -20 or -80°C (sera and plasma) or under liquid nitrogen (cells), or as otherwise applicable according to stability requirements. These freezers are located onsite in the BPC and offsite at NCI Frederick Central Repository Services in Frederick, MD. Visitors to the laboratory are required to be accompanied by laboratory staff at all times.

Access to stored clinical samples is restricted. Samples will be stored until requested by a researcher named on the protocol. All requests are monitored and tracked in Labmatrix. All researchers are required to sign a form stating that the samples are only to be used for research purposes associated with this trial (as per the IRB approved protocol) and that any unused samples must be returned to the BPC. It is the responsibility of the NCI Principal Investigator to ensure that the samples requested are being used in a manner consistent with IRB approval.

## 5.2.1.1 Protocol Completion/Sample Destruction

Following completion of this study, samples will remain in storage as detailed above. Access to these samples will only be granted following IRB approval of an additional protocol, granting the rights to use the material.

If, at any time, a patient withdraws from the study and does not wish for their existing samples to be utilized, the individual must provide a written request. Following receipt of this request, the samples will be destroyed or returned to the participant, if so requested. The PI will record any loss or unanticipated destruction of samples as a deviation. Reporting will be per the requirements of section 7.27.2.

#### 6 DATA COLLECTION AND EVALUATION

#### **6.1 DATA COLLECTION**

The PI will be responsible for overseeing entry of data into a 21 CFR Part 11-compliant data capture system provided by the NCI CCR and ensuring data accuracy, consistency and timeliness. The principal investigator, associate investigators/research nurses and/or a contracted


data manager will assist with the data management efforts. Primary and final analyzed data will have identifiers so that research data can be attributed to an individual human subject participant.

All adverse events, including clinically significant abnormal findings on laboratory evaluations, regardless of severity, will be followed until return to baseline or stabilization of event. Patients will be followed for adverse events for a minimum of 30 days after the last administration of investigational agent/intervention and have an attribution of at least possibly related to the agent/intervention should be recorded and reported as per sections 7.2, 7.3 and 7.4 or until removal from study treatment, whichever comes first.

An abnormal laboratory value will be considered an AE if the laboratory abnormality is characterized by any of the following:

- Results in discontinuation from the study
- Is associated with clinical signs or symptoms
- Requires treatment or any other therapeutic intervention
- Is associated with death or another serious adverse event, including hospitalization.
- Is judged by the Investigator to be of significant clinical impact
- If any abnormal laboratory result is considered clinically significant, the investigator will provide details about the action taken with respect to the test drug and about the patient's outcome.

**End of study procedures:** Data will be stored according to HHS, FDA regulations, and NIH Intramural Records Retention Schedule as applicable.

Loss or destruction of data: Should we become aware that a major breech in our plan to protect subject confidentiality and trial data has occurred, the IRB will be notified.

## 6.1.1 Eligibility Checklist

The eligibility checklist is to be completed at study entry and forwarded to protocol research nurse who will forward the checklist to the Central Registration Office.

### 6.1.2 Protocol Deviations and Non-Compliance

Any protocol non-compliance or deviations should be directly reported to the PI and to the NIH IRB per Section 7.2.

## 6.1.3 Follow-up

All persons will be followed for SAEs for 30 days after last dose of pomalidomide. Patients who discontinue therapy for any reason will be invited for a follow up visit at 3 months after last dose, then followed up by a phone call to the patient and/or the primary physician's office at 12 and 24 months after starting the first dose of pomalidomide. The phone call will focus on a) survival status and cause of death if pertinent, b) ongoing systemic treatment for cGvHD and date of discontinuation, c) primary malignancy progression, d) any second primary malignancy, e) return to work part-time or full-time. Primary and contributing causes of death are to be recorded in the CRF and the patient's medical record.


#### **6.2** RESPONSE CRITERIA

## 6.2.1 Definitions

Evaluable for efficacy: Patients who complete 6 months of therapy will be evaluable for the secondary endpoint of efficacy assessment. Patients who progress earlier will be also included in the analysis of efficacy.

### 6.2.2 Efficacy Analysis

The primary evaluation point is overall response at 6 months using the NIH cGvHD response criteria measures.<sup>29</sup> The overall response score will be assessed as CR, PR, SD or PD as per NIH guidelines. The organ-specific and other subcomponents of the overall response score will be analyzed individually and absolute values recorded.

Up to 2 corticosteroid pulses will be allowed, one for initial flares and one for late flares as described in Section 4.1.

Response will be assessed every 3 months from the start of pomalidomide. To ensure comparability, baseline and on-study methods for response assessment will be performed using identical grading, scale or techniques. The Chronic GVHD Assessment (Clinician) Form will be completed at each 3-month evaluation visit [Appendix G]. Included in that form are both organ-specific primary measurements and clinician-assessed secondary measurements. The response of each affected organ will be evaluated and an overall response (CR, PR, stable disease) will be determined.

## 6.2.2.1 Response Criteria

Efficacy will be assessed using NIH consensus criteria measuring for therapeutic response in clinical trials for cGvHD<sup>29</sup>:

- **CR** is defined as complete resolution in all of signs and symptoms at all affected organs or tissues.
- **PR** is defined as improvement in ≥ 1 organ or tissue with no progression in any other affected organ or tissue. The calculations for PR and progressive disease (PD) are provided in Appendix H and Appendix I.
- **Response** < **PR** is defined as change towards improvement from the pre-treatment baseline but not meeting the criteria for CR or PR.
- **Stable Disease** is defined as no change in cGvHD, SD will be considered as response in patients with documented cGvHD progression over preceding 3 months.
- **Flare** is defined as exacerbation of cGvHD manifestations during withdrawal of immunosuppressive therapy which do not exceed those at the beginning of the trial and improves after reinstatement of previous treatment.
- **Progressive disease** is defined as failure of therapy to control cGvHD. The calculations for progressive disease (PD) are provided in <u>Appendix I</u>. Assessment by Organ-Specific Criteria. Patients who progress prior to 6 months evaluation will be also evaluable for the primary efficacy endpoint.
- **Mixed response** (improvement in some organs but worsening in others) will be categorized as progressive disease.


As outlined in Section 3.5, type of involved organ, location and its measurements will be recorded at scheduled evaluations and reported on the appropriate CRF, equal to "Chronic GVHD Assessment (Clinician) Form," (Appendix G). All other measurements not being included in primary assessment but clinically related to cGvHD (e.g., change of pigmentation) will be reported in the source documents.

**Skin and skin appendages:** Skin assessments include 4 anatomic level of skin involvement:

- (1) erythematous rash (epidermal),
- (2) movable sclerosis (dermal),
- (3) non-moveable sclerosis, hidebound skin, or involvement of subcutaneous tissue and fascia (subcutaneous) and
- (4) ulceration (full thickness loss of epidermal tissue).

The first 3 measurements should be taken separately and recorded in metric notation using a body surface area (BSA). A cutaneous assessment worksheet for recording the BSA is provided (Appendix J). The size of ulcer should be measured the longest diameter (LD) of the largest ulcer.

**Eyes:** The primary measurement of lacrimal gland function in cGvHD is using the Schirmer's test. The test should be performed without anesthesia for both eyes (OU) unless physically inapplicable. The measurement of each eye and the average of measurements will be recorded in the CRF.

**Mouth:** Mouth assessments include:

(1) mucosal erythema by 0-3 grading based on the color intensity, (2) lichen-type hyperkeratosis by 0-3 grading based on the percentage of oral surface area,(3 ulceration by 0-6 based on percentage of oral surface area, and (4) mucoceles by 0-3 grading based on its total number of presence.

**Hematopoietic:** The measurements of hematopoietic response include:

- (1) platelet count,
- (2) eosinophil count and percentage.

White blood cell (WBC) count will be recorded on the Assessment Form but will not be used for response assessment.

**Gastrointestinal tract:** Gastrointestinal (GI) symptoms are graded through interview by the investigator according to 0-3 severity scales.

**Liver:** Involvement of liver is graded according to the levels of bilirubin and liver enzymes (AST and ALT).

**Lung:** The forced expiratory volume in the first second (FEV1) and single breath diffusion lung capacity for carbon monoxide (DLCO) is included as components for the lung function score (LFS). LFS is computed by the extent of FEV1 and DLCO compromise (>80% = 1, 70 - 79% = 2, 60 - 69% = 3, 50 - 59% = 4, 40 - 49% = 5, <40% = 6). Scores for FEV1 and DLCO are added and the sum reduced to an overall category according to following table (Table 5). Absolute values of both FEV1 and DLCO should be recorded in the CRF.

**Table 5. Categories of the Lung Function Score** 


| Category | Lung Function | Lung Function Score |
|----------|-------------------|---------------------|
| I | Normal | 2 |
| II | Mild decrease | 3 – 5 |
| III | Moderate decrease | 6 – 9 |
| IV | Severe decrease | 10 – 12 |

**Global chronic GVHD Rating:** The overall clinical impression of patient's cGvHD will be recorded on a 4-point (0-3) scale on the Chronic GVHD Assessment (Clinician) Form.

Chronic GVHD Improvement Scale: The overall changes of patient's cGvHD symptoms <u>during</u> <u>previous 3 months</u> will be recorded on a 7-point (-3 to +3) scale on the Chronic GVHD Assessment (Clinician) Form.

**Chronic GVHD Symptom Severity Scale:** The overall severity of patient's cGvHD symptoms will be recorded on an 11-point (0-10) numeric scale on the Chronic GVHD Assessment (Clinician) Form.

**Karnofsky Performance Scale:** The Karnofsky Performance Scale will be only recorded on the Chronic GVHD Assessment (Clinician) Form but <u>not</u> used as a measure of response.

**Lee symptom scale** was developed as a 30-item symptom scale with 7 subscales to capture the cGvHD-specific symptom burden (<u>Appendix K</u>). This symptom scale showed to correlate with persons' self-assessed mild, moderate, and severe cGvHD manifestations in cross-sectional validation analysis. "Lee total score" will be calculated per Lee et al. <sup>75</sup> Longitudinal assessments showed that changes in overall health status correlated best with changes in quality of life as measured by the SF-36 and FACT-BMT. We will not use "Lee symptom scale" as a measure of pomalidomide efficacy but as supplemental information on the quality of life.

**NIH organ 0-3 scoring** (Appendix E) will be also collected at the evaluation endpoints.<sup>22</sup> Although not initially developed for response assessments, the evidence is emerging in some domains (skin, eyes) about potential use of this scale as a simple and valid assessment of cGvHD change over time.

## 6.2.2.2 Summary of Response Measures

- i. Primary response measures
  - 1. Skin (BSA), erythema, moveable, non-moveable
  - 2. Eyes (Schirmer)
  - 3. Mouth (modified OMRS)
  - 4. Liver (bilirubin, AST, ALT)
  - 5. GI tract (GI response scale)


- 6. Lung (FEV, DLCO, LFS)
- 7. Clinician assessment scale (3-point, 7-point change, 11-point global)
- 8. ROM visual Carpenter scale (1-7 and 1-4)
- 9. NIH organ scoring
- ii. Secondary assessments
  - 1. Platelet count, CRP, C3, C4, albumen
  - 2. 2 and 6 minute walk time
  - 3. Grip strength
  - 4. Lee symptom scale
  - 5. HAP, SF-36, Karnofsky
  - 6. MRI (if positive baseline)
  - 7. Disabilities of the Arm Hand and Shoulder (DASH)
- 6.2.2.3 Other endpoints to be recorded at the evaluation time points: Need for secondary systemic therapy for GvHD, malignancy progression, discontinuation of immune suppression, steroid doses, other immunosuppressive drug doses, intensity of immunosuppression, NIH global severity (<u>Appendix P</u>), survival, progression-free/malignancy-free survival, disability-free survival.

### **6.3** TOXICITY CRITERIA

The following adverse event management guidelines are intended to ensure the safety of each patient while on the study. The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for AE reporting. All appropriate treatment areas should have access to a copy of the CTCAE version 4.0. A copy of the CTCAE version 4.0 can be downloaded from the CTEP web site: (http://ctep.cancer.gov/protocolDevelopment/electronic\_applications/ctc.htm#ctc\_40).

## 7 NIH REPORTING REQUIREMENTS/DATA AND SAFETY MONITORING PLAN

#### 7.1 **DEFINITIONS**

Please refer to definitions provided in Policy 801: Reporting Research Events found at: <a href="https://irbo.nih.gov/confluence/pages/viewpage.action?pageId=36241835#Policies&Guidance-800Series-ComplianceandResearchEventReportingRequirements">https://irbo.nih.gov/confluence/pages/viewpage.action?pageId=36241835#Policies&Guidance-800Series-ComplianceandResearchEventReportingRequirements</a>.


#### 7.2 OHSRP OFFICE OF COMPLIANCE AND TRAINING / IRB REPORTING

### 7.2.1 Expedited Reporting

Please refer to the reporting requirements in Policy 801: Reporting Research Events and Policy 802 Non-Compliance Human Subjects Research found at:

https://irbo.nih.gov/confluence/pages/viewpage.action?pageId=36241835#Policies&Guidance-800Series-ComplianceandResearchEventReportingRequirements.. Note: Only IND Safety Reports that meet the definition of an unanticipated problem will need to be reported per these policies.

## 7.2.2 IRB Requirements for PI Reporting at Continuing Review

Please refer to the reporting requirements in Policy 801: Reporting Research Events found at: <a href="https://irbo.nih.gov/confluence/pages/viewpage.action?pageId=36241835#Policies&Guidance-800Series-ComplianceandResearchEventReportingRequirements">https://irbo.nih.gov/confluence/pages/viewpage.action?pageId=36241835#Policies&Guidance-800Series-ComplianceandResearchEventReportingRequirements</a>.

## 7.3 NCI CLINICAL DIRECTOR REPORTING

Problems expeditiously reviewed by the OHSRP in the NIH eIRB system will also be reported to the NCI Clinical Director/designee; therefore, a separate submission for these reports is not necessary.

In addition to those reports, all deaths that occur within 30 days after receiving a research intervention should be reported via email unless they are due to progressive disease.

To report these deaths, please send an email describing the circumstances of the death to NCICCRQA@mail.nih.gov within one business day of learning of the death.

### 7.4 NIH REQUIRED DATA AND SAFETY MONITORING PLAN

Serious adverse events potentially attributable to the study medication or procedures will be reported to IRB. If trends are noted and/or risks warrant it, accrual will be interrupted and/or the protocol and/or consent document will be amended accordingly.

## 7.4.1 Principal Investigator/Research Team

The clinical research team will meet on a regular weekly basis when participants are being actively treated on the trial to discuss each participant. Decisions about dose level enrollment and dose escalation if applicable will be made based on the toxicity data from prior participants.

All data will be collected in a timely manner and reviewed by the principal investigator or a lead associate investigator. Events meeting requirements for expedited reporting as described in section 7.2.1 will be submitted within the appropriate timelines.

The principal investigator will review adverse event and response data on each participant to ensure safety and data accuracy. The principal investigator will personally conduct or supervise the investigation and provide appropriate delegation of responsibilities to other members of the research staff.


#### 8 SPONSOR PROTOCOL/SAFETY REPORTING

#### 8.1 **DEFINITIONS**

#### 8.1.1 Adverse Event

Any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An adverse event (AE) can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product (ICH E6 (R2))

## 8.1.2 Serious Adverse Event (SAE)

An adverse event or suspected adverse reaction is considered serious if in the view of the investigator or the sponsor, it results in any of the following:

- Death,
- A life-threatening adverse event (see section **8.1.3**)
- Inpatient hospitalization or prolongation of existing hospitalization
  - A hospitalization/admission that is pre-planned (i.e., elective or scheduled surgery arranged prior to the start of the study), a planned hospitalization for pre-existing condition, or a procedure required by the protocol, without a serious deterioration in health, is not considered a serious adverse event.
  - A hospitalization/admission that is solely driven by non-medical reasons (e.g., hospitalization for patient or subject convenience) is not considered a serious adverse event.
  - Emergency room visits or stays in observation units that do not result in admission to the hospital would not be considered a serious adverse event. The reason for seeking medical care should be evaluated for meeting one of the other serious criteria.
- Persistent or significant incapacity or substantial disruption of the ability to conduct normal life functions
- A congenital anomaly/birth defect
- Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered a serious adverse drug experience when, based upon appropriate medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.

### 8.1.3 Life-threatening

An adverse event or suspected adverse reaction is considered "life-threatening" if, in the view of either the investigator or sponsor, its occurrence places the patient or subject at immediate risk of death. It does not include an adverse event or suspected adverse reaction that, had it occurred in a more severe form, might have caused death. (21CFR312.32)


### 8.1.4 Severity

The severity of each Adverse Event will be assessed utilizing the CTCAE version 4.0.

## 8.1.5 Relationship to Study Product

All AEs will have their relationship to study product assessed using the terms: related or not related.

- <u>Related</u> There is a reasonable possibility that the study product caused the adverse event. Reasonable possibility means that there is evidence to suggest a causal relationship between the study product and the adverse event.
- Not Related There is not a reasonable possibility that the administration of the study product caused the event.

#### 8.2 ASSESSMENT OF SAFETY EVENTS

AE information collected will include event description, date of onset, assessment of severity and relationship to study product and alternate etiology (if not related to study product), date of resolution of the event, seriousness and outcome. The assessment of severity and relationship to the study product will be done only by those with the training and authority to make a diagnosis and listed on the Form FDA 1572 as the site principal investigator or sub-investigator. AEs occurring during the collection and reporting period will be documented appropriately regardless of relationship. AEs will be followed through resolution.

#### SAEs will be:

- Assessed for severity and relationship to study product and alternate etiology (if not related to study product) by a licensed study physician listed on the Form FDA 1572 as the site principal investigator or sub-investigator.
- Recorded on the appropriate SAE report form, the medical record and captured in the clinical database.
- Followed through resolution by a licensed study physician listed on the Form FDA 1572 as the site principal investigator or sub-investigator.

For timeframe of recording adverse events, please refer to section **** All serious adverse events recorded from the time of first investigational product administration must be reported to the sponsor.

#### 8.3 REPORTING OF SERIOUS ADVERSE EVENTS

Any AE that meets protocol-defined serious criteria or meets the definition of Adverse Event of Special Interest that require expedited reporting must be submitted immediately (within 24 hours of awareness) to OSRO Safety using the CCR SAE report form.

All SAE reporting must include the elements described in section 8.2.

SAE reports will be submitted to the Center for Cancer Research (CCR) at: <a href="https://osroosafety@mail.nih.gov">Osroosafety@mail.nih.gov</a> and to the CCR PI and study coordinator. CCR SAE report form


and instructions can be found at: <a href="https://nih.sharepoint.com/:u:/r/sites/NCI-CCR-OCD-Communications/SitePages/Forms-and-Instructions.aspx?csf=1&web=1&e=uWBXtI">https://nih.sharepoint.com/:u:/r/sites/NCI-CCR-OCD-Communications/SitePages/Forms-and-Instructions.aspx?csf=1&web=1&e=uWBXtI</a>

Following the assessment of the SAE by OSRO, other supporting documentation of the event may be requested by the OSRO Safety and should be provided as soon as possible.

#### 8.4 SAFETY REPORTING CRITERIA TO THE PHARMACEUTICAL COLLABORATORS

Reporting will be per the collaborative agreement.

#### 8.5 REPORTING PREGNANCY

All required pregnancy reports/follow-up to OSRO will be submitted to: <a href="https://nih.gov">OSROSafety@mail.nih.gov</a> and to the CCR PI and study coordinator. Forms and instructions can be found here: <a href="https://nih.sharepoint.com/:u:/r/sites/NCI-CCR-OCD-Communications/SitePages/Forms-and-Instructions.aspx?csf=1&web=1&e=uWBXtI">https://nih.sharepoint.com/:u:/r/sites/NCI-CCR-OCD-Communications/SitePages/Forms-and-Instructions.aspx?csf=1&web=1&e=uWBXtI</a>

## 8.5.1 Maternal exposure

If a participant becomes pregnant during the course of the study, the study treatment should be discontinued immediately, and the pregnancy reported to the Sponsor no later than 24 hours of when the Investigator becomes aware of it. The Investigator should notify the Sponsor no later than 24 hours of when the outcome of the Pregnancy becomes known.

Pregnancy itself is not regarded as an SAE. However, congenital abnormalities or birth defects and spontaneous miscarriages that meet serious criteria (section **8.1.2**) should be reported as SAEs.

The outcome of all pregnancies occurring from the first dose of study therapy until 28 days after the last dose of study therapy should be followed up and documented.

## 8.5.2 Paternal exposure

Male participants should refrain from fathering a child or donating sperm during the study and for 28 days after the last dose of Pomalidomide.

Pregnancy of the participant's partner is not considered to be an AE. However, the outcome of all pregnancies occurring from the date of the first dose until 28 days after the last dose should, if possible, be followed up and documented. Pregnant partners may be offered the opportunity to participate in an institutional pregnancy registry protocol (e.g., the NIH IRP pregnancy registry study) to provide data about the outcome of the pregnancy for safety reporting purposes.

## 8.6 REGULATORY REPORTING FOR STUDIES CONDUCTED UNDER CCR-SPONSORED IND

Following notification from the investigator, CCR, the IND sponsor, will report any suspected adverse reaction that is both serious and unexpected. CCR will report an AE as a suspected adverse reaction only if there is evidence to suggest a causal relationship between the study product and the adverse event. CCR will notify FDA and all participating investigators (i.e., all investigators to whom the sponsor is providing drug under its INDs or under any investigator's IND) in an IND safety report of potential serious risks from clinical trials or any other source, as soon as possible, in accordance to 21 CFR Part 312.32.

All serious events will be reported to the FDA at least annually in a summary format.


#### 8.7 SPONSOR PROTOCOL DEVIATION REPORTING

A Protocol Deviation is defined as any non-compliance with the clinical trial Protocol, Manual of Operational Procedures (MOP) and other Sponsor approved study related documents, GCP, or protocol-specific procedural requirements on the part of the participant, the Investigator, or the study site staff inclusive of site personnel performing procedures or providing services in support of the clinical trial.

It is the responsibility of the study Staff to document any protocol deviation identified by the Staff or the site Monitor in the CCR Protocol Deviation Tracking System (PDTS) online application. The entries into the PDTS online application should be timely, complete, and maintained per CCR PDTS user requirements.

In addition, any deviation to the protocol should be documented in the participant's source records and reported to the reviewing IRB per their guidelines. OSRO required protocol deviation reporting is consistent with E6(R2) GCP: Integrated Addendum to ICH E6(R1): 4.5 Compliance with Protocol; 5.18.3 (a), and 5.20 Noncompliance; and ICH E3 16.2.2 Protocol deviations.

### 9 CLINICAL MONITORING

As a sponsor for clinical trials, FDA regulations require the CCR to maintain a monitoring program. The CCR's program allows for confirmation of: study data, specifically data that could affect the interpretation of primary and secondary study endpoints; adherence to the protocol, regulations, ICH E6, and SOPs; and human subjects protection. This is done through independent verification of study data with source documentation focusing on:

- Informed consent process
- Eligibility confirmation
- Drug administration and accountability
- Adverse events monitoring
- Response assessment.

The monitoring program also extends to multi-site research when the CCR is the coordinating center.

This trial will be monitored by personnel employed by a CCR contractor. Monitors are qualified by training and experience to monitor the progress of clinical trials. Personnel monitoring this study will not be affiliated in any way with the trial conduct.

### 10 STATISTICAL CONSIDERATIONS

It is known from prior trials that the pomalidomide MTD is about 3 mg/d in persons with bone marrow disorders receiving therapies for cancer. Due to high frequency of pomalidomide dose de-escalation observed in preliminary cGvHD experiences when given at 3 mg/d, this study will explore clinical toxicity of gradual escalation doses below 3.0 mg.

The primary objective of this study is to determine if patients with cGVHD will experience an acceptable level of clinical response when treated with either a constant low dose of pomalidomide (0.5 mg/day) for six months or a strategy of increasing dose of pomalidomide from 0.5 mg/d up through each individual patients' maximum tolerated dose, with escalations by


0.5 mg/d every 2 weeks to a maximum of 2.0 mg/d. The study will thus randomize patients between fixed low dose and escalating dose to tolerance, and will be considered a randomized phase II trial with a selection design component.

In each of the two arms, the trial will be conducted using a single stage design. With 16 patients on each arm, an exact binomial test would have 90% power to detect a difference between a 5% response rate and a 30% response rate using a 0.10 one-sided significance level and an exact binomial test. In addition, after the trial has ended, the 80% and 95% confidence limits will be determined for each arm about the observed response proportion in order to aid in interpretation of the results. If there are 3 or more responses in 16 patients, this would be sufficient to rule out a 5% response rate and demonstrate consistency with 30% or better response rates.

At the conclusion of the study, if both arms are able to accrue to the full 16 patients, the arm with the greater number of responses will be selected for further investigation subsequently. That is, if the fixed, low-dose arm, or the increasing dose level arm, has the greater number of responses, then that arm would be studied further. In the event of a tie, the lower dose arm would likely be preferred. As an example, if the true probabilities of response on the two arms were 0.10 and 0.30, then the probability of correctly selecting the superior arm would be 93%, and if the true probabilities on the two arms were 0.15 and 0.30, the probability of correct selection would be 84%.

As an early stopping rule for futility, if after 7 patients have enrolled on either arm, 0 have responded, then no further patients will be accrued to that arm as soon as this can be determined. In practice, this means that patients may continue to be accrued beyond 7 in an arm, but no more patients would be registered and treated on that arm once the first 7 were evaluated and no PRs or CRs were identified in those first 7.

To protect patient safety, an early stopping rule will be implemented as follows. For patients treated on either arm, if 2 patients in the first 6, or 33% of the patients at any time experience a DLT at a given dose level, no further patients will be treated at that given level on the trial. Furthermore, when more than 6 patients have received a given dose level, if at any time 33% or more patients experience a DLT when treated at that dose level, then no further patients will be treated at that dose level. Thus, as an example, should there be 2 patients with a DLT in the first 6 who are able to receive 2.0 mg/day on the dose escalating arm, then subsequent patients treated on that arm will not be escalated beyond 1.5 mg/day.

With two arms, each of which has a maximal accrual of 16 patients, up to 32 evaluable patients will be randomized. In order to allow for a very small number of patients who are not able to be evaluated at all for response, the accrual ceiling will be set at 35.

#### 11 COLLABORATIVE AGREEMENTS

## 11.1 COOPERATIVE RESEARCH AND DEVELOPMENT AGREEMENT (CRADA)

Pomalidomide is provided by Celgene Corporation under CRADA # 02328 Celgene/NCI Clinical Research Leader: "Preclinical and Clinical Development of Celgene Corporation's Proprietary Immunomodulatory Agent, CC4047 (Pomalidomide), as a Therapy for Graft-Versus-Host Disease (GVHD)," executed July 13, 2010.


#### 12 HUMAN SUBJECTS PROTECTIONS

### 12.1 RATIONALE FOR SUBJECT SELECTION

No subjects will be excluded from participation based on sex, race or ethnicity. The study will be open to all subjects who satisfy the inclusion criteria and provide an informed consent to the protocol.

#### 12.2 Participation of Children

As there is no experience with pomalidomide in children, this study will be limited to subjects age 18 years or older.

## 12.3 PARTICIPATION OF NIH SUBJECTS UNABLE TO GIVE CONSENT

Adults unable to give consent are excluded from enrolling in the protocol. However re-consent may be necessary and there is a possibility, though unlikely, that subjects could become decisionally impaired. For this reason and because there is a prospect of direct benefit from research participation (section 10.5), all subjects  $\geq$  age 18 will be offered the opportunity to fill in their wishes for research and care, and assign a substitute decision maker on the "NIH Advance Directive for Health Care and Medical Research Participation" form so that another person can make decisions about their medical care in the event that they become incapacitated or cognitively impaired during the course of the study. Note: The PI or AI will contact the NIH Ability to Consent Assessment Team (ACAT) for evaluation as needed for the following: an independent assessment of whether an individual has the capacity to provide consent; assistance in identifying and assessing an appropriate surrogate when indicated; and/or an assessment of the capacity to appoint a surrogate. For those subjects that become incapacitated and do not have pre-determined substitute decision maker, the procedures described in MEC Policy 87-4 and NIH HRPP 403 for appointing a surrogate decision maker for adult subjects who are (a) decisionally impaired, and (b) who do not have a legal guardian or durable power of attorney, will be followed.

#### 12.4 EVALUATION OF BENEFITS AND RISKS/DISCOMFORTS

## 12.4.1 Related to Pomalidomide

Potential risks of pomalidomide include the range of toxicities described in Section 11.1.9 and the consent form. There may also be unexpected side effects. All subjects will be carefully monitored for side effects.

#### 12.4.2 Related to Blood Collection

Minor complications including bleeding, pain, and hematoma formation at the site of blood draws, or infections may rarely occur.

## 12.4.3 Related to Tissue Biopsy

Skin and oral punch biopsy is a minor surgical procedure that may be associated with temporary bleeding, hematoma at the site, local infection and postoperative discomfort. These risks are small (generally <5%) and transient.


### 12.4.4 Related to Pregnancy

Pomalidomide is in a class of agents that is known to be teratogenic. Women of child-bearing potential and men must agree to adhere to methods of contraception and other fertility control measures as prescribed by the protocol. This will include counseling about pregnancy precautions and the potential risks of fetal exposure conducted at a minimum of every 28 days. Women of child-bearing potential must also undergo regular pregnancy testing.

## 12.5 RISKS/BENEFITS ANALYSIS

Risks of participating in this trial include side effects from pomalidomide and risks of medical procedures (blood draws, oral and skin biopsy). Patients may receive benefit from the clinical monitoring or potentially experience improvement in cGvHD symptoms or quality of life. Therefore, this research represents more than minimal risk to subjects with prospect of direct benefit to individual subjects.

### 12.6 CONSENT PROCESS AND DOCUMENTATION

The investigational nature and research objectives of this trial, the procedure and its attendant risks and discomforts will be carefully explained to the subject. The potential subject will be educated regarding the nature of the condition, proposed intervention, and outcome measures. Study subjects will be informed that participation is entirely voluntary and that withdrawal from the study can be made at any time without penalty of benefits to which they may be entitled. Informed consent will be obtained by Dr. Steven Pavletic or his designee. At any time during participation in the protocol if new information becomes available relating to risks, adverse events, or toxicities, this information will be provided orally or in writing to all enrolled or prospective participants. Documentation will be provided to the IRB and if necessary the informed consent amended to reflect relevant information.

### 12.6.1 Telephone re-consent procedure

Reconsent on this study may be obtained via telephone according to the following procedure: the informed consent document will be sent to the subject. An explanation of the study will be provided over the telephone after the subject has had the opportunity to read the consent form. The subject will sign and date the informed consent. A witness to the subject's signature will sign and date the consent. The original informed consent document will be sent back to the consenting investigator who will sign and date the consent form with the date the consent was obtained via telephone. A fully executed copy will be returned via mail for the subject's records. The informed consent process will be documented on a progress note by the consenting investigator.

## 12.6.2 Short form consent process for non-English speaking patients

If there is an unexpected enrollment of a research participant for whom there is no translated extant IRB approved consent document, the principal investigator and/or those authorized to obtain informed consent will use the Short Form Oral Consent Process as described in MAS Policy M77-2, OSHRP SOP 12, and 45 CFR 46.117 (b) (2). The summary that will be used is the English version of the extant IRB approved consent document. Signed copies of both the English version of the consent and the translated short form will be given to the subject or their legally authorized representative and the signed original will be filed in the medical record.


Unless the PI is fluent in the prospective subject's language, an interpreter will be present to facilitate the conversation. Preferably someone who is independent of the subject (i.e., not a family member) will assist in presenting information and obtaining consent. Whenever possible, interpreters will be provided copies of the relevant consent documents well before the consent conversation with the subject (24 to 48 hours if possible).

We request prospective IRB approval of the use of the short form process and will notify the IRB at the time of continuing review of the frequency of the use of the Short Form.

#### 13 REGULATORY AND OPERATIONAL CONSIDERATIONS

### 13.1 STUDY DISCONTINUATION AND CLOSURE

This study may be temporarily suspended or prematurely terminated if there is sufficient reasonable cause. Written notification, documenting the reason for study suspension or termination, will be provided by the suspending or terminating party to study participants, investigators, funding agency, the Investigational New Drug (IND) and regulatory authorities. If the study is prematurely terminated or suspended, the Principal Investigator (PI) will promptly inform study participants, the Institutional Review Board (IRB), and sponsor and will provide the reason(s) for the termination or suspension. Study participants will be contacted, as applicable, and be informed of changes to study visit schedule.

Circumstances that may warrant termination or suspension include, but are not limited to:

- Determination of unexpected, significant, or unacceptable risk to participants
- Demonstration of efficacy that would warrant stopping
- Insufficient compliance to protocol requirements
- Data that are not sufficiently complete and/or evaluable
- Determination that the primary endpoint has been met
- Determination of futility

Study may resume once concerns about safety, protocol compliance, and data quality are addressed, and satisfy the sponsor, IRB and as applicable, Food and Drug Administration (FDA).

### 13.2 QUALITY ASSURANCE AND QUALITY CONTROL

Each clinical site will perform internal quality management of study conduct, data and biological specimen collection, documentation and completion. An individualized quality management plan will be developed to describe a site's quality management.

Quality control (QC) procedures will be implemented beginning with the data entry system and data QC checks that will be run on the database will be generated. Any missing data or data anomalies will be communicated to the site(s) for clarification/resolution.

Following written Standard Operating Procedures (SOPs), the monitors will verify that the clinical trial is conducted and data are generated and biological specimens are collected, documented (recorded), and reported in compliance with the protocol, International Council for Harmonisation Good Clinical Practice (ICH GCP), and applicable regulatory requirements (e.g., Good Laboratory Practices (GLP), Good Manufacturing Practices (GMP)).


The investigational site will provide direct access to all trial related sites, source data/documents, and reports for the purpose of monitoring and auditing by the sponsor, and inspection by local and regulatory authorities.

### 13.3 CONFLICT OF INTEREST POLICY

The independence of this study from any actual or perceived influence, such as by the pharmaceutical industry, is critical. Therefore, any actual conflict of interest of persons who have a role in the design, conduct, analysis, publication, or any aspect of this trial will be disclosed and managed. Furthermore, persons who have a perceived conflict of interest will be required to have such conflicts managed in a way that is appropriate to their participation in the design and conduct of this trial. The study leadership in conjunction with the National Cancer Institute has established policies and procedures for all study group members to disclose all conflicts of interest and will establish a mechanism for the management of all reported dualities of interest.

#### 13.4 CONFIDENTIALITY AND PRIVACY

Participant confidentiality and privacy is strictly held in trust by the participating investigators, their staff, and the sponsor(s). This confidentiality is extended to cover testing of biological samples and genetic tests in addition to the clinical information relating to participants. Therefore, the study protocol, documentation, data, and all other information generated will be held in strict confidence. No information concerning the study or the data will be released to any unauthorized third party without prior written approval of the sponsor.

All research activities will be conducted in as private a setting as possible.

The study monitor, other authorized representatives of the sponsor, representatives of the Institutional Review Board (IRB), and/or regulatory agencies may inspect all documents and records required to be maintained by the investigator, including but not limited to, medical records (office, clinic, or hospital) and pharmacy records for the participants in this study. The clinical study site will permit access to such records.

The study participant's contact information will be securely stored at the/each clinical site for internal use during the study. At the end of the study, all records will continue to be kept in a secure location for as long a period as dictated by the reviewing IRB, Institutional policies, or sponsor requirements.

Study participant research data, which is for purposes of statistical analysis and scientific reporting, will be stored at the NCI CCR. This will not include the participant's contact or identifying information. Rather, individual participants and their research data will be identified by a unique study identification number. The study data entry and study management systems used by the clinical site(s) and by NCI CCR research staff will be secured and password protected. At the end of the study, all study databases will be archived at the NCI CCR.

To further protect the privacy of study participants, a Certificate of Confidentiality has been issued by the National Institutes of Health (NIH). This certificate protects identifiable research information from forced disclosure. It allows the investigator and others who have access to research records to refuse to disclose identifying information on research participation in any civil, criminal, administrative, legislative, or other proceeding, whether at the federal, state, or local level. By protecting researchers and institutions from being compelled to disclose


information that would identify research participants, Certificates of Confidentiality help achieve the research objectives and promote participation in studies by helping assure confidentiality and privacy to participants.

#### 14 PHARMACEUTICAL INFORMATION

#### 14.1 POMALIDOMIDE

### 14.1.1 Description

Pomalidomide, 4-amino-2-(2,6-dioxo-3-piperidyl)isoindoline-1'-one)-1,3-dione, is a novel immunomodulatory drug. The Chemical Abstract Service (CAS) registry number for pomalidomide is 19171-19-8. Pomalidomide is also known as CC-4047. The chemical structure of the active pharmaceutical ingredient is as follows:

$$NH_2$$

Pomalidomide has an asymmetric carbon atom and can therefore exist as the optically active forms S (-) and R (+). Pomalidomide is being developed as a racemate.

Pomalidomide shares a number of the beneficial pharmacologic properties of thalidomide and lenalidomide, but it is a more potent anti-proliferative immunomodulating agent than either drug.

### 14.1.2 Source

Celgene Corporation will supply pomalidomide 0.5 mg, 1.0 mg, and 2.0 mg capsules. Pomalidomide will be packaged in bottles containing capsules for 28 days of every 28-day cycle. Only a 28-day supply of pomalidomide may be provided to the patient for each 28-day cycle. Site will utilize commercial supply of anti-thrombotic agents for prophylactic purposes.

Celgene will supply drug free of charge. The initial drug shipment will be sent to NIH pharmacy. NIH pharmacy will order all subsequent drug orders.

## 14.1.3 Formulation and Preparation

Pomalidomide will be administered as 2.0 mg, 1.0 mg and/or 0.5 mg capsules to be taken orally. Each daily dose of pomalidomide should be taken at approximately the same time of day. No modification of capsules is necessary.

### 14.1.4 Study Drug Packaging and Labeling

Pomalidomide investigational supplies are dispensed to the persons in individual bottles of capsules. Each bottle will identify the contents as study medication. The label for study drug supplied by Celgene will bear the Celgene Corporation name and address, the protocol number,


the quantity of study drug contained, and the standard caution statement, as follows: "Caution: New Drug - Limited by Federal Law to Investigational Use."

Pomalidomide should not be handled by FCBP unless wearing gloves. All bottles will contain the following warning label: "WARNING: POTENTIAL FOR HUMAN BIRTH DEFECTS."

### 14.1.5 Study Drug Receipt and Storage

The PI is responsible for taking an inventory of each shipment of study drug received, and comparing it with the accompanying study drug accountability form. The PI or their designee will verify the accuracy of the information on the form, sign and date it, retain a copy in the study file, and return a copy to Celgene.

At the study site, all investigational study drugs will be stored in a locked, safe area to prevent unauthorized access.

The study drug should be stored at room temperature away from direct sunlight and protected from excessive heat and cold.

#### 14.1.6 Administration Procedures

Females of childbearing potential should not handle or administer pomalidomide unless they are wearing gloves. Pomalidomide capsules should be swallowed whole, and should not be broken, chewed or opened. Pomalidomide should be taken without food, at least 2 hours before or 2 hours after a meal.

If a dose of pomalidomide is missed, it should be taken as soon as possible on the same day. If it is missed for the entire day, it should <u>not</u> be made up, rather it should be taken at the next scheduled time point.

Patients who take more than the prescribed dose of pomalidomide should be instructed to seek emergency medical care if needed and contact study staff immediately.

Accurate recording of all study drug administration (including dispensing and dosing) will be made in the source documents.

## 14.1.7 Study Drug Accountability

The PI or designee(s) is responsible for accounting for all study drug that is issued to and returned by the patient during the course of the study.

## 14.1.8 Study Drug Handling and Disposal

Celgene will instruct the Investigator(s) on the return or destruction of unused study drug. If any study drug is lost or damaged, its disposition should be documented in the patient's CRF and source documents. Study drug supplies will be retained at the clinical site pending instructions for disposition by Celgene. Patients will be instructed to return empty bottles or unused capsules.

### 14.1.9 Expected Toxicities

Likely (more than 20%): Constipation, fatigue, myalgia, and rash.

Less Likely (less than 20%): Anemia, thrombocytopenia, neutropenia, productive cough, dyspnea (with or without exertion), lung pain, nose bleeds, sore throat, discolored sputum, bloody sputum,


irritation of the upper respiratory tract, other respiratory infections, fever, headache, bacterial or viral infections, bone pain, muscle cramps, joint swelling, parasthesias, nausea, diarrhea, bloating, dry mouth and irritation of the mouth, dry skin, redness of the skin, and itching, unusual weakness or dizziness, hypotension, flushing, and chest pain.

Rare (Less than 3%): pneumonia, vomiting, blood clots in persons receiving combination therapy with other cancer drug, erythropoeitin, and/or steroids.

Experience with pomalidomide in humans and animals is detailed in the background section. Neutropenia was the most frequently reported grade 3/4 AE in subjects with relapsed/refractory multiple myeloma. The majority of these occurred without associated infection and was the dose-limiting toxicity observed during the dose finding portion of the study. Neutropenia was also the most frequently reported AE and SAE in subjects with multiple myeloma followed by thrombocytopenia and anemia. Subjects receiving pomalidomide have developed venous thromboembolic events (DVTs and pulmonary emboli) reported as SAEs. Anticoagulant prophylaxis is recommended as a precaution per protocol.

Pomalidomide was found to be teratogenic in a developmental study in rabbits. Precautions against fetal exposure are detailed throughout the protocol.

## 14.1.10Incompatibilities

Based on in vitro metabolism data, pomalidomide is not likely to precipitate drug-drug interactions especially due to inhibition or induction when co-administered with cytochrome P-450, substrates.

A food effect study with pomalidomide has not been conducted.


### 15 REFERENCES

1. Lee SJ VG, Flowers ME. Chronic graft-versus-host disease. *Biol Blood Marrow Transplant*. 2003;9(4):215-233.

- 2. Lee SJ KJ, Barrett AJ, Ringden O, Antin JH, Cahn JY, Carabasi MH, Gale RP, Giralt S, Hale GA, Ilhan O, McCarthy PL, Socie G, Verdonck LF, Weisdorf DJ, Horowitz MM. Severity of chronic graft-versus-host disease: association with treatment-related mortality and relapse. *Blood*. 2002;100(2):406-414.
- 3. Filipovich AH WD, Pavletic S, Socie G, Wingard JR, Lee SJ, Martin P, Chien J, Przepiorka D, Couriel D, Cowen EW, Dinndorf P, Farrell A, Hartzman R, Henslee-Downey J, Jacobsohn D, McDonald G, Mittleman B, Rizzo JD, Robinson M, Schubert M, Schultz K, Shulman H, Turner M, Vogelsang G, Flowers ME. National Institutes of Health consensus development project on criteria for clinical trials in chronic graft-versus-host disease: I. Diagnosis and staging working group report. *Biol Blood Marrow Transplant*. 2005;11(12):945-956.
- 4. Vogelsang GB PS. Chronic Graft Versus Host Disease

Interdisciplinary Management. Cambridge University Press; 2009.

- 5. Pavletic SZ CS, Kernan NA, Henslee-Downey J, Mendizabal AM, Papadopoulos E, Gingrich R, Casper J, Yanovich S, Weisdorf D. Influence of T-cell depletion on chronic graft-versus-host disease: results of a multicenter randomized trial in unrelated marrow donor transplantation. *Blood.* 2005;106(9):3308-3313.
- 6. Baird K PS. Chronic graft versus host disease. *Curr Opin Hematol.* 2006;13(6):426-435.
- 7. Socie G RJ, Martin PJ. Current challenges in chronic graft-versus-host disease. *Biol Blood Marrow Transplant*. 2010;16:146-151.
- 8. Le NT CN. Regulating regulatory T cells. Bone Marrow Transplant. 2007;39(1)::1-9.
- 9. Koreth J, Matsuoka K, Kim HT, et al. Interleukin-2 and regulatory T cells in graft-versus-host disease. *N Engl J Med*. 2011;365(22):2055-2066.
- 10. Skert C DD, Michelutti A, Patriarca F, Arpinati M, Filì C, Lucchi P, Malagola M, Bergonzi C, Roccaro A, Peli A, Ricotta D, Caimi L, Fanin R, Baccarani M, Russo D. Kinetics of Th1/Th2 cytokines and lymphocyte subsets to predict chronic GVHD after allo-SCT: results of a prospective study. *Bone Marrow Transplant*. 2009;44(11):729-737.
- 11. Barak V L-SF, Nisman B, Nagler A. Cytokine dysregulation in chronic graft versus host disease. *Leuk Lymphoma*. 1995;17((1-2)):169-173.
- 12. Liem LM FW, van Houwelingen HC, Goulmy E. Serum transforming growth factor-beta1 levels in bone marrow transplant recipients correlate with blood cell counts and chronic graft-versus-host disease. *Transplantation*. 1999;67(1).
- 13. Bogunia-Kubik K MA, Wysoczanska B, Lange A. Recipient interferon-gamma 3/3 genotype contributes to the development of chronic graft-versus-host disease after allogeneic hematopoietic stem cell transplantation. *Haematologica*. 2005;90(3):425-426.
- 14. Zhang C TI, Zhang Z, Liu Y, Kandeel F, Forman S, Strober S, Zeng D. Donor CD4+ T and B cells in transplants induce chronic graft-versus-host disease with autoimmune manifestations. *Blood*. 2006;107(7):2993-3001.


15. Trendelenburg M GM, Passweg J, Tichelli A, Tyndall A, Gratwohl A. "Altered immunity syndrome", a distinct entity in long-term bone marrow transplantation survivors? *Bone Marrow Transplant*. 2001;28(12):1175-1176.

- 16. Patriarca F SC, Sperotto A, Zaja F, Falleti E, Mestroni R, Kikic F, Calistri E, Filì C, Geromin A, Cerno M, Fanin R. The development of autoantibodies after allogeneic stem cell transplantation is related with chronic graft-vs-host disease and immune recovery. *Exp Hematol.* 2006;34(3):389-396.
- 17. Svegliati S OA, Campelli N, Luchetti M, Poloni A, Trappolini S, Moroncini G, Bacigalupo A, Leoni P, Avvedimento EV, Gabrielli A. Stimulatory autoantibodies to PDGF receptor in patients with extensive chronic graft-versus-host disease. *Blood.* 2007;110(1):237-241.
- 18. Sarantopoulos S SK, Kim HT, Bhuiya NS, Cutler CS, Soiffer RJ, Antin JH, Ritz J. High levels of B-cell activating factor in patients with active chronic graft-versus-host disease. *Clin Cancer Res.* 2007;13(20):6107-6114.
- 19. Fujii H CG, She K, Aslanian S, Shimizu H, Kariminia A, Krailo M, Chen Z, McMaster R, Bergman A, Goldman F, Grupp SA, Wall DA, Gilman AL, Schultz KR. Biomarkers in newly diagnosed pediatric-extensive chronic graft-versus-host disease: a report from the Children's Oncology Group. *Blood*. 2008;111(6):3276-3285.
- 20. Cutler C, Miklos D, Kim HT, et al. Rituximab for steroid-refractory chronic graft-versus-host disease. *Blood.* 2006;108(2):756-762.
- 21. Bhushan V, Collins RH, Jr. Chronic graft-vs-host disease. *JAMA*. 2003;290(19):2599-2603.
- 22. Filipovich AH, Weisdorf D, Pavletic S, et al. National Institutes of Health consensus development project on criteria for clinical trials in chronic graft-versus-host disease: I. Diagnosis and staging working group report. *Biol Blood Marrow Transplant*. 2005;11(12):945-956.
- 23. Lee SJ. New approaches for preventing and treating chronic graft-versus-host disease. *Blood.* 2005;105(11):4200-4206.
- 24. Shlomchik WD. Graft-versus-host disease. *Nat Rev Immunol*, 2007;7(5):340-352.
- 25. Shlomchik WD, Lee SJ, Couriel D, Pavletic SZ. Transplantation's greatest challenges: advances in chronic graft-versus-host disease. *Biol Blood Marrow Transplant*. 2007;13(1 Suppl 1):2-10.
- 26. Wolff D, Schleuning M, von Harsdorf S, et al. Consensus Conference on Clinical Practice in Chronic GVHD: Second-Line Treatment of Chronic Graft-versus-Host Disease. *Biol Blood Marrow Transplant*. 2011;17(1):1-17.
- 27. Couriel D, Carpenter PA, Cutler C, et al. Ancillary therapy and supportive care of chronic graft-versus-host disease: national institutes of health consensus development project on criteria for clinical trials in chronic Graft-versus-host disease: V. Ancillary Therapy and Supportive Care Working Group Report. *Biol Blood Marrow Transplant*. 2006;12(4):375-396.
- 28. Martin PJ, Weisdorf D, Przepiorka D, et al. National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: VI. Design of Clinical Trials Working Group report. *Biol Blood Marrow Transplant*. 2006;12(5):491-505.


29. Pavletic SZ, Martin P, Lee SJ, et al. Measuring therapeutic response in chronic graft-versus-host disease: National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: IV. Response Criteria Working Group report. *Biol Blood Marrow Transplant*. 2006;12(3):252-266.

- 30. Schultz KR, Miklos DB, Fowler D, et al. Toward biomarkers for chronic graft-versus-host disease: National Institutes of Health consensus development project on criteria for clinical trials in chronic graft-versus-host disease: III. Biomarker Working Group Report. *Biol Blood Marrow Transplant*. 2006;12(2):126-137.
- 31. Shulman HM, Kleiner D, Lee SJ, et al. Histopathologic diagnosis of chronic graft-versus-host disease: National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: II. Pathology Working Group Report. *Biol Blood Marrow Transplant*. 2006;12(1):31-47.
- 32. Flowers ME, Martin PJ. Evaluation of thalidomide for treatment or prevention of chronic graft-versus-host disease. *Leuk Lymphoma*. 2003;44(7):1141-1146.
- 33. Flowers ME, Storer B, Carpenter P, et al. Treatment change as a predictor of outcome among patients with classic chronic graft-versus-host disease. *Biol Blood Marrow Transplant*. 2008;14(12):1380-1384.
- 34. Flowers ME MP. Evaluation of thalidomide for treatment or prevention of chronic graft-versus-host disease. *Leuk Lymphoma*. 2003;44(7):1141-1146.
- 35. Martin PJ, Inamoto Y, Carpenter PA, Lee SJ, Flowers ME. Treatment of chronic graft-versus-host disease: Past, present and future. *Korean J Hematol.* 2011;46(3):153-163.
- 36. Vogelsang GB FE, Hess AD, Altamonte V, Beschorner WE, Jabs DA, Corio RL, Levin LS, Colvin OM, Wingard JR, et al. Thalidomide for the treatment of chronic graft-versus-host disease. *N Engl J Med.* 1992;326(16):1055-1058.
- 37. Tefferi A VS, Barosi G, Passamonti F, Roboz GJ, Gisslinger H, Paquette RL, Cervantes F, Rivera CE, Deeg HJ, Thiele J, Kvasnicka HM, Vardiman JW, Zhang Y, Bekele BN, Mesa RA, Gale RP, Kantarjian HM. Pomalidomide is active in the treatment of anemia associated with myelofibrosis. *J Clin Oncol.* 2009;27(27):4563-4569.
- 38. Heney D ND, Wheeldon J, Bailey CC, Lewis IJ, Barnard DL. Thalidomide treatment for chronic graft-versus-host disease. *Br J Haematol.* 1991;78(1):23-27.
- 39. Rovelli A AC, Nesi F, Balduzzi A, Nicolini B, Locasciulli A, Vassallo E, Miniero R, Uderzo C. The role of thalidomide in the treatment of refractory chronic graft-versus-host disease following bone marrow transplantation in children. *Bone Marrow Transplant*. 1998;21(6):577-581.
- 40. Forsyth CJ, Cremer PD, Torzillo P, Iland HJ, Young GA. Thalidomide responsive chronic pulmonary GVHD. *Bone Marrow Transplant.* 1996;17(2):291-293.
- 41. Staumont-Salle D, Magro L, Piette F, Thomas P, Jouet JP, Catteau B. Chronic graft-versus-host disease revealed by lichenoid vulvar lesions successfully treated with thalidomide. *Acta Derm Venereol.* 2003;83(4):302-303.
- 42. Browne PV WD, DeFor T, Miller WJ, Davies SM, Filipovich A, McGlave PB, Ramsay NK, Wagner J, Enright H. Response to thalidomide therapy in refractory chronic graft-versus-host disease. *Bone Marrow Transplant*::26(8):865-869.


43. Cole CH RP, Pritchard S, Phillips G, Chan KW. Thalidomide in the management of chronic graft-versus-host disease in children following bone marrow transplantation. *Bone Marrow Transplant*. 1994;14(6):937-942.

- 44. Mehta P, Kedar A, Graham-Pole J, Skoda-Smith S, Wingard JR. Thalidomide in children undergoing bone marrow transplantation: series at a single institution and review of the literature. *Pediatrics*. 1999;103(4):e44.
- 45. Arora M WJ, Davies SM, Blazar BR, Defor T, Enright H, Miller WJ, Weisdorf DF. Randomized clinical trial of thalidomide, cyclosporine, and prednisone versus cyclosporine and prednisone as initial therapy for chronic graft-versus-host disease. *Biol Blood Marrow Transplant*. 2001;7(5):265-273.
- 46. Koc S LW, Flowers ME, Anasetti C, Deeg HJ, Nash RA, Sanders JE, Witherspoon RP, Appelbaum FR, Storb R, Martin PJ. Thalidomide for treatment of patients with chronic graft-versus-host disease. *Blood.* 2000;96(12):3995-3996.
- 47. Chao NJ, Parker PM, Niland JC, et al. Paradoxical effect of thalidomide prophylaxis on chronic graft-vs.-host disease. *Biol Blood Marrow Transplant.* 1996;2(2):86-92.
- 48. Parker PM CN, Nademanee A, O'Donnell MR, Schmidt GM, Snyder DS, Stein AS, Smith EP, Molina A, Stepan DE, Kashyap A, Planas I, Spielberger R, Somlo G, Margolin K, Zwingenberger K, Wilsman K, Negrin RS, Long GD, Niland JC, Blume KG, Forman SJ. Thalidomide as salvage therapy for chronic graft-versus-host disease. *Blood*. 1995;86(9):3604-3609.
- 49. Kulkarni S PR, Sirohi B, Treleaven J, Saso R, Horton C, Atra A, Ortin M, Rudin C, Goyal S, Sankpal S, Meller S, Pinkerton CR, Mehta J, Singhal S. Thalidomide after allogeneic haematopoietic stem cell transplantation: activity in chronic but not in acute graft-versushost disease. *Bone Marrow Transplant*. 2003;32(2):165-170.
- 50. Payvandi F, Wu L, Haley M, et al. Immunomodulatory drugs inhibit expression of cyclooxygenase-2 from TNF-alpha, IL-1beta, and LPS-stimulated human PBMC in a partially IL-10-dependent manner. *Cell Immunol.* 2004;230(2):81-88.
- 51. Corral LG, Haslett PA, Muller GW, et al. Differential cytokine modulation and T cell activation by two distinct classes of thalidomide analogues that are potent inhibitors of TNF-alpha. *J Immunol.* 1999;163(1):380-386.
- 52. Dredge K, Marriott JB, Todryk SM, et al. Protective antitumor immunity induced by a costimulatory thalidomide analog in conjunction with whole tumor cell vaccination is mediated by increased Th1-type immunity. *J Immunol.* 2002;168(10):4914-4919.
- 53. Schafer PH, Gandhi AK, Loveland MA, et al. Enhancement of cytokine production and AP-1 transcriptional activity in T cells by thalidomide-related immunomodulatory drugs. *J Pharmacol Exp Ther.* 2003;305(3):1222-1232.
- 54. Schey SA, Fields P, Bartlett JB, et al. Phase I study of an immunomodulatory thalidomide analog, CC-4047, in relapsed or refractory multiple myeloma. *J Clin Oncol.* 2004;22(16):3269-3276.
- 55. Galustian C, Klaschka DC, Meyer B, Labarthe M-C, Bartlett JB, Dalgleish AG. Lenalidomide (Revlimid(R), CC-5013) and ActimidTM (CC-4047) inhibit the function and expansion of T regulatory (Treg) cells in vitro: Implications for anti-tumor activity in vivo. *AACR Meeting Abstracts.* 2006;2006(1):1147-a-.


56. Verhelle D, Corral LG, Wong K, et al. Lenalidomide and CC-4047 inhibit the proliferation of malignant B cells while expanding normal CD34+ progenitor cells. *Cancer Res.* 2007;67(2):746-755.

- 57. Suppiah R, Srkalovic JG, Hussein MA. Immunomodulatory analogues of thalidomide in the treatment of multiple myeloma. *Clin Lymphoma Myeloma*. 2006;6(4):301-305.
- 58. Ito T, Ando H, Suzuki T, et al. Identification of a primary target of thalidomide teratogenicity. *Science*. 2010;327(5971):1345-1350.
- 59. Zhu YX, Braggio E, Shi CX, et al. Cereblon expression is required for the antimyeloma activity of lenalidomide and pomalidomide. *Blood*. 2011;118(18):4771-4779.
- 60. Brustle A, Heink S, Huber M, et al. The development of inflammatory T(H)-17 cells requires interferon-regulatory factor 4. *Nat Immunol*. 2007;8(9):958-966.
- 61. Mudter J, Yu J, Zufferey C, et al. IRF4 regulates IL-17A promoter activity and controls RORgammat-dependent Th17 colitis in vivo. *Inflamm Bowel Dis.* 2011;17(6):1343-1358.
- 62. Bartlett JB DK, Dalgleish AG. The evolution of thalidomide and its IMiD derivatives as anticancer agents. *Nat Rev Cancer*. 2004;4(4):314-322.
- 63. Xu W CM, Sankar S, Webb DR, Bennett BL. CC-4047 promotes Th1 cell differentiation and reprograms polarized human Th2 cells by enhancing transcription factor T-bet. *Clin Immunol.* 2008;128(3):392-399.
- 64. Streetly MJ GK, Daniel Y, Zeldis JB, Kazmi M, Schey SA. Alternate day pomalidomide retains anti-myeloma effect with reduced adverse events and evidence of in vivo immunomodulation. *Br J Haematol.* 2008;141(1):41-51.
- 65. Schey SA FP, Bartlett JB, Clarke IA, Ashan G, Knight RD, Streetly M, Dalgleish AG. Phase I study of an immunomodulatory thalidomide analog, CC-4047, in relapsed or refractory multiple myeloma. *J Clin Oncol.* 2004;22(16):3269-3276.
- 66. Rusten LS JS. Tumor necrosis factor (TNF)-alpha directly inhibits human erythropoiesis in vitro: role of p55 and p75 TNF receptors. *Blood.* 1995;154(8):3732-3741.
- 67. Pusic I, DiPersio JF, Goran SL, et al. Pomalidomide (POM) In Advanced Corticosteroid-Resistant Chronic Graft-Versus-Host Disease (cGVHD). *Biology of Blood and Marrow Transplantation: Journal of the American Society for Blood and Marrow Transplantation.* 2010;16(2):S311.
- 68. Mesa RA PA, Hussein K, Wu W, Schwager S, Litzow MR, Hogan WJ, Tefferi A. Phase1/-2 study of Pomalidomide in myelofibrosis. *Am J Hematol.* 2010 Feb;85(2):129-130.
- 69. Lacy MQ HS, Gertz MA, Dispenzieri A, Buadi F, Kumar S, Greipp PR, Lust JA, Russell SJ, Dingli D, Kyle RA, Fonseca R, Bergsagel PL, Roy V, Mikhael JR, Stewart AK, Laumann K, Allred JB, Mandrekar SJ, Rajkumar SV. Pomalidomide (CC4047) plus low-dose dexamethasone as therapy for relapsed multiple myeloma. *J Clin Oncol*. 2009;27(30):5008-5014.
- 70. Begna KH MR, Pardanani A, Hogan WJ, Litzow MR, McClure RF, Tefferi A. A phase-2 trial of low-dose pomalidomide in myelofibrosis. *Leukemia*. 2011;25(2):301-304.
- 71. Arai S, Jagasia M, Storer B, et al. Global and organ-specific chronic graft-versus-host disease severity according to the 2005 NIH Consensus Criteria. *Blood*. 2011;118(15):4242-4249.


72. Kuzmina Z, Eder S, Bohm A, et al. Significantly worse survival of patients with NIH-defined chronic graft-versus-host disease and thrombocytopenia or progressive onset type: results of a prospective study. *Leukemia*. 2011.

- 73. Mitchell SA, Jacobsohn D, Thormann Powers KE, et al. A multicenter pilot evaluation of the National Institutes of Health chronic graft-versus-host disease (cGVHD) therapeutic response measures: feasibility, interrater reliability, and minimum detectable change. *Biol Blood Marrow Transplant*. 2011;17(11):1619-1629.
- 74. Lyman GH, Khorana AA, Falanga A, et al. American Society of Clinical Oncology guideline: recommendations for venous thromboembolism prophylaxis and treatment in patients with cancer. *J Clin Oncol*. 2007;25(34):5490-5505.
- 75. Lee S, Cook EF, Soiffer R, Antin JH. Development and validation of a scale to measure symptoms of chronic graft-versus-host disease. *Biol Blood Marrow Transplant*. 2002;8(8):444-452.


# 16 APPENDICES

## 16.1 APPENDIX A: PERFORMANCE STATUS CRITERIA

| ECOG Performance Status Scale | | Karnofsky Performance Scale | |
|---|---|---|---|
| Grade | Descriptions | Percent | Description |
| 0 | Normal activity. Fully active, able to carry on all pre-disease performance without restriction. | 100 | Normal, no complaints, no evidence of disease. |
| | | 90 | Able to carry on normal activity; minor signs or symptoms of disease. |
| | Symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able to | 80 | Normal activity with effort; some signs or symptoms of disease. |
| 1 | carry out work of a light or sedentary nature (e.g., light housework, office work). | 70 | Cares for self, unable to carry o normal activity or to do activ work. |
| 2 | In bed <50% of the time.<br>Ambulatory and capable of all self-<br>care, but unable to carry out any<br>work activities. Up and about<br>more than 50% of waking hours. | 60 | Requires occasional assistance, but is able to care for most of his/her needs. |
| | | 50 | Requires considerable assistance and frequent medical care. |
| 2 | In bed >50% of the time. Capable of only limited self-care, confined | 40 | Disabled, requires special care and assistance. |
| 3 | to bed or chair more than 50% of waking hours. | 30 | Severely disabled, hospitalization indicated. Death not imminent. |
| 4 | 100% bedridden. Completely disabled. Cannot carry on any self- | 20 | Very sick, hospitalization indicated. Death not imminent. |
| | care. Totally confined to bed or chair. | 10 | Moribund, fatal processes progressing rapidly. |
| 5 | Dead. | 0 | Dead. |


#### 16.2 APPENDIX B: MEASUREMENT OF POMALIDOMIDE SERUM LEVELS

## **Blood and Plasma Sample Labeling**

Labels must contain the following information:

- Protocol No.:
- Subject ID number:
- Nominal Time Point:

All blood and plasma collection tubes and storage vials should be labeled and chilled on wet ice **prior to** sample collection and processing.

## **Blood Sample Collection**

- Research nurses will give the Figg lab 24 hours advance notice on PK blood draws.
- Fill an ice bucket with a sufficient amount of ice to pre-chill all collection tubes before blood draw.
- Collect approximately 6 mL of whole blood into a pre-chilled 6-mL K<sub>3</sub>EDTA tube to which 1% hydrochloric acid has been added (supplied by Figg Laboratory). Blood can be collected via direct vein puncture or indwelling catheter.
- Accurately record the time of blood collection.
- Gently invert the tube 3-5 times and immerse it into ice immediately to prevent possible compound degradation at room temperature.
- The date, cycle day, and **exact** time of each blood draw should be recorded on the sample tube and the PK sheet containing the study number and unique patient identifier.
- Please page 102-11964 (Gareth Peters or alternate tech) for immediate pick-up. (Contact the Clinical Pharmacology Program (CPP) processing group in 10/5A09 at 301-594-6131 or 301-402-3622 with any questions).

## **Blood Sample Processing to Obtain Plasma**

- Within 30 minutes of collection, the blood sample must be centrifuged at 1,500 g (about 3,000 rpm dependent upon the type of centrifuge) for 10 min at 4°C to obtain plasma.
- Using Eppendorf pipettes (or equivalent) to transfer approximately 0.7 mL of plasma into each of the two pre-labeled, pre-chilled, citric acid-containing polypropylene storage vials (one primary and one back-up, provide by Celgene). Keep storage vials on ice before they are ready to be transferred into a freezer.
- Within 60 minutes of blood collection, transfer plasma samples in storage vials into a -80°C freezer, where they will remain stored until analysis.
- Immediately record the time of sample entry into the freezer.
- Patient data will be entered into a secure and encrypted LabSamples database maintained by the Clinical Pharmacology Program, Office of the Clinical Director

**Abbreviated Title:** Pomalidomide for cGvHD **Version Date:** 4/29/2025

# 16.3 APPENDIX C: DIAGNOSTIC CRITERIA OF CHRONIC GVHD

| Organ or Site | Diagnostic<br>Features <sup>1</sup> | Distinctive<br>Features <sup>2</sup> | Others <sup>3</sup> | Common Features <sup>4</sup> |
|---|---|---|---|---|
| Skin | Poilkiloderma Lichen planus- like features Sclerotic features Morphea-like features Lichen sclerosus-like features | Depigmentatio<br>n | Sweat impairment Ichthyosis Keratosis pilaris Hypopigmentation Hyperpigmentatio n | Erythema Maculopapular rash Pruritus |
| Nails | | Dystrophy Longitudinal ridging, splitting, or brittle features Onycholysis Pterygium unguis Nail loss 5,6 | | |
| Scalp and body hair | | New onset of scarring or nonscarring scalp alopecia <sup>7</sup> Scaling, papulosquamo us lesion | Thinning scalp<br>hair, typically<br>patchy, coarse, or<br>dull <sup>8</sup><br>Premature grey<br>hair | |


| Organ or Site | Diagnostic<br>Features <sup>1</sup> | Distinctive<br>Features <sup>2</sup> | Others <sup>3</sup> | Common Features <sup>4</sup> |
|---|---|---|---|---|
| Mouth | Lichen-type features Hyperkeratotic plaques Restriction of mouth opening from sclerosis | Xerostomia Mucocele Mucosal atrophy Pseudomembra nes <sup>6</sup> Ulcers <sup>6</sup> | | Gingivitis Mucositis Erythema Pain |
| Eyes | | New onset dry, gritty, or painful eyes <sup>9</sup> Cicatricial conjunctivitis Keratoconjunct ivitis sicca <sup>9</sup> Confluent areas of punctuate keratopathy | Photophobia Periorbital hyperpigmentation Blepharitis <sup>10</sup> | |
| Genitalia | Lichen planus-<br>like features<br>Vaginal<br>scarring or<br>stenosis | Erosions <sup>6</sup> Fissures <sup>6</sup> Ulcers <sup>6</sup> | | |
| Lung | Bronchiolitis<br>obliterans<br>diagnosed with<br>lung biopsy | Bronchiolitis<br>obliterans<br>diagnosed with<br>PFTs <sup>12</sup> and<br>radiology <sup>9</sup> | | BOOP 13 |
| Muscle,<br>Fascia, joints | Fasciitis Joint stiffness or contractures secondary to sclerosis | Myositis or polymyositis | Edema Muscle cramps Arthralgia or arthritis | |


| Organ or Site | Diagnostic<br>Features <sup>1</sup> | Distinctive<br>Features <sup>2</sup> | Others <sup>3</sup> | Common Features <sup>4</sup> |
|---|---|---|---|---|
| Hematopoiet ic and immune | | | | Thrombocytopenia Eosinophilia Lymphopenia Hypo- or hypergammaglobilin emia Autoantibodies (AIHA and ITP) 14 |
| Other | | | | Pericardial or pleural effusions Ascites Peripheral neuropathy Nephrotic syndrome Myasthenia gravis Cardiac conduction abnormality or cardiomyopathy |

- 1.Sufficient to establish the diagnosis of cGvHD
- 2. Seen in cGvHD, but insufficient alone to establish a diagnosis of cGvHD
- 3.Can be acknowledged as part of the cGvHD symptomatology if the diagnosis is confirmed
- 4. Seen with both acute and cGvHD
- 5. Usually symmetric, affects most nails
- 6.In all cases, infection, drug effects, malignancy, or other causes must be excluded.
- 7. After recovery from chemoradiation therapy
- 8. Not explained by endocrine or other causes
- 9. Diagnosis of cGvHD requires biopsy or radiology confirmation (or Schirmer test for eyes)
- 10.Erythema of the eyelids with edema
- 11.Infants and children
- 12.Pulmonary function tests
- 13. Bronchiolitis obliterans-organizing pneumonia


14.AIHA: autoimmune hemolytic anemia; ITP: idiopathic thrombocytopenic purpura


# 16.4 APPENDIX D: CLINICAL DIFFERENTIATION OF ACUTE AND CHRONIC GVHD

| Category | Time of<br>Symptoms After<br>HCT or DLI | | Presence of<br>Chronic GVHD<br>Features <sup>2</sup> |
|---|---|---|---|
| Acute GVHD | | | |
| Classic acute GVHD | ≤ 100 days | Yes | No |
| Persistent, recurrent, or late-onset acute GVHD | > 100 days | Yes | No |
| Chronic GVHD | | | |
| Classic cGvHD | No time limit | No | Yes |
| Overlap syndrome | No time limit | Yes | Yes |

1. Abbreviations: HCT: hematopoietic cell transplantation; DLI: donor lymphocyte infusion

2. See Appendix C for features

## 16.5 APPENDIX E: ORGAN SPECIFIC AND GLOBAL SCORING OF CHRONIC GVHD

| | SCORE 0 | SCORE 1 | SCORE 2 | SCORE 3 |
|---|---|---|---|---|
| PERFORMANCE SCORE: KPS ECOG LPS | Asymptomatic and fully active (ECOG 0; KPS or LPS 100%) | Symptomatic, fully<br>ambulatory, restricted<br>only in physically<br>strenuous activity<br>(ECOG 1, KPS or<br>LPS 80-90%) | Symptomatic,<br>ambulatory, capable<br>of self-care, >50% of<br>waking hours out of<br>bed (ECOG 2, KPS<br>or LPS 60-70%) | Symptomatic,<br>limited self-care,<br>>50% of waking hours<br>in bed (ECOG 3-4,<br>KPS or LPS <60%) |
| SKIN Clinical features: Maculopapular rash Lichen planus-like features Papulosquamous lesions or ichthyosis Hyperpigmentation Hypopigmentation Keratosis pilaris Erythema Erythroderma Poikiloderma Sclerotic features Pruritus Hair involvement Nail involvement | No Symptoms | <18% BSA with disease signs but NO sclerotic features | 19-50% BSA OR involvement with superficial sclerotic features "not hidebound" (able to pinch) | >50% BSA OR deep sclerotic features "hidebound" (unable to pinch) OR impaired mobility, ulceration or severe pruritus |
| involved | | | | |
| Моитн | No symptoms | Mild symptoms<br>with disease signs but<br>not limiting oral<br>intake significantly | Moderate<br>symptoms with<br>disease signs with<br>partial limitation of<br>oral intake | Severe symptoms<br>with disease signs on<br>examination with<br>major limitation of oral<br>intake |
| LIP Print Name: | | LIP Signature: | | |
| Date of Evaluation: | | | | |
| Timepoint: Baseline | Off Study | | | |


| | SCORE 0 | SCORE 1 | SCORE 2 | SCORE 3 |
|---|---|---|---|---|
| GI TRACT | No symptoms | Symptoms such as dysphagia, anorexia, nausea, vomiting, abdominal pain or diarrhea without significant weight loss (<5%) | Symptoms<br>associated with mild<br>to moderate weight<br>loss (5-15%) | Symptoms associated with significant weight loss >15%, requires nutritional supplement for most calorie needs <b>OR</b> esophageal dilation |
| Liver | Normal LFT | Elevated Bilirubin,<br>AP*, AST or ALT <2<br>x ULN | Bilirubin >3 mg/dl<br>or Bilirubin,<br>enzymes 2-5 x ULN | Bilirubin or enzymes > 5 x ULN |
| Lungs* | No symptoms | Mild symptoms<br>(shortness of breath<br>after climbing one<br>flight of steps) | Moderate<br>symptoms (shortness<br>of breath after<br>walking on flat<br>ground) | Severe symptoms (shortness of breath at rest; requiring $0_2$ ) |
| FEV1 DLCO | FEV1 > 80%<br><b>OR</b> LFS=2 | FEV1 60-79% <b>OR</b><br>LFS 3-5 | FEV1 40-59%<br><b>OR</b> LFS 6-9 | FEV1 ≤39% <b>OR</b><br>LFS 10-12 |
| EYES Mean tear test (mm): >10 6-10 ≤5 Not done | No symptoms | Mild dry eye symptoms not affecting ADL (requiring eyedrops ≤ 3 x per day) <b>OR</b> asymptomatic signs of keratoconjunctivitis sicca | Moderate dry eye symptoms partially affecting ADL (requiring drops > 3 x per day or punctal plugs), WITHOUT vision impairment | Severe dry eye symptoms significantly affecting ADL (special eyeware to relieve pain) <b>OR</b> unable to work because of ocular symptoms <b>OR</b> loss of vision caused by keratoconjunctivitis sicca |
| LIP Print Name: Date of Evaluation: | | LIP Signature: | | |
| Timepoint: Baseline | Off Study | | | |

SCORE 0


range of 2-12.

JOINTS AND FASCIA Mild tightness of No symptoms Tightness of arms Contractures WITH arms or legs, normal or legs **OR** joint significant decrease of contractures, or mild decreased ROM AND significant range of motion erythema due to limitation of ADL (ROM) AND not fasciitis, moderate (unable to tie shoes, affecting ADL decrease ROM AND button shirts, dress self mild to moderate etc.) limitation of ADL GENITAL TRACT Symptomatic with Symptomatic with Symptomatic WITH No symptoms mild signs on exam moderate signs on advanced signs AND no effect on exam AND with (stricture, labial coitus and minimal mild dyspareunia or agglutination or severe discomfort with discomfort with ulceration) AND gynecologic exam gynecologic exam severe pain with coitus or inability to insert vaginal speculum \* AP may be elevated in growing children, and not reflective of liver dysfunction Other indicators, clinical manifestations or complications related to cGVHD (check all that apply and assign a score to its severity (0-3) based on its functional impact (none – 0,mild -1, moderate -2, severe – 3) Sesophageal stricture or web Pericardial Effusion Pleural Effusion(s) Nephrotic syndrome Peripheral Neuropathy Ascites (serositis) Cardiomyopathy <sup>1</sup> Eosinophilia > 500μl\_\_\_\_ Myasthenia Gravis Polymyositis Cardiac conduction defects Coronary artery involvement ¶ Platelets <100,000/μl \_\_\_\_ Progressive onset OTHERS: LIP Print Name: LIP Signature: **Date of Evaluation:** Timepoint: Baseline Off Study When discrepancy exists between pulmonary symptom or PFT scores the higher value should be used for final scoring. Scoring using the Lung Function Score (LFS) is preferred, but if DLCO is not available, grading using FEV1 should be used. The percent predicted FEV1 and DLCO (adjusted for hematocrit but not alveolar volume) should be converted to a numeric score as follows:

>80% = 1; 70-79% = 2; 60-69% = 3; 50-59% = 4; 40-49% = 5; <40% = 6. The LFS = FEV1 score + DLCO score, with a possible

SCORE 1

SCORE 2

**SCORE 3** 


## 16.6 APPENDIX F: GLOBAL SCORING OF CGVHD

| Stage | Definition |
|---|---|
| Mild | Only 1 or 2 organs or site (except the lung) No clinically significant functional impairment (maximum of score 1 in all affected organs or sites) |
| Moderate | At least 1 organ or site with clinically significant but no major disability (maximum score of 2 in any affected organ or site), or 3 or more organs or sites with no clinically significant functional impairment (maximum score of 1 in all affected organs or sites) |
| Severe | Major disability caused by cGvHD (score of 3 in any organ or site) Lung function score ≥ 2 |


## 16.7 APPENDIX G: CHRONIC GVHD ASSESSMENT (CLINICIAN) FORM

| Current ration: Young S Date: Wik#/Name: | Current Patient Weight: | Today's Date: | MR#/Name: |
|---|---|---|---|
|---|---|---|---|

| Component | Findings | | | | | | Scoring (see skin score worksheet) | | |
|---|---|---|---|---|---|---|---|---|---|
| Skin | Erythemator | Erythematous rash of any sort | | | | | | % BSA (max 100%) | |
| 19 Front 18 Back | Moveable so | elerosis | | | | | | % | BSA (max 100%) |
| | Non-moveable sclerosis (hidebound/non-pinchable) or subcutaneous sclerosis/fasciitis | | | | | % BSA (max 100%) | | | |
| | Ulcer(s): select the largest ulcerative lesion, and measure its longest dimension in cm and mark location of ulcer | | | | | | | | |
| | | | | | | | Longest dime | ensi | on:cm |
| <b>Eyes</b> Bilateral Schirmer's Tear Test | Right Eye: wetting | | | mm of | Left<br>wetti | • | | | mm of |
| (without anesthesia) in persons 9 years or older | | | | | | | | | |
| Mouth | Mucosal<br>change | No evid<br>of CGVH | | | derate | | Severe | | |
| | Erythema | None | 0 | Mild erythema<br>moderate erythen<br>(<25%) | | or | derate (≥25%)<br>Severe<br>hema (<25%) | l . | Severe erythema 3 (≥25%) |

| Mouth Hard Palate Soft Palate | Lichenoid | None 0 | Hyperkeratotic changes(<25%) | 1 | Hyperkeratotic changes(25-50%) | 2 Hyperker changes ( | |
|---|---|---|---|---|---|---|---|
| Pharynx - Uvula - Tongue | Ulcers | None 0 | None | 0 | Ulcers involving 3 (≤20%) | Severe ulceration (>20%) | as 6 |
| | Mucoceles* | None 0 | 1-5 mucoceles | 1 | 6-10 scattered 2 mucoceles | Over mucocele | s 10 3 |
| | | | *Mucoceles sco<br>lower labial an<br>palate only | | | Total sc<br>all<br>changes | ore for<br>mucosal |
| Blood Counts Platelet (K/uL) | Count U | LN (K/uL) | Total WBC (K/uL) ULN (K/uL) | | Eosinophil | s (%) | |
| Liver Function Total bilirubin ( | | LN (mg/dL) | ALT (U/L) | ULN (U/L) Alkaline Phosphatase | | | JLN (U/L) |
| Gastrointestinal-Upper GI | $0=no\ symp$ | otoms | 1 | | | | |
| 1.1 | 1=mild, occasional symptoms, with little reduction in oral intake during the past week 2=moderate, intermittent symptoms, with some reduction in oral intake during the past week | | | | | | |

| Nausea & Vomiting | 3=more severe or persistent symptoms throughout the day, with marked reduction in oral intake, on almost every day of the past week | | |
|---|---|---|---|
| Gastrointestinal- | 0= no esophageal symptoms | | |
| Esophageal | 1=Occasional dysphagia or odynoph | agia with solid food or pills duri | ng the past week |
| <ul><li>Dysphagia OR</li><li>Odynophagia</li></ul> | 2=Intermittent dysphagia or odynophagia with solid foods or pills, but not for liquids or soft foods, during the past week | | |
| | 3=Dysphagia or odynophagia for aln | nost all oral intake, on almost ev | ery day of the past week |
| Gastrointestinal-Lower GI | $\theta$ = no loose or liquid stools during th | e past week | |
| • Diarrhea | l = occasional loose or liquid stools, | on some days during the past we | ek |
| | 2=intermittent loose or liquid stools throughout the day, on almost every day of the past week, without requiring intervention to prevent or correct volume depletion | | |
| | 3=voluminous diarrhea on almost ev correct volume depletion | very day of the past week, requir | ing intervention to prevent or |
| Lungs • Bronchiolitis Obliterans | Pulmonary Function Tests with Diffusing Capacity (attach report for person> 5 yrs old) | FEV-1 | Single Breath DLCO (adjusted for hemoglobin) |
| | | (% Predicted) | (%Predicted) |
| Health Care Provider Global Ratings: In your opinion, do you | Where would you rate the sever symptoms on the following scale, we that are not at all severe and 10 | where 0 is CGVHD symptoms | Over the past month would you say that this patient's CGVHD is |
| think that this patient's | symptoms possible: | | +3= Very much better |
| cGvHD is mild, moderate or severe? | | | +2= Moderately better |
| 0=none | 0 1 2 3 4 5 6 | 7 8 9 10 | +1= A little better |
| o none | | | 0= About the same |

| 1= mild<br>2=moderate<br>3=severe | cGvHD symptoms<br>not at all severe | | cGvHD symptoms<br>most severe<br>possible | -1=A little worse<br>-2=Moderately worse<br>-3=Very much worse |
|---|---|---|---|---|
| Karnofsky Performance | Score | Performance Status Scale D<br>16 years old) | efinitions (Use Lansky Pla | y Performance for persons < |
| Able to carry on normal | | | | |
| activity and to work; no special care needed. | 90 | Able to carry on normal activ | Able to carry on normal activity; minor signs or symptoms of disease | |
| | 80 Normal activity with effort; some signs or symptoms of disease | | | |
| Unable to work; able to live at | 70 | Cares for self; unable to carry on normal activity or to do active work | | |
| home and care for most personal needs; varying | 60 | Requires occasional assistance but is able to care for most personal needs | | |
| amount of assistance needed. | 50 | Requires considerable assistance and frequent medical care | | |
| Unable to care for self; | 40 | Disabled; requires special car | e and assistance | |
| requires equivalent of institutional or hospital care; | 30 | Severely disabled; hospital ad | lmission is indicated althou | gh death not imminent |
| disease may be progressing rapidly. | 20 | Very sick; hospital admission necessary; active supportive treatment necessary | | |
| | 10 | Moribund; fatal processes progressing rapidly | | |


## 16.8 APPENDIX H: CALCULATIONS FOR PARTIAL RESPONSE IN CHRONIC GVHD

| Organ and Starting Score or Value at Baseline | Partial Response Criterion <sup>1</sup> |
|---|---|
| Skin (% of BSA) | |
| > 50 | $e/s \le 0.5 \text{ and } e > 0$ |
| 25-50 | $s - e \ge 25$ and $e > 0$ |
| < 25 | Only CR; no PR possible |
| Eye (mm Schirmer's test) | |
| < 5 mm | $e - s \ge 5$ mm and $e < LLN$ |
| 5-10 mm | Only CR; no PR possible |
| Mouth (Schubert Scale 0-15) | |
| > 8 | $e/s \le 0.5$ and $e > 0$ |
| 4-7 | $s - e \ge 4$ and $e > 0$ |
| < 4 | Only CR; no PR possible |
| Hematology | |
| Platelet count | $e-s \ge 100,000/\mu L$ and $e < LLN$ |
| Eosinophil count | |
| ≥3 X ULN | $e/s \le 0.5$ and $e > ULN$ |
| < 3 X ULN | Only CR; no PR possible |
| Gastrointestinal (0 -3 scales) | |
| 3 | e = 1 or 2 |
| 2 | e = 1 |
| 1 | Only CR; no PR possible |
| Liver function | |
| (ALT, alkaline phosphatase and bilirubin) | |
| ≥ 3 X ULN | $e/s \le 0.5$ and $e > ULN$ |
| < 3 X ULN | Only CR; no PR possible |

Abbreviations: s: starting score or value; e: ending score or value; ULN: upper limit of normal; LLN: lower limit of normal


## 16.9 APPENDIX I: CALCULATIONS FOR PROGRESSION IN CHRONIC GVHD

| Organ and Starting Score or Value | Progression Criterion <sup>1</sup> |
|---|---|
| Skin (% of BSA) | $e-s \ge 25$ |
| Eye (mm Schirmer's test) | $s - e \ge 5 \text{ mm}$ |
| Mouth (Schubert Scale 0-15) | $e-s \ge 3$ |
| Hematology Platelet count Eosinophil count | $s-e \geq 50,\!000/\mu L$ and $e < LLN$ |
| $\geq 3 \times \text{ULN}$ | $e - s \ge 3 \times ULN$ |
| < 3 X ULN | e - s ≥ 2 X ULN |
| Gastrointestinal (0 -3 scales) | $e-s \ge 1$ |
| Liver function (ALT, alkaline phosphatase and bilirubin) | 2 V I II N |
| $s \ge 3 \times ULN$ | $e - s \ge 3 \times ULN$ |
| s < 3 X ULN | $e - s \ge 2 X ULN$ |
| Lungs (Lung function scale 12 points) <sup>2</sup> | $e-s \ge 3$ |

<sup>1.</sup> Abbreviations: starting score or value; e: ending score or value; ULN: upper limit of normal; LLN: lower limit of normal

<sup>2.</sup> If the starting lung function score is  $\geq$  10, progression is defined as  $\geq$  5% decrease of FEV1 in two tests measured at least 2 weeks apart.


## 16.10 APPENDIX J: CHRONIC GVHD CUTANEOUS ASSESSMENT WORKSHEET (ADULT)

| | Erythematous changes | | | Moveable-sclerosis/Dermal sclerosis | | | Non-moveable/subcutaneous sclerosis or fasciitis | | |
|---|---|---|---|---|---|---|---|---|---|
| | % region involved | Multiplier | Total<br>BSA | % region involved | Multiplier | Total<br>BSA | % region involved | Multiplier | Total<br>BSA |
| Head/neck/scalp | | 0.09 | | | 0.09 | | | 0.09 | |
| Anterior torso | | 0.18 | | | 0.18 | | | 0.18 | |
| Posterior torso | | 0.18 | | | 0.18 | | | 0.18 | |
| L. upper extrem. | | 0.09 | | | 0.09 | | | 0.09 | |
| R. upper extrem. | | 0.09 | | | 0.09 | | | 0.09 | |
| L. lower extrem. (incl. L. buttock) | | 0.18 | | | 0.18 | | | 0.18 | |
| R. lower extrem. (incl. R. buttock) | | 0.18 | | | 0.18 | | | 0.18 | |
| Genitalia | | 0.01 | | | 0.01 | | | 0.01 | |




## 16.11 APPENDIX K: LEE SYMPTOM SCALE

| | Not at all | Slightly | Moderately | Quite a bit | Extremely |
|---|---|---|---|---|---|
| SKIN: | | | | | |
| a. Abnormal skin color | 0 | 1 | 2 | 3 | 4 |
| b. Rashes | 0 | 1 | 2 | 3 | 4 |
| c. Thickened skin | 0 | 1 | 2 | 3 | 4 |
| d. Sores on skin | 0 | 1 | 2 | 3 | 4 |
| e. Itchy skin | 0 | 1 | 2 | 3 | 4 |
| EYES AND MOUTH: | | | | | |
| f. Dry eyes | 0 | 1 | 2 | 3 | 4 |
| g. Need to use eyedrops frequently | 0 | 1 | 2 | 3 | 4 |
| h. Difficulty seeing clearly | 0 | 1 | 2 | 3 | 4 |
| i. Need to avoid certain foods due to mouth pain | 0 | 1 | 2 | 3 | 4 |
| j. Ulcers in mouth | 0 | 1 | 2 | 3 | 4 |
| k. Receiving nutrition from an intravenous line or feeding tube | 0 | 1 | 2 | 3 | 4 |
| BREATHING: | | | | | |
| 1. Frequent cough | 0 | 1 | 2 | 3 | 4 |
| m. Colored sputum | 0 | 1 | 2 | 3 | 4 |
| n. Shortness of breath with exercise | 0 | 1 | 2 | 3 | 4 |
| o. Shortness of breath at rest | 0 | 1 | 2 | 3 | 4 |
| p. Need to use oxygen | 0 | 1 | 2 | 3 | 4 |
| EATING AND DIGESTION: | | | | | |


| | Not at all | Slightly | Moderately | Quite a bit | Extremely |
|---|---|---|---|---|---|
| q. Difficulty swallowing solid foods | 0 | 1 | 2 | 3 | 4 |
| r. Difficulty swallowing liquids | 0 | 1 | 2 | 3 | 4 |
| s. Vomiting | 0 | 1 | 2 | 3 | 4 |
| t. Weight loss | 0 | 1 | 2 | 3 | 4 |
| MUSCLES AND JOINTS: | | | | | |
| u. Joint and muscle aches | 0 | 1 | 2 | 3 | 4 |
| v. Limited joint movement | 0 | 1 | 2 | 3 | 4 |
| w. Muscle cramps | 0 | 1 | 2 | 3 | 4 |
| x. Weak muscles | 0 | 1 | 2 | 3 | 4 |
| ENERGY: | | | | | |
| y. Loss of energy | 0 | 1 | 2 | 3 | 4 |
| z. Need to sleep more/take naps | 0 | 1 | 2 | 3 | 4 |
| aa. Fevers | 0 | 1 | 2 | 3 | 4 |
| MENTAL AND EMOTIONAL: | | | | | |
| bb. Depression | 0 | 1 | 2 | 3 | 4 |
| cc. Anxiety | 0 | 1 | 2 | 3 | 4 |
| dd. Difficulty sleeping | 0 | 1 | 2 | 3 | 4 |


#### 16.12 APPENDIX L: POMALIDOMIDE PREGNANCY PREVENTION RISK MANAGEMENT PLANS

This Appendix applies to all patients receiving pomalidomide therapy. The following Pregnancy Risk Minimization Plan documents are included in this Appendix:

- 1) Pomalidomide Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods (<u>Appendix M</u>);
- 2) Pomalidomide Information Sheet (Appendix N).
- 1. The Pomalidomide Risks of Fetal Exposure, Pregnancy Testing Guidelines and Acceptable Birth Control Methods document (Appendix M) provides the following information:
  - Potential risks to the fetus associated with pomalidomide exposure
  - Definition of Female of Childbearing Potential (FCBP)
  - Pregnancy testing requirements for patients receiving Pomalidomide who are females of childbearing potential
  - Acceptable birth control methods for both female of childbearing potential and male patients receiving pomalidomide in the study
  - Requirements for counselling of all study patients receiving pomalidomide about pregnancy precautions and the potential risks of fetal exposure to pomalidomide
- 2. The Pomalidomide Information Sheet (<u>Appendix N</u>) will be given to each patient receiving pomalidomide study therapy. The patient must read this document prior to starting pomalidomide study treatment and each time they receive a new supply of study drug.


# 16.13 APPENDIX M: POMALIDOMIDE RISKS OF FETAL EXPOSURE, PREGNANCY TESTING GUIDELINES AND ACCEPTABLE BIRTH CONTROL METHODS

#### **Risks Associated with Pregnancy**

Pomalidomide was found to be teratogenic in a developmental study in rabbits. Pomalidomide is an analogue of thalidomide. Thalidomide is a known human teratogen that causes severe lifethreatening human birth defects. If pomalidomide is taken during pregnancy, it may cause birth defects or death to an unborn baby.

## Criteria for females of childbearing potential (FCBP)

This protocol defines a female of childbearing potential as a sexually mature woman who is menstruating, amenorrheic from previous medical treatments, under 50 years of age and/or perimenopausal and do not qualify for the females not of reproductive potential category.

Criteria for females not of reproductive potential:

Defined as females who have been in natural menopause for at least 24 consecutive months, or who have had a hysterectomy and/or bilateral oophorectomy.

#### Counselling

For a female of childbearing potential, pomalidomide is contraindicated unless all of the following are met (ie, all females of childbearing potential must be counselled concerning the following risks and requirements prior to the start of pomalidomide study therapy):

- She understands the potential teratogenic risk to the unborn child
- She understands the need for effective contraception, without interruption, 28 days before starting study treatment, throughout the entire duration of study treatment, dose interruption and 28 days after the end of study treatment
- She should be capable of complying with effective contraceptive measures
- She is informed and understands the potential consequences of pregnancy and the need to notify her study doctor immediately if there is a risk of pregnancy
- She understands the need to commence the study treatment as soon as study drug is dispensed following a negative pregnancy test
- She understands the need and accepts to undergo pregnancy testing based on the frequency outlined in this protocol (Section 2.2)
- She acknowledges that she understands the hazards and necessary precautions associated with the use of pomalidomide

The investigator must ensure that females of childbearing potential:

- Comply with the conditions for pregnancy risk minimization, including confirmation that she has an adequate level of understanding
- Acknowledge the aforementioned requirements


For a female NOT of childbearing potential, pomalidomide is contraindicated unless all of the following are met (ie, all females NOT of childbearing potential must be counselled concerning the following risks and requirements prior to the start of pomalidomide study therapy):

• She acknowledges that she understands the hazards and necessary precautions associated with the use of pomalidomide

The effect of pomalidomide on spermatogenesis is not known and has not been studied. Therefore, male patients taking pomalidomide must meet the following conditions (ie, all males must be counselled concerning the following risks and requirements prior to the start of pomalidomide study therapy):

- Understand the potential teratogenic risk if engaged in sexual activity with a pregnant female or a female of childbearing potential
- Understand the need for the use of a condom even if he has had a vasectomy, if engaged in sexual activity with a pregnant female or a female of childbearing potential.

#### Contraception

Females of childbearing potential (FCBP) enrolled in this protocol must agree to use two reliable forms of contraception simultaneously or to practice complete abstinence from heterosexual contact during the following time periods related to this study: 1) for at least 28 days before starting study drug; 2) while participating in the study; 3) during dose interruptions; and 4) for at least 28 days after study treatment discontinuation.

The two methods of reliable contraception must include one highly effective method and one additional effective (barrier) method. FCBP must be referred to a qualified provider of contraceptive methods if needed. The following are examples of highly effective and additional effective methods of contraception:

- Highly effective methods:
  - o Intrauterine device (IUD)
  - o Hormonal (birth control pills, injections, implants)
  - Tubal ligation
  - o Partner's vasectomy
- Additional effective methods:
  - Male condom
  - o Diaphragm
  - o Cervical Cap

Because of the increased risk of venous thromboembolism in patients taking pomalidomide and dexamethasone, combined oral contraceptive pills are not recommended. If a patient is currently using combined oral contraception the patient should switch to another one of the effective methods listed above. The risk of venous thromboembolism continues for 4–6 weeks after discontinuing combined oral contraception. The efficacy of contraceptive steroids may be reduced during co-treatment with dexamethasone.


Implants and levonorgestrel-releasing intrauterine systems are associated with an increased risk of infection at the time of insertion and irregular vaginal bleeding. Prophylactic antibiotics should be considered particularly in patients with neutropenia.

#### Pregnancy testing

Medically supervised pregnancy tests with a minimum sensitivity of 25 mIU/mL must be performed for females of childbearing potential, including females of childbearing potential who commit to complete abstinence, as outlined below.

#### Before starting study drug

#### Female Patients:

FCBP must have two negative pregnancy tests (sensitivity of at least 25 mIU/mL) prior to starting study drug. The first pregnancy test must be performed within 10-14 days prior to the start of study drug and the second pregnancy test must be performed within 24 hours prior to the start of study drug. The patient may not receive study drug until the study doctor has verified that the results of these pregnancy tests are negative.

#### Male Patients:

Must practice complete abstinence or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for at least 28 days following study drug discontinuation, even if he has undergone a successful vasectomy.

#### During study participation and for 28 days following study drug discontinuation

#### Female Patients:

- FCBP with regular or no menstrual cycles must agree to have pregnancy tests weekly for the first 28 days of study participation and then every 28 days while on study, at study discontinuation, and at day 28 following study drug discontinuation. If menstrual cycles are irregular, the pregnancy testing must occur weekly for the first 28 days and then every 14 days while on study, at study discontinuation, and at days 14 and 28 following study drug discontinuation.
- At each visit, the Investigator must confirm with the FCBP that she is continuing to use two reliable methods of birth control.
- Counselling about pregnancy precautions and the potential risks of fetal exposure must be conducted at a minimum of every 28 days.
- If pregnancy or a positive pregnancy test does occur in a study patient, study drug must be immediately discontinued.
- Pregnancy testing and counselling must be performed if a patient misses her period or if her pregnancy test or her menstrual bleeding is abnormal. Study drug treatment must be discontinued during this evaluation.
- Females must agree to abstain from breastfeeding during study participation and for at least 28 days after study drug discontinuation.


#### Male Patients:

• Counselling about the requirement for complete abstinence or condom use during sexual contact with a pregnant female or a female of childbearing potential and the potential risks of fetal exposure to pomalidomide must be conducted at a minimum of every 28 days.

• If pregnancy or a positive pregnancy test does occur in the partner of a male study patient during study participation, the investigator must be notified immediately.

## Additional precautions

- Patients should be instructed never to give this medicinal product to another person and to return any unused capsules to the study doctor at the end of treatment.
- Patients should not donate blood during therapy and for at least 28 days following discontinuation of study drug.
- Male patients should not donate semen or sperm during therapy or for at least 28 days following discontinuation of study drug.
- Only enough study drug for one cycle of therapy may be dispensed with each cycle of therapy.


#### 16.14 APPENDIX N: POMALIDOMIDE INFORMATION SHEET

#### FOR PATIENTS ENROLLED IN CLINICAL RESEARCH STUDIES

Please read this Pomalidomide Information Sheet before you start taking study drug and each time you get a new supply. This Pomalidomide Information Sheet does not take the place of an informed consent to participate in clinical research or talking to your study doctor or healthcare provider about your medical condition or your treatment.

### What is the most important information I should know about pomalidomide?

- 1. Pomalidomide may cause birth defects (deformed babies) or death of an unborn baby. Pomalidomide is similar to the medicine thalidomide. It is known that thalidomide causes life-threatening birth defects. Pomalidomide has not been tested in pregnant women but may also cause birth defects. Pomalidomide was found to cause birth defects when tested in pregnant rabbits. If you are a female who is able to become pregnant:
  - Do not take study drug if you are pregnant or plan to become pregnant
  - You must either not have any sexual relations with a man or use two reliable, separate forms of effective birth control at the same time:
    - o for 28 days before starting study drug
    - o while taking study drug
    - o during dose interruptions of study drug
    - o for 28 days after stopping study drug
  - You must have pregnancy testing done at the following times:
    - $\circ$  within 10 14 days and again 24 hours prior to the first dose of study drug
    - o weekly for the first 28 days
    - o every 28 days after the first month or every 14 days if you have irregular menstrual periods
    - o if you miss your period or have unusual menstrual bleeding
    - 28 days after the last dose of study drug (14 and 28 days after the last dose if menstrual periods are irregular)
    - o at discontinuation of study drug
  - Stop taking study drug if you become pregnant during treatment
    - o If you suspect you are pregnant at any time during the study, you must stop study drug immediately and immediately inform your study doctor. The study doctor will report all cases of pregnancy to Celgene Corporation.
  - Do not breastfeed while taking study drug
  - The study doctor will be able to advise you where to get additional advice on contraception.


#### If you are a female not of childbearing potential:

In order to ensure that an unborn baby is not exposed to pomalidomide, your study doctor will confirm that you are not able to become pregnant.

#### If you are a male:

The effect of pomalidomide on sperm development is not known and has not been studied. The risk to the fetus in females of child bearing potential whose male partner is receiving pomalidomide is unknown at this time.

- 1. Male patients (including those who have had a vasectomy) must either **not** have any sexual relations with a pregnant female or a female who can become pregnant, or must use a condom during sexual contact with a pregnant female or a female that can become pregnant:
  - o While you are taking study drug
  - o During dose interruptions of study drug
  - o For 28 days after you stop taking study drug
- 2. **Male patients should not donate sperm or semen** while taking study drug and for 28 days after stopping study drug.
- 3. If you suspect that your partner is pregnant any time during the study, you must immediately inform your study doctor. The study doctor will report all cases of pregnancy to Celgene Corporation. Your partner should call their healthcare provider immediately if they get pregnant.
- 2. Restrictions in sharing study drug and donating blood:
  - 1. Do not share study drug with other people. It must be kept out of the reach of children and should never be given to any other person.
  - **2. Do not donate blood** while you take study drug and for 28 days after stopping study drug.
  - 3. Do not break, chew, or open study drug capsules.
  - 4. You will be supplied with no more than one cycle of study drug
  - **5.** Return unused study drug capsules to your study doctor.

Additional information is provided in the informed consent form and you can ask your study doctor for more information.


## 16.15 APPENDIX O: MEDICATION DIARY

| Today's date |
|--------------|
|--------------|

| Patie | nt | | Name | | | | Patient Study |
|---|---|---|---|---|---|---|---|
| ID_ | | | | • | CTION | S TO TH | E PATIENT: |
| 1.<br>2.<br>3. | Complete one form for each cycle. You will take your dose of pomalidomide each day at approximately the same time. Pomalidomide capsules should be swallowed whole, and should not be broken, chewed or opened. Caregivers who are women able to become pregnant should not handle pomalidomide unless wearing gloves. You will take0.5 mg capsules,1 mg capsules and2 mg capsules each day. Record the date, the number of capsules of each size you took, and when you took them. | | | | | | |
| 4.<br>5. | | | | | | | blease record them in the Comments column. |
| <u> </u> | Time of # of capsules taken | | | ician when you go for your next appointment. | | | |
| Date | | Day | daily dose | 0.5<br>mg | 1 mg | 2 mg | Comments |
| | | 1 | | | | | |
| | | 2 | | | | | |
| | | 3 | | | | | |
| | | 4 | | | | | |
| | | 5 | | | | | |
| | | 6 | | | | | |
| | | 7 | | | | | |
| | | 8 | | | | | |
| | | 9 | | | | | |
| | | 10 | | | | | |
| | | 11 | | | | | |
| | | 12 | | | | | |
| | | 13 | | | | | |
| | | 14 | | | | | |

Abbreviated Title: Pomalidomide for cGvHD **Version Date:** 4/29/2025 Patient Name Patient Study ID (initials acceptable) INSTRUCTIONS TO THE PATIENT: 1. Complete one form for each cycle. 2. You will take your dose of pomalidomide each day at approximately the same time. Pomalidomide capsules should be swallowed whole, and should not be broken, chewed or opened. Caregivers who are women able to become pregnant should not handle pomalidomide unless wearing gloves. You will take \_\_\_\_\_0.5 mg capsules, \_\_\_\_\_1 mg capsules and \_\_\_\_\_2 mg capsules each day. 3. Record the date, the number of capsules of each size you took, and when you took them. 4. If you have any comments or notice any side effects, please record them in the Comments column. 5. Please bring your pill bottle and this form to your physician when you go for your next appointment. Time # of capsules taken of daily dose **Comments Date** Da 0.5 1 mg 2 mg y mg 15 16 17 18 19 20 21 22 23 24 25 26

| | 27 | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | 28 | | | | | | | | | |
| Patient's | S | ignature: | | | | | | | | Date: |
| Physician's | Office | will complet | e this sec | ction: | | | | | | |
| 1. Date p | atient | started prote | ocol trea | tment | <br>_ Date | patient | was | removed | from | study |


| 2. Patient's planned daily dose | Total number | er of pills | taken th | nis month |
|---|---|---|---|---|
| Physician/Nurse/Data | Manager's | | | Signature |


#### 16.16 APPENDIX P: DATA COLLECTION ELEMENTS REQUIRED BY PROTOCOL

ALL OF THE FOLLOWING ELEMENTS WILL BE RECORDED IN THE C3D DATABASE.

#### A. PATIENT ENROLLMENT

#### **Recipient**

- Date of birth, age, sex, race, ethnicity
- Height
- Weight
- Karnofsky Performance Status
- Date of original diagnosis of the underlying disease (month/year)
- Diagnosis for which transplant was performed
- Date and type of transplant
- Conditioning regimen
- Acute GVHD yes/no
- Chronic GVHD date of diagnosis
- Chronic GVHD classification (late, overlap, classic)
- Prior systemic therapy for cGVHD
- Prior therapy for cGVHD
- Date of Informed Consent signature, consent version and date of registration
- Baseline History/Physical
- Baseline Symptoms
- Intensity of current immunosupression: None, Mild (single agent prednisone ≤0.5 mg/kg/day), Moderate (prednisone ≥0.5 mg/kg/day and or any single agent/modality), High (2 or more agents/modalities +prednisone >0.5 mg/kg/day)
- Clinician's impression of activity: Inactive, off systemic therapy or topical immunosupression; Inactive, on systemic therapy or topical immunosupression; Active, irrespective of the level of current therapy; Highly Active, irrespective of the level of current therapy
- Findings of consultations done at screening

#### Donor

- Age at transplant
- Relationship, sex
- Degree and type of HLA match (allele or serologic)
- CMV status


# B. STUDY DRUG ADMINISTRATION AND RESPONSE FOR EACH COURSE OF THERAPY GIVEN

- Dates study drug given
- Actual dose given
- Response assessment

#### C. LABORATORY AND DIAGNOSTIC TEST DATA

- All Clinical laboratory and diagnostic test results done at screening except diagnostic tests which are not specified in the protocol, and if the results are not needed to document the start or end of an adverse event that requires reporting.
- All tests done to document resolution of adverse events
- Serologies-CMV and HSV

#### D. ADVERSE EVENTS

- All unexpected serious adverse events that are possibly, probably, or definitely related to the research
- All deaths, except deaths due to progressive disease
- All Protocol Violations or Deviations
- All Unanticipated Problems

#### E. CONCOMITANT MEASURES

- Baseline immunosuppresive medications
- Other therapy for recorded adverse events

#### F. Off study

- Date and reason for off study
- Date and cause of death
- Autopsy findings


#### 16.17 APPENDIX Q:CHRONIC GVHD COMPOSITE ASSESSMENT SCALE – EVALUATION TOOLS

### 16.17.1Component 1: Skin

| Patient Name: | Patient MR #: |
|---------------------|---------------|
| Date of Assessment: | |

#### 1. CAS - Initial assessment

- a. Extent (% body surface area, BSA) of involvement are estimated for lichenoid, sclerotic, and fascial disease.
- b. A score 0-3 (none, mild, moderate, severe) are given that directly correlates with BSA affected (see table below)
- c. The highest score in any skin sub-type are used to determine the overall stage of involvement

## • Check appropriate box in each row

| Sub-type | Norma | l=0 | MILD=1 | MILD=1 | MILD=1 | MODERAT | E=2 | SEVERE=3 |
|---|---|---|---|---|---|---|---|---|
| Erythema /<br>Lichenoid | 0 | | 1-25%<br>BSA | 25<br>50%BSA | 3 = > 50% BSA | | | |
| Sclerosis,<br>movable | 0 | | 1-25%<br>BSA | 25<br>50%BSA | 3 = > 50% BSA | | | |
| Sclerosis, fixed (fasciitis) | 0 | | 1-25%<br>BSA | 25 –<br>50%BSA | 3 = > 50% BSA | | | |

| Overall stage (max 3): | | |
|------------------------|--------------|-----------|
| Signature | Printed Name | Date/Time |

2. Not in CAS - Objective ancillary data (presence or absence)


| Pigment a<br>(% | | | ions/<br>ations | Nail dy | strophy | Alop | oecia | Ede | ema | Xe | rosis |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Present | Absent | Presen | Absent | Presen | Absent | Presen | Absent | Presen | Absent | Presen | Absent |
| | | t | | t | | t | | t | | t | |
| % | | | | | | | | | | | |

3. Not in CAS - Subjective assessments --- Patient Visual Analog Scales

Pain

O

Itching

O

10



**Definitions:** 

Pain due to <u>skin</u> disease from zero (no pain) to 10 (worst imaginable pain) Itching is level of discomfort from itching from zero (no itching) to 10 (worst imaginable itching)

10

Clinical severity is patient's assessment of degree of disease activity on the skin

| Pain<br>(0-10) | Pruritus<br>(0-10) | Clinical severity (0-10) | |
|---|---|---|---|
| | | Patient | Physician |

| Date of bx | Clinical findings | Group received | Location<br>of bx | Affected/<br>Unaffected | Bx<br>reason<br>(D, R,<br>D/R)* |
|---|---|---|---|---|---|

| *D- Diagnostic; R-R | esearch, D/R- Diagnostic/Research | 1 |
|---------------------|-----------------------------------|---------------|
| Signature | Printed Name | <br>Date/Time |


## 16.17.2Component 2: Mouth

1. <u>CAS – Initial assessment</u>

• Please, check off the box.

| Instrument | Clinical Sign or<br>Symptom | Nor | mal=0 | Mil | d=1 | Modera | ate=2 | Severe | =3 |
|---|---|---|---|---|---|---|---|---|---|
| Oral<br>Mucositis | Oral signs of cGVHD | 0 | | 1 to 34 | | 35-69 | | 70-103+ | |
| Rating Scale (CAS) | | | | | | | | | |

| OMRS | S Score: | | |
|--------|------------------------------------|------------------|----------|
| Stage: | | | |
| 2. | Biopsy of oral mucosa (please chee | ck off the box): | |
| A. | Research Biopsy (Dr. Hakim's lab) | □ YES □NO | Size(mm) |
| B. | Clinical Biopsy (Pathology) | □ YES □NO | Size(mm) |
| C. | Minor Salivary Gland | □ YES □NO | |
| 3. | Amount of saliva collected in 5 mi | <u>n</u> : | |
| Date: | /LIP print name: _ | | |
| I IP | Signatur | ٠۵٠ | |

| <b>Version Da</b> | te: 4/29/2025 |
|-------------------|---------------|
|-------------------|---------------|

| Schube | rt Oral Mucositis R | atin | g Scale | 9 | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | //LII | | | | | | | | | _LIP_ | | |
| | UCTIONS: Assess e | | | | | | | | | stated | clinical | |
| | | | | J | LIPS | | | ABIA<br>COS | | | BUCC<br>MUCO | |
| | | | Lowe | r | Upp | oer | Low | ver | Upp | er | Right | Left |
| | Atrophy | | | | | | | | | | | |
| | Pseudomembrane | : | | | | | | | | | | |
| | Erythema | | | | | | | | | | | |
| | Hyperkeratosis | | | | | | | | | | | |
| | Lichenoid | | | | | | | | | | | |
| | Ulceration | | | | | | | | | | | |
| | <b>Edema/Cellulitis</b> | | | | | | | | | | | |
| | | | | T | ONG | UE | | FLO<br>OF | OOR | PA | LATE | GINGIVA |
| | | D | orsal | T . | ater | Vor | ıtral | _ | OUT | Har | Soft | |
| | | יע | JI SAI | al | | V CI | iti ai | H | 701 | d | Soit | |
| | Atrophy | | | | | | | | | | | |
| | Pseudomembran<br>e | | | | | | | | | | | |
| | Erythema | | | | | | | | | | | |
| | Hyperkeratosis | | | | | | | | | | | |
| | Lichenoid | | | | | | | | | | | |
| | Ulceration | | | | | | | | | | | |
| | <b>Edema/Cellulitis</b> | | | | | | | | | | | |
| Instruc | tions for Rating: | su | m all it | ems | | otal ( | OMRS | S Sco | ore: _ | | (range: | 0 – 273; |
| _ | y, erythema, hyperk<br>eudomembrane | kera | tosis, li | iche | enoid, | and | edema | ì | | | Ulcera | ation |
| Change | e is rated from norm | al. | | | | | | | | | | |
| $0 = N_0$ | ormal/No change | | | | | | | | 0 | = Non | e | |
| 1 = M | ild change | | | | | | | | | | out ≤ 1cm | |
| 2 = M | oderate change | | | | | | | | 2 | = >1 c | $m^2$ but $\leq$ | 2 cm <sup>2</sup> |
| 3 = Se | vere change | | | | | | | | 3 | =>2c | $m^2$ | |

| If an | y area cannot be | assesse | d, circle one | of the follow | ing: | | | |
|---|---|---|---|---|---|---|---|---|
| | Unable to visual | lize/asse | ess due to se | verity | 09 = | = Un | able to ass | ess because |
| - | ent is | | | | | | | |
| 05 = | Unable to assess | s becaus | se patient is | sedated | edated not | | available. | Explain: |
| 06 | =Unable | to | assess | because | pat | tient | is | disoriented |
| 07 = | Unable to assess | becaus | se patient is | comatose | 10 | = | Other. | Explain: |
| 08 = | Unable to assess | | se patient is | unwilling | | 99 = | - Missing | |
| | ck (√) type of lig | • | ce used to vi | isualize the o | ral cavit | y: | | (1) |
| | water rinse used | | | | <b>(2)</b> | | | (0) |
| | (1) Otoscope | | Dental Ligh | nt | _ (3) ( | <b>Ither</b> | | (2) |
| Loca | al anesthetic used | | | | | | | |
| | es: Patient asked<br>ne to 10= worst): | to rate | oral pain us | ing the Paino | ometer a | nd to | rate dryness | s verbally (0 |
| 110 | Oral pain: | | | | | | | |
| | Pain on swallo | wing - | | | | | | |
| | Dryness in mo | uth | | | | | | |
| | Dryness in thro | oat: | | | | | | |
| Mou | th Opening: | | mm | | | | | |

LIP print name:

Qualitative change of

the gingival soft

tissues


Gingival Index

(Harald Löe)

Date:

| Instrument | Variable Assessed | Mild | Moderate | Severe |
|---|---|---|---|---|
| | | Inflammation=0 | Inflammation=1 | Inflammation= |
| | | .1-1.0 | .1-2.0 | 2.1-3.0 |

LIP Signature:

| Instrument | Variable Assessed | Excellent<br>Plaque<br>Control=0 | Good<br>Plaque<br>Control=0.1<br>-0.9 | Fair Plaque<br>Control=1.0<br>-1.9 | Poor Plaque<br>Control=2.0-<br>3.0 |
|---|---|---|---|---|---|
| Plaque Index<br>(Silness and Löe) | The severity and location of the soft debris aggregates | | | | |

## Instructions: Gingival Index

Upon palpation of the gingiva and running a blunt instrument (periodontal probe) along the soft tissue wall of the entrance of the gingival crevice the gingiva is examined and categorized the following way:

GI=0: is the score given to the gingiva the color of which is pale pink to pink. The surface after drying is matt. The degree of stippling may vary. The gingival margin may be located on the enamel or at various levels apical to the cemento-enamel junction. Although the margin should be thin, the buccal and lingual gingiva may present a rounded termination against the tooth, thereby forming the entrance or orifice of the gingival crevice. The form of the interdental gingiva depends on the space and size of the interdental areas. The tip of the papilla should be the most incisally or occlusally located part of the gingiva. On palpation, the gingival should be firm.

GI=1: is the score given when the gingiva is subject to mild inflammation. The gingival margin is slightly more reddish or bluish-reddish than normal and there is slight edema of the margin. A colorless gingival exudate may be observed or collected at the entrance of the crevice. Bleeding is not provoked.

GI=2: This is the score for a moderately inflamed gingiva. The gingiva is red or reddish-blue and glazy. There is enlargement of the margin due to edema. Bleeding is provoked.

GI=3: is the score for severe inflammation. The gingiva is markedly red or reddish-blue and enlarged. There is a tendency to spontaneous bleeding. Ulceration may be seen.

#### Plaque Index

PI=0: This score is given when the gingival area of the tooth surface is literally free of plaque. The surface is tested by running a pointed probe across the tooth surface at the entrance of the gingival crevice after the tooth has been properly dried, and if no soft matter adheres to the point of the probe, the area is considered clean.


PI=1: This score is given when no plaque can be observed in situ by the unarmed eye, but when the plaque is made visible on the point of the probe after this has been moved across the tooth surface at the entrance of the gingival crevice.

PI=2: This score is given when the gingival area is covered with a thin to moderately thick layer of plaque. The deposit is visible to the naked eye.

PI=3: Heavy accumulation of soft matter, the thickness of which fills out the niche produced by the gingival margin and the tooth surface. The interdental area is stuffed with soft debris.

Scoring For both indices, scores are given for distal, buccal, mesial and lingual surfaces. The

**Scoring** For both indices, scores are given for distal, buccal, mesial and lingual surfaces. The scores are added together and divided by the number of surfaces scored (4), and then divided by the number of teeth scored (6). This is your Gingival Index or Plaque Index score.

#### VISUAL ANALOG SCALE FOR XEROSTOMIA

| | , ' |
|-----------------------------------------------|--------------------|
| e the difficulty you experience in swallowing | ng due to dryness. |
| Not difficult at all | Very difficult |
| e the dryness of your mouth. | |
| Not dry at all | Very dry |

Date: \_\_\_/\_\_\_ LIP print name: \_\_\_\_\_\_LIP Signature: \_\_\_\_

NUMERIC RATING SCALES (0-10) FOR ORAL PAIN, SENSITIVITY, AND DRYNESS **ORAL PAIN/SENSITIVITY** On a 0 to 10 scale, how SENSITIVE or PAINFUL was your mouth at its WORST in the past month? Please circle the number. 0 1 2 5 6 7 9 8 10 No sensitivity Worst sensitivity **ORAL DRYNESS** On a 0 to 10 scale, how DRY is your mouth at its WORST in the past month? Please circle the number. 0 1 2 3 5 6 7 8 9 4 10 No dryness Worst dryness Global Scale Compared to one month ago, what is the overall condition of your mouth? Please circle. A little worse A little better Much worse Same Much better LIP Print Name: \_\_\_\_\_LIP Signature: \_\_\_\_\_

Abbreviated Title: Pomalidomide for cGvHD


Date of Evaluation:\_\_\_\_\_


| ORAL HEALTH I | MPACT PROFILE (C | )HIP-14) | |
|---------------|------------------|----------|-----|
| Date://_ | LIP print name:_ | • | LIP |
| Signature: | | | |

| # | Because of problems with your teeth, denture or mouth have you | Never (0) | Hardly<br>ever (1) | Occasionally (2) | Often (3) | Very<br>Often<br>(4) |
|---|---|---|---|---|---|---|
| 1 | Had trouble pronouncing words | | | | | |
| 2 | Felt sense of taste has worsened | | | | | |
| 3 | Had painful aching in the mouth | | | | | |
| 4 | Found it uncomfortable to eat any foods | | | | | |
| 5 | Have been self-conscious | | | | | |
| 6 | Felt tense | | | | | |
| 7 | Had an unsatisfactory diet | | | | | |
| 8 | Had to interrupt meals | | | | | |
| 9 | Found it difficult to relax | | | | | |
| 10 | Have been a bit embarrassed | | | | | |
| 11 | Have been irritable with other people | | | | | |
| 12 | Had difficulty doing usual jobs | | | | | |
| 13 | Felt life in general was less satisfying | | | | | |
| 14 | Have been totally unable to function | | | | | |

| Total |
|-------|


16.17.3Component 3: Vaginal/Vulvar

16.17.3.1 Vaginal/Vulvar-Initial assessment form

Note: patient won't be referred if less than 16

| Patient Name: | Patient MR #: |
|---------------|---------------|

Date of Assessment: \_\_\_\_\_

#### 1. CAS – Initial assessment

Please, check all boxes that pertain

| NORMAL=0 | MILD=1 | MODERATE=2 | SEVERE=3 | |
|---|---|---|---|--|
| Vulva OR Vagina | Vulva | Vulva | Severe Vulva OR Vagina | |
| No symptoms | Erythema around openings of vestibular glands OR | Erosions on flat surfaces most notable on vulva OR | Vulvar architectural changes such as nearly complete resorption of the labia minora and clitoral agglutination OR | |
| | Generalized erythema / edema of vulva including vestibule OR | Fissures in vulvar folds (e.g. interlabial sulci; fourchette) OR | Vaginal synechiae including shortened vagina OR | |
| | Periurethral or other patchy erythema OR | Increased friability of vulvar mucosa | Hematocolpos OR | |
| NORMAL=0 | MILD=1 | MODERATE=2 | SEVERE=3 |
|---|---|---|---|
| | Leukokeratosis<br>(r/o HPV) | | Introital stenosis OR |
| | | | Myofascial pain/spasm of levator or pelvic floor muscles |

| | muscl |
|----------------------------------------------------------------------|-------|
| Overall stage (determined by most severe finding): | |
| 2. Not in CAS – Gynecologic history | |
| Reason for BMT:: | |
| Type of BMT: | |
| Date(s) of BMT: | |
| Current immunosuppressive medications: | |
| 3. Menstrual history: How old were you when you first had a period? | |
| Were your periods regular before you had your BMT? Yes/No | |
| Are you still getting periods? Yes/No | |
| When was your last menstrual period? | |

| Did ' | your BMT | or other | treatment affect | your periods? | Yes/No |
|-------|----------|----------|------------------|---------------|--------|
|-------|----------|----------|------------------|---------------|--------|

| - | |
|-------------------------|----------------------------------|
| If yes, how? Less f | Frequent/ More frequent/ Stopped |
| Describe | |
| 4. Hormone use: | |
| Did you use hormones as | fter your BMT? Yes/No |
| If yes, which ones (C | heck all that apply) |
| 5. Combined horm | nones |
| Birth control pills: | Yes / No Dates: |
| Prempro: | Yes / No Dates: |
| Estradiol/prog (FemHR7 | Γ) Yes / No Dates: |
| | Yes / No Dates: |
| Other: | Dates: |
| 6. Menopausal hor | rmones – estrogens: |
| Estrogen oral pill: | Yes/No Dates: |
| Estrogen topical cream: | Yes/No Dates: |
| Estrogen vaginal pill: | Yes/No Dates: |
| Estrogen patch: | Yes/No Dates: |
| Estrogen ring: | Yes/No Dates: |
| Other: | Dates: |
| 7. Menopausal hor | rmones – progesterone: |
| Progesterone: | Yes/No Dates: |
| Provera: | Yes/No Dates: |
| Other: | Dates: |

| <b>Abbreviated Title:</b> Pomalidomide for cGvHD <b>Version Date:</b> 4/29/2025 | |
|---|---|
| Are you currently taking hormones? Yes/No | |
| Specify | |
| Any contraindications to hormone use? Yes/No | |
| Specify | |
| 8. Gynecologic surgery history: | |
| Have you ever had gynecology surgery? Yes/No | |
| Specify what surgery and year | _ |
| Do you still have a uterus? Yes/No | |
| Do you still have your ovaries? Yes/No | |
| 9. Pap smear history: | |
| Have you ever had an abnormal pap? Yes/No; if yes, when? | |
| What was done? | |
| When was your last pap smear? | |
| Was it normal or abnormal? | |
| 10. STD history: | |
| Have you ever been told you have had any of the following? | |
| Chlamydia: Yes/No | |
| Gonorrhea: Yes/No | |
| Genital herpes: Yes/No | |

Warts or HPV: Yes/No


Dysplasia: Yes/No

### 11. Obstetric history:

Have you ever been pregnant? Yes/No How many times?

### 12. Sexual history:

Have you ever been sexually active? Yes/No

Are you sexually active currently? Yes/No

Have you had intercourse since your transplant? Yes/No

Describe \_\_\_\_\_

#### 13. Not in CAS - Questions addressing pain when the vulva is touched

Do you have pain when nothing is touching the vulva? Yes/No

Do you have vulvar pain or burning when you urinate? Yes/No

If yes, is this when the urine touches the vulva? Yes/No

If yes, does the pain makes you want to urinate? Yes/No

Do you have vulvar pain or burning when you:

Insert a tampon: Yes/No/NA

Wear tight jeans or pants: Yes/No/NA

When you ride a bike: Yes/No/NA

During foreplay: Yes/No/NA

When the penis touches the vulva: Yes/No/NA

Does the vulvar pain prevent or interrupt intercourse? Yes/No/NA

Do you have pain with deep penetration of the penis? Yes/No/NA

Have you been told there is scarring in the vagina? Yes/No/NA

| <b>Abbreviated Title:</b> Pomalidomide for cGvHD <b>Version Date:</b> 4/29/2025 | | |
|---|---|---|
| Do you think there is scarring in the vagina? | | Yes/No/unknown |
| Signature | Printed Name | Date |


## 16.17.3.2 Vaginal/Vulvar-follow-up form

## 1. **CAS – Initial assessment**

• Please check all boxes that pertain

| NORMAL=0 | MILD=1 | MODERATE=2 | SEVERE=3 |
|---|---|---|---|
| Vulva OR Vagina | Vulva | Vulva | Severe Vulva OR Vagina |
| No symptoms | Erythema around openings of vestibular glands OR | Erosions on flat surfaces most notable on vulva OR | Vulvar architectural changes such as nearly complete resorption of the labia minora and clitoral agglutination OR |
| | Generalized erythema / edema of vulva including vestibule OR | Fissures in vulvar folds (e.g. interlabial sulci; fourchette) OR | Vaginal synechiae including shortened vagina OR |
| | Periurethral or other patchy erythema <u>OR</u> | Increased<br>friability of<br>vulvar mucosa | Hematocolpos OR |
| | Leukokeratosis (r/o HPV) | | Introital stenosis OR |
| | | | Myofascial pain/spasm of levator or pelvic floor muscles |

Overall stage (determined by most severe finding):

| Version Date: 4/29/2025 | V۵ | ersion | Date: | 4/29/2025 |
|-------------------------|----|--------|-------|-----------|
|-------------------------|----|--------|-------|-----------|

| Current systemic immunosuppressive medications_ | |
|---|---|
| Have you used topical temovate on the vulva | a since your last visit? Yes / No |
| Describe use and effect | |
| Have you used hormone therapy since your limits. | ast visit? Yes / No |
| Specify | |
| Describe use and effect | |
| Pap smear: | |
| When was your last pap smear? | |
| Was it normal or abnormal? | |
| Sexual history: | |
| | st visit? Yes / No |
| Have you been sexually active since your last | VISIC. TOSTINO |
| • If yes, was it painful? | Yes / No |
| | Yes / No<br>Yes / No |

Do you have vulvar pain or burning when you urinate? Yes / No/ NA

If yes, is this when the urine touches the vulva? Yes / No/ NA If yes, does the pain makes you want to urinate? Yes / No/ NA Do you have vulvar pain or burning when you: • Wear tight jeans or pants: Yes / No/ NA • When you ride a bike: Yes / No/ NA • During foreplay: Yes / No / NA • When the penis touches the vulva: Yes / No/ NA Since the last visit: • Does the vulvar pain prevent or interrupt intercourse? Yes / No/ NA • Do you have pain with deep penetration of the penis? Yes / No/ NA • Have you been told there is scarring in the vagina? Yes / No/ NA • Do you think there is scarring in the vagina? Yes / No/ unknown RECOMMENDATIONS:

Printed Name

Date

Abbreviated Title: Pomalidomide for cGvHD


Signature


#### 16.17.4 Component 3: Function

#### **Description**

There are standard ranges for all tests. Every joint has an established range of motion (ROM). For example, the normal ROM for shoulder flexion is 180 degrees, each quartile is 45 degrees. If the shoulder can be put through 125 degrees it is 75% of normal. Similar is for grip strength (in Kg or pounds of pressure) and for walk time. The velocity is established based on norms for age and sex. For example if 18 feet/second, if divided by 4 and gets quartiles.

| Patient Name: | Patient MR #: |
|---------------------------------|---------------|
| Date of Assessment: | |
| Assessed: Yes/No | |
| Assessed Partially: Yes/No | |
| Reason if "No": age restriction | |

#### 1. CAS – Initial Assessment

PLEASE ASSESS in according to age restrictions for each parameter

• Please, check off the appropriate box

| | Musculoskeletal findings | | | |
|---|---|---|---|---|
| Parameter | NORMAL=0 | MILD=1 | MODERATE=2 | SEVERE=3 |
| ROM* Assess if patient ≥ 4 | 0-25% | 26-50% | 51-75% | >75% |
| grip strength* Assess if patient $\geq 6$ | 0-25% | 26-50% | 51-75% | I. 75% |
| walk velocity* Assess if patient ≥ 6 | 0-25% | 26-50% | 51-75% | II. > 75% |
| HAP* Assess if patient ≥ 16 | >81 | 73-81 | 61-72 | <61 |

\* Reduction in maximal performance Overall stage (max3): Total score (max 12): **Actual Number\*\*** % of predicted\*\*\* Parameter ROM Trial 2 Trial 1 grip strength Trial 3 Average Right Dominant Hand Left R Circle One walk velocity Total Distance Walked in 2 Minutes: feet walked in 2 minutes feet walked in 6 minutes HAP MAS AAS \*\* Please provide the actual result of reduction in maximal performance \*\*\* Please provide the actual result as % of predicted

Printed Name

Date

Abbreviated Title: Pomalidomide for cGvHD


Signature

## 2. P-ROM



## 3. Occupational Therapy

| 1. CAS outcome measures: Dx: | | |
|-----------------------------------------|-----------------------|---------|
| Date of transplant: | | |
| Date of evaluation: Timepoint: | | |
| Instrumental Activities of Daily Living | g: | |
| Frenchay Activities Index: | | |
| Activity Card Sort: | | |
| Basic Self Care: | | |
| Barthel Index: | | |
| Motor Function: | | |
| Disabilities of the Arm Hand and Sho | oulder (DASH) score : | |
| Manual Abilities Measure: | | |
| Grooved Peg board | | |
| 1. Total time dominant hand: | | seconds |
| 2. Total time non dominant hand:_ | | seconds |
| Recommendations: | | |
| Date of Evaluation: | _LIP | |
| Signature: | /phone::301-451-7502 | |

## 2. Manual Ability Measure (MAM-36)

| Patient ID: | | Today's Date: |
|---|---|---|
| Age: | Sex: | Highest Level of Education: |
| Race<br>know) | (White, African | n American, American Indian, Asian-Pacific, Mixed Races, Don't |
| Are you Hi | spanic? | _Yes,No |
| Are you cu | rrently employe | ed? If so, what is your occupation Gob title)? |
| If not, what | t was your occu | apation before you were diagnosed with your current condition? |
| What is yo | ur diagnosis for | coming to the clinic? |
| How long a | ago were you di | iagnosed with this condition? |
| Do you hav | e any other me | edical problems that affect the use of your hands? |
| | had hand surge<br>what was/will | ery, or if you have surgery scheduled, please indicate the be done: |
| • | our dominant ha | and?<br>, Ambidextrous, Don't know |
| Which hand | d(s) has limited | function or hand use? Both_, Right_, Left, |
| Do you live<br>Yes | e alone now? | |


#### **INSTRUCTIONS:**

Please circle one response regarding how easy or how hard it is for you to perform the following tasks.

Easy (4) = I can do the activity without any problem.

A little hard (3) = I usually do the task myself, although it takes longer or more effort now than before (i.e., before having current diagnosis/condition/disability). Sometimes, there is pain or discomfort when I do the task.

Very hard (2) = It is very hard for me to do the task and I usually ask others to do it for me unless no one is around.

Cannot do (1) =I am unable to do the task all by myself.

Almost Never do (0) = I have not done and almost will never do the task, even though I think I can do it.

| Task | Easy | A little hard | Very hard | Cannot do | Never do |
|---|---|---|---|---|---|
| Eat a sandwich | 4 | 3 | 2 | 1 | 0 |
| Drink a glass of water | 4 | 3 | 2 | 1 | 0 |
| Pick up a half-full water pitcher | 4 | 3 | 2 | 1 | 0 |
| Use a spoon or fork | 4 | 3 | 2 | 1 | 0 |
| Butter bread (Put butter or jam on | 4 | 3 | 2 | 1 | 0 |
| Cut meat on a plate with a knife | 4 | 3 | 2 | 1 | 0 |
| Squeeze toothpaste | 4 | 3 | 2 | 1 | 0 |
| Brush teeth : | 4 | 3 | 2 | 1 | 0 |
| Brush or comb hair | 4 | 3 | 2 | 1 | 0 |
| Wash hands | 4 | 3 | 2 | 1 | 0 |
| Wring a towel ' | 4 | 3 | 2 | 1 | 0 |
| Zip pants | 4 | 3 | 2 | 1 | 0 |
| Zip a jacket | 4 | 3 | 2 | 1 | 0 |
| Button clothes | 4 | 3 | 2 | 1 | 0 |
| Fasten a clothes snap or hook | 4 | 3 | 2 | 1 | 0 |
| Cut nails with a nail clipper | 4 | 3 | 2 | 1 | 0 |
| Tie shoes with laces | 4 | 3 | 2 | 1 | 0 |

| Task | Easy | A little hard | Very hard | Cannot do | Never do |
|---|---|---|---|---|---|
| Use a remote control | 4 | 3 | 2 | 1 | 0 |
| Key in telephone numbers | 4 | 3 | 2 | 1 | 0 |
| Turn door knob to open a door | 4 | 3 | 2 | 1 | 0 |
| Turn key to open a lock | 4 | 3 | 2 | 1 | 0 |
| Carry a shopping bag with a hand loop | 4 | 3 | 2 | 1 | 0 |
| Open a previously-opened wide-<br>mouth jar (jam, pickle) | 4 | 3 | 2 | 1 | 0 |
| Open a previously-unopened carton<br>box (milk, cereal) | 4 | 3 | 2 | 1 | 0 |
| Pour liquid from a bottle into a glass | 4 | 3 | 2 | 1 | 0 |
| Open a medicine bottle with child-<br>proof top | 4 | 3 | 2 | 1 | 0 |
| Open an envelope without a letter<br>Opener | 4 | 3 | 2 | 1 | 0 |
| Peel vegetables or fruits | 4 | 3 | 2 | 1 | 0 |
| Count money (bills and coins) | 4 | 3 | 2 | 1 | 0 |
| Take things out of a wallet (bills, papers, credit cards) | 4 | 3 | 2 | 1 | 0 |
| Write 3 to 4 sentences legibly | 4 | 3 | 2 | 1 | 0 |
| Tum pages of a book | 4 | 3 | 2 | 1 | 0 |
| Use a hammer or screwdriver | 4 | 3 | 2 | 1 | 0 |
| Fold clothes after laundering | 4 | 3 | 2 | 1 | 0 |
| Take a CD/DVD out of its case and put it onto a player/drive | 4 | 3 | 2 | 1 | 0 |


#### 3. Human Activity Profile

## **Instructions**

• Please check each activity according to these directions:

- Check Column 1 ("Still Doing This Activity") if:
- You completed the activity unassisted the last time you had the need or opportunity to do so.
- Check Column 2 ("Have Stopped Doing This Activity") if:
- You have engaged in the activity in the past, but you probably would not perform the activity today even if the opportunity should arise.
- Check Column 3 ("Never Did This Activity") if:
- You have never engaged in the specific activity.

| Human Activity Profile Test | Still doing | Have stopped | Never did |
|---|---|---|---|
| | this activity | doing this activity | this activity |
| 1. Getting in and out of chairs | | | |
| or bed (without assistance) | | | |
| 2. Listening to the radio | | | |
| 3. Reading books, magazines or newspapers | | | |
| 4. Writing (letters, notes) | | | |
| 5. Working at a desk or table | | | |
| 6. Standing (for more than one minute) | | | |
| 7. Standing (for more than five minutes) | | | |
| 8. Dressing or undressing (without assistance) | | | |
| 9. Getting clothes from | | | |
| drawers or closets | | | |
| 10. Getting in or out of a car | | | |
| (without assistance) | | | |
| 11. Dining at a restaurant | | | |

| Human Activity Profile Test | Still doing | Have stopped | Never did |
|---|---|---|---|
| | this activity | doing this activity | this activity |
| 12. Playing cards/table games | | | |
| 13. Taking a bath (no assistance needed) | | | |
| 14. Putting on shoes, stockings or socks (no assistance needed) | | | |
| 15. Attending a movie, play, church event or sports activity | | | |
| 16. Walking 30 yards (27 meters) | | | |
| 17. Walking 30 yards (non-stop) | | | |
| 18. Dressing/undressing (no rest or break needed) | | | |
| 19.Using public transportation or | | | |
| driving a car (100 miles or less) | | | |
| 20. Using public transportation or | | | |
| driving a car (99 miles or more) | | | |
| 21. Cooking your own meals | | | |
| 22. Washing or drying dishes | | | |
| 23. Putting groceries on shelves | | | |
| 24. Ironing or folding clothes | | | |
| 25. Dusting/polishing furniture | | | |
| or polishing cars | | | |
| 26. Showering | | | |
| 27. Climbing six steps | | | |
| 28. Climbing six steps (non-stop) | | | |
| 29. Climbing nine steps | | | |
| 30. Climbing 12 steps | | | |

| Human Activity Profile Test | Still doing this activity | Have stopped doing this activity | Never did<br>this activity |
|---|---|---|---|
| 31. Walking ½ block on level ground | child deciving | doing this activity | this deal (10) |
| 32. Walking ½ block on | | | |
| level ground (non-stop) | | | |
| 33. Making a bed (not changing sheets) | | | |
| 34. Cleaning windows | | | |
| 35. Kneeling, squatting to do light work | | | |
| 36. Carrying a light load of groceries | | | |
| 37. Climbing nine steps (non-stop) | | | |
| 38. Climbing 12 steps (non-stop) | | | |
| 39. Walking ½ block uphill | | | |
| 40. Walking ½ block uphill (non-stop) | | | |
| 41. Shopping (by yourself) | | | |
| 42. Washing clothes (by yourself) | | | |
| 43. Walking one block on level | | | |
| ground | | | |
| 44. Walking two blocks on level ground | | | |
| 45. Walking one block on level | | | |
| ground (non-stop) | | | |
| 46. Walking two blocks on level | | | |
| ground (non-stop) | | | |
| 47. Scrubbing (floors, walls or cars) | | | |
| 48. Making beds (changing sheets) | | | |

| Human Activity Profile Test | Still doing this activity | Have stopped doing this activity | Never did this activity |
|---|---|---|---|
| 49. Sweeping | this activity | doing this activity | this activity |
| 50. Sweeping (five minutes non-stop) | | | |
| 51. Carrying a large suitcase or bowling (one line) | | | |
| 52. Vacuuming carpets | | | |
| 53. Vacuuming carpets (five minutes non-stop) | | | |
| 54. Painting (interior/exterior) | | | |
| 55. Walking six blocks on level ground | | | |
| 56. Walking six blocks on level ground (non-stop) | | | |
| 57. Carrying out the garbage | | | |
| 58. Carrying a heavy load of groceries | | | |
| 59. Climbing 24 steps | | | |
| 60. Climbing 36 steps | | | |
| 61. Climbing 24 steps (non-stop) | | | |
| 62. Climbing 36 steps (non-stop) | | | |
| 63. Walking one mile | | | |
| 64. Walking one mile (non-stop) | | | |
| 65. Running 110 yards (100 meters) or playing softball/baseball | | | |


| Human Activity Profile Test | Still doing | Have stopped | Never did |
|---|---|---|---|
| | this activity | doing this activity | this activity |
| 66. Dancing (social) | | | |
| 67. Doing calisthenics or aerobic | | | |
| dancing (5 minutes non-stop) | | | |
| 68. Mowing the lawn (power mower, | | | |
| but not a riding mower) | | | |
| 69. Walking two miles | | | |
| 70. Walking two miles (non-stop) | | | |
| 71. Climbing 50 steps | | | |
| 72. Shoveling, digging or spading | | | |
| 73. Shoveling, digging or spading | | | |
| (five minutes non-stop) | | | |
| 74. Climbing 50 steps (non-stop) | | | |
| 75. Walking three miles or golfing | | | |
| 18 holes without a riding cart | | | |
| 76. Walking three miles (non-stop) | | | |
| 77. Swimming 25 yards | | | |
| 78. Swimming 25 yards (non-stop) | | | |
| 79. Bicycling one mile | | | |
| 80. Bicycling two miles | | | |
| 81. Bicycling one mile (non-stop) | | | |
| 82. Bicycling two miles (non-stop) | | | |
| 83. Running or jogging ¼ mile | | | |
| 84. Running or jogging ½ mile | | | |

| Human Activity Profile Test | Still doing this activity | Have stopped doing this activity | Never did<br>this activity |
|---|---|---|---|
| 85. Playing tennis or racquetball | | | |
| 86. Playing basketball (game play) | | | |
| 87. Running or jogging ¼ mile (non-stop) | | | |
| 88. Running or jogging ½ mile (non-stop) | | | |
| 89. Running or jogging one mile | | | |
| 90. Running or jogging two miles | | | |
| 91. Running or jogging three miles | | | |
| 92. Running or jogging one mile in 12 minutes or less | | | |
| 93. Running or jogging two miles in 20 minutes or less | | | |
| 94. Running or jogging three miles in 30 minutes or less | | | |


| 16.17. | .5Com | ponent | 4: | Eves |
|--------|-------|--------|----|------|

| Patient Na | me: | | | Patient MR#: |
|------------|---------|-----|-----------------|--------------|
| Date of As | sessmer | nt: | | |
| Assessed: | Yes | No | Age Restriction | |

## 1. CAS - Initial assessment

Reason if "NO":

## PLEASE ASSESS if patient is 9 years old and older

Please Check off the boxes (grade the worst eye)

1+ = few separated spots

2+ = many separated spots

**3+ = confluent spots** 

| None = 0 | | Mild = 1 | Moderate = 2 | _ | Severe = 3 | |
|---|---|---|---|---|---|---|
| Schirmer's without<br>Anesthesia<br>> 10 mm | | Schirmer's without<br>Anesthesia<br>7 to 10 mm | Schirmer's without<br>Anesthesia<br>3 to 6 mm | | Schirmer's without<br>Anesthesia<br>< 3 mm | X |
| No<br>punctate<br>keratopath | | Mild<br>punctate<br>keratopathy | Moderate<br>punctate<br>keratopathy | | Severe<br>punctate<br>keratopathy | X |
| Grade 0 No conjunctival disease | X | Grade 1 conjunctival hyperemia occuring on the bulbar or palpebral conjuctiva. | Grade 2 palpebral conjunctival fibrovascular changes occuring along the superior border of the upper eyelid, or the lower border of the tarsal plate of the lower eyelid, with or without conjuctival epithelial sloughing, involving < 25 % of the total surface area OR Grade 3 palpebral conjunctival fibrovascular changes occuring along the superior border of the upper eyelid, or the lower border of the tarsal plate of the lower eyelid, involving 25 to 75 % of | | Grade 3 > 75 % of the total surface area with or without a cicatricial entropion. | |


Schirmer's without Anesthesia: Rt eye\_\_\_mm Lf eye\_\_mm Schirmer's with Anesthesia\*: Rt eye\_\_mm Lf eye\_\_mm

Overall Stage (max 3):-----

**Total Score (max 9): -----**

### 2. Not in CAS - Ocular Symptoms

| | Dryness | | | Redness | | | Irritation | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | None | Mild | Moderate | Severe | None | Mild | Moderate | Severe | None | Mild | Moderate | Severe |
| Right<br>Eye | | X | | | | X | | | | X | | |
| Left<br>Eye | | X | | | | X | | | | X | | |

#### 3. Not in CAS - Recommended therapy:

| | Recommended Therapy | | | |
|---|---|---|---|---|
| None | Ocular<br>lubrication | topical restasis<br>or<br>topical<br>corticosteroids | Punctual<br>occlusion | Other |
| | X | X | X | discussed ASED and scleral contact lenses |

## 4. Composite Assessment Scale:

| Test | Grade 0 (none) | Grade 1 (mild) | Grade 2 (moderate) | Grade 3 (severe) |
|---|---|---|---|---|
| Schirmer's Tear<br>Test (without<br>Anesthesia) | > 10 mm | 7-10 mm | 3-6 mm | < 3 mm |
| Punctate<br>Keratopathy | None | 1+ = few separated spots | 2+ = many separated spots | 3+ = confluent spots |


| | Conjunctival Inflammation and Scarring (see scheme below) | No conjunctival<br>disease | Grade 1 | Grade 2 or 3 | Grade 4 |
|---|---|---|---|---|---|
| I | Examined by: | | | <br>Date | |
| - | Signature | Printed | Name | <br>Date | |

## 16.18 APPENDIX R: CHRONIC GVHD COMPOSITE ASSESSMENT SCALE BARTHEL INDEX SCORE

| Patient Name: | MR #: |
|---------------|-------|
| Rater Name: | Date: |

| Activity | Score | Ratings |
|---|---|---|
| Feeding | | 0=unable 5=needs help cutting, spreading butter, etc., or requires modified diet 10= independent |
| Bathing | | 0=dependent<br>5=independent |
| Grooming | | 0=needs help with personal care 5=independent with face/hair/teeth/shaving (implements provided) |

| T | |
|---|---|
| Dressing | 0=dependent 5=needs help but can do about half unaided 10= independent (including buttons, zippers, laces, etc.) |
| Bowels | 0=incontinent (or needs to be given enemas) 5=occasional accidents 10= continent |
| Bladder | 0=incontinent, or catherized and unable to manage alone 5=occasional accidents 10= continent |
| Toilet Use | 0=dependent 5=needs some help, but can do something alone 10= independent (on and off, dressing and wiping) |
| Transfers (Bed to chair and Back) | 0=Unable, no sitting balance 5=major help (one or two people, physical), can sit 10=Minor help (verbal or physical) 15=independent |
| Mobility (on level surfaces) | 0=Immobile < 50 yards) 5=wheelchair independent, including corners>50 yards 10=walks with help of one person (verbal or physical)>50 yards 15=independent (may use any aid; for example cane or walker)>50 yards |
| Stairs | 0=unable 5=needs help (verbal, physical, carrying aid) 10= independent |

| Signature: | | <b>Printed Name:</b> | Date: |
|---|---|---|---|
| Total Score | e: (0-100) _ | | |
| | | 10= independent | |
| | | 5=needs help (verbal, physical, carrying ai | d) |
| Stairs | | 0=unable | |


## 16.19 APPENDIX S: CHRONIC GVHD COMPOSITE ASSESSMENT SCALE FRENCHAY ACTIVITIES INDEX

| Patient Name | <b>:</b> | MR #:_ | |
|---|---|---|---|
| Rater Name: | | _ Date: | |
| In the last 3 mon | ths, how often have you undertaken: | | |
| Task<br>Number | Task Description: Domestic Chores | Score | Ratings: 0=Never 1= Less than once a week 2=1-2 times per week 3=Most days |
| 1. | Preparing main meals | | |
| 2. | Washing up after meals | | |

In the last 3 months, how often have you undertaken:

**Subtotal Domestic Chores : (\_\_/6)** 

| Task Number | Task Description: Leisure/work | Score | Ratings: 0=Never 1= 1-2 times in 3 months 2= 3-12 times in 6 months 3=At least weekly |
|---|---|---|---|
| 3. | Washing clothes | | |
| 4. | Light Housework | | |
| 5. | Heavy Housework | | |
| 6. | Local Shopping | | |
| 7. | Social Occasions | | |
| 8. | Walking outside for >15 minutes | | |
| 9. | Actively pursuing a hobby | | |
| 10. | Driving a car/going on bus | | |

| Subtotal Leisure/Work: (/24) |
|------------------------------|
|------------------------------|

In the last 6 months how often have you undertaken:

| Task<br>Number | Task Description: Outdoor | Score | Ratings: |
|---|---|---|---|
| 11. | Travel outing/car ride | | 0=Never $1=1-2$ times in 6 months $2=3-12$ times in 6 months $3=$ at last weekly |
| 12. | Gardening | | 0=Never<br>1=Light<br>2=Moderate<br>3=Heavy/All necessary |
| 13. | Household Maintenance | | 0=Never<br>1=Light<br>2=Moderate<br>3=Heavy/All necessary |
| 14. | Reading Books | | 0=None<br>1=1 in 6 months<br>2=Less than 1 in 2 weeks<br>3= More than 1 every 2 weeks |
| 15. | Gainful Work | | 0=None<br>1=Up to 10 hours/week<br>2=10-30 hours/week<br>3=Over 30 hours/week |
| | Subtotal Outdoor: (/15) | | |

| Total Score:/45 | | |
|-----------------|---------------|-------|
| | Printed Name: | Date: |


#### Revised guidelines for using the Frenchay Activities Index

The aim is to record activities which require some initiative from the patient. It is important to concentrate upon the patient's actual frequency of activity over the recent past, not distant past performance nor potential performance. One activity can only score on one item.

#### **Specific item information:**

- 1. Needs to play a substantial part in the organization, preparation and cooking of main meal. Not just making snacks or reheating prepared food.
- 2. Must do all or share equally, e.g. washing or wiping and putting away. Not just rinsing an occasional item.
- 3. Organization of washing and drying clothes, whether in washing machine, or by hand or at laundromat. Sharing task equally, e.g. loading, unloading, hanging, folding.
- 4. Dusting, polishing, ironing, tidying small objects or bedclothes. Anything heavier is included in item 5.
- 5. All heavier housework including changing beds, cleaning floors, fires and windows, vacuuming, moving chairs, etc.
- 6. Playing a substantial role in organizing and buying groceries, whether small or large amounts. Must go to the shop and not just push a cart. Can include collection of pension or going to the Post Office.
- 7. Going out to clubs, church activities, cinema, theatre, drinking, to dinner with friends, etc. May be transported there, provided patient takes an active part once arrived. Includes social activities at home, initiated by the patient, e.g. visits from family or friends not where main purpose is to provide care.
- 8. Sustained walking for at least 15 minutes (allowed short stops for breath). About one mile. Can include walking to do shopping, provided walks far enough.
- 9. Must require some 'active' participation and thought, e.g. propagating or caring for houseplants, knitting, painting, games, sports (not just watching sport on television). Can be mental activities, e.g. reading specialist magazines, doing the stocks and shares or window shopping for pleasure.
- 10. Must drive a car (not just be a passenger), or get to a bus/coach and travel on it independently.
- 11. Coach or rail trips or car rides to some place for pleasure. Not for a routine 'social outing' (i.e. shopping, going to local friends). Must involve some organization and decision-making by the patient. Excludes trips organized passively by institutions unless patient exercises choice on whether to go. The common factor is travel for pleasure. Holidays within the six months are divided into days per month e.g. a 7-day holiday equals 1 or 2 days per month.
- 12. Gardening outside:
  - a. Light = occasional weeding or sweeping paths
  - b. Moderate = regular weeding, raking, pruning, etc.
  - c. Heavy = all necessary work including heavy digging.
- 13. Household maintenance:
  - a. Light = repairing small items, replacing lamp lightbulb or plug
  - b. Moderate = spring cleaning, hanging a picture, routine car maintenance
  - c. Heavy = painting/decorating, most necessary household/car maintenance.


14. Must be full-length books, not periodicals, magazines or newspapers. Can be talking books.

15. Work for which the patient is paid, not voluntary work. The time worked should be averaged out over six months. For example, one month working for 18 hours/week over the six-month period would be scored as 'up to 10 hours/week'.

# 16.20 APPENDIX T: QUALITY OF LIFE ASSESSMENTS (OBTAINED AT BASELINE THEN YEARLY)

#### FACT-BMT (Version 4)

By circling one (1) number per line, please indicate how true each statement has been for you during the past 7 days.

| <u>-</u> | ADDITIONAL CONCERNS | Not<br>at all | A little<br>bit | Some-<br>what | Quite<br>a bit | Very<br>much |
|---|---|---|---|---|---|---|
| BMT1 | I am concerned about keeping my job (include work at home) | 0 | 1 | 2 | 3 | 4 |
| BMT2 | I feel distant from other people | | 1 | 2 | 3 | 4 |
| BMT3 | I worry that the transplant will not work | 0 | 1 | 2 | 3 | 4 |
| BMT4 | The effects of treatment are worse than I had imagined | 0 | 1 | 2 | 3 | 4 |
| C6 | I have a good appetite | 0 | 1 | 2 | 3 | 4 |
| C7 | I like the appearance of my body | 0 | 1 | 2 | 3 | 4 |
| BMT5 | I am able to get around by myself | 0 | 1 | 2 | 3 | 4 |
| BMT6 | I get tired easily | 0 | 1 | 2 | 3 | 4 |
| BL4 | I am interested in sex | 0 | 1 | 2 | 3 | 4 |
| BMT7 | I have concerns about my ability to have children | 0 | 1 | 2 | 3 | 4 |
| BMT8 | I have confidence in my nurse(s) | 0 | 1 | 2 | 3 | 4 |
| BMT9 | I regret having the bone marrow transplant | 0 | 1 | 2 | 3 | 4 |
| BMT | I can remember things | 0 | 1 | 2 | 3 | 4 |
| 10<br>Br1 | I am able to concentrate (e.g., reading) | 0 | 1 | 2 | 3 | 4 |
| BMT | I have frequent colds/infections | 0 | 1 | 2 | 3 | 4 |
| 11<br>BMT<br>12 | My eyesight is blurry | 0 | 1 | 2 | 3 | 4 |
| BMT<br>13 | I am bothered by a change in the way food tastes | 0 | 1 | 2 | 3 | 4 |
| BMT<br>14 | I have tremors | 0 | 1 | 2 | 3 | 4 |
| B1 | I have been short of breath | 0 | 1 | 2 | 3 | 4 |
| BMT<br>15 | I am bothered by skin problems (e.g., rash, itching) | 0 | 1 | 2 | 3 | 4 |
| BMT<br>16 | I have trouble with my bowels | 0 | 1 | 2 | 3 | 4 |
| BMT | My illness is a personal hardship for my close family | | | | | |
| 17 | members | | 1 | 2 | 3 | 4 |
| BMT<br>18 | The cost of my treatment is a burden on me or my family | 0 | 1 | 2 | 3 | 4 |

US English
Copyright 1987, 1997
Page 3 of

## FACT-BMT (Version 4)

By circling one (1) number per line, please indicate how true each statement has been for you during the past 7 days.

| | EMOTIONAL WELL-BEING | Not<br>at all | A little<br>bit | Some-<br>what | Quite<br>a bit | Very<br>much |
|---|---|---|---|---|---|---|
| GE1 | I feel sad | 0 | 1 | 2 | 3 | 4 |
| GE2 | I am satisfied with how I am coping with my illness | 0 | 1 | 2 | 3 | 4 |
| GE3 | I am losing hope in the fight against my illness | 0 | 1 | 2 | 3 | 4 |
| GE4 | I feel nervous | 0 | 1 | 2 | 3 | 4 |
| GE5 | I worry about dying | 0 | 1 | 2 | 3 | 4 |
| GE6 | I worry that my condition will get worse | 0 | 1 | 2 | 3 | 4 |

| | × | FUNCTIONAL WELL-BEING | Not<br>at all | A little<br>bit | Some-<br>what | Quite<br>a bit | Very<br>much |
|---|---|---|---|---|---|---|---|
| | GF1 | I am able to work (include work at home) | 0 | 1 | 2 | 3 | 4 |
| | GF2 | My work (include work at home) is fulfilling | 0 | 1 | 2 | 3 | 4 |
| | GF3 | I am able to enjoy life | 0 | 1 | 2 | 3 | 4 |
| | GF4 | I have accepted my illness | 0 | 1 | 2 | 3 | 4 |
| | GF5 | I am sleeping well | 0 | 1 | 2 | 3 | 4 |
| | GF6 | I am enjoying the things I usually do for fun | 0 | 1 | 2 | 3 | 4 |
| | GF7 | I am content with the quality of my life right now | 0 | 1 | 2 | 3 | 4 |
| 1 | | | | | | | |

US English Copyright 1987, 1997

FACT-BMT (Version 4)

By circling one (1) number per line, please indicate how true each statement has been for you during the past 7 days.

| | ADDITIONAL CONCERNS | Not<br>at all | A little<br>bit | Some-<br>what | Quite<br>a bit | Very<br>much |
|---|---|---|---|---|---|---|
| BMT1 | I am concerned about keeping my job (include work at home) | 0 | 1 | 2 | 3 | 4 |
| BMT2 | I feel distant from other people | 0 | 1 | 2 | 3 | 4 |
| BMT3 | I worry that the transplant will not work | 0 | 1 | 2 | 3 | 4 |
| BMT4 | The effects of treatment are worse than I had imagined | 0 | 1 | 2 | 3 | 4 |
| C6 | I have a good appetite | 0 | 1 | 2 | 3 | 4 |
| C7 | I like the appearance of my body | 0 | 1 | 2 | 3 | 4 |
| BMT5 | I am able to get around by myself | 0 | 1 | 2 | 3 | 4 |
| BMT6 | I get tired easily | 0 | 1 | 2 | 3 | 4 |
| BL4 | I am interested in sex | 0 | 1 | 2 | 3 | 4 |
| BMT7 | I have concerns about my ability to have children | 0 | 1 | 2 | 3 | 4 |
| BMT8 | I have confidence in my nurse(s) | 0 | 1 | 2 | 3 | 4 |
| вмт9 | I regret having the bone marrow transplant | 0 | 1 | 2 | 3 | 4 |
| BMT<br>10 | I can remember things | 0 | 1 | 2 | 3 | 4 |
| Br1 | I am able to concentrate (e.g., reading) | 0 | 1 | 2 | 3 | 4 |
| BMT<br>11 | I have frequent colds/infections | 0 | 1 | 2 | 3 | 4 |
| BMT<br>12 | My eyesight is blurry | 0 | 1 | 2 | 3 | 4 |
| BMT<br>13 | I am bothered by a change in the way food tastes | 0 | 1 | 2 | 3 | 4 |
| BMT<br>14 | I have tremors | 0 | 1 | 2 | 3 | 4 |
| B1 | I have been short of breath | 0 | 1 | 2 | 3 | 4 |
| BMT<br>15 | I am bothered by skin problems (e.g., rash, itching) | 0 | 1 | 2 | 3 | 4 |
| BMT<br>16 | I have trouble with my bowels | 0 | 1 | 2 | 3 | 4 |
| BMT<br>17 | My illness is a personal hardship for my close family | | | | | |
| -17 | members | | 1 | 2 | 3 | 4 |
| BMT<br>18 | The cost of my treatment is a burden on me or my family | 0 | 1 | 2 | 3 | 4 |

US English Copyright 1987, 1997

3/10/03 Page 3 of 3


## Your Health and Well-Being

This survey asks for your views about your health. This information will help keep track of how you feel and how well you are able to do your usual activities. *Thank you for completing this survey!* 

For each of the following questions, please mark an  $\boxtimes$  in the one box that best describes your answer.

1. In general, would you say your health is:



2. <u>Compared to one year ago</u>, how would you rate your health in general <u>now</u>?



SF-36v2 TM Health Survey © 1996, 2000 by QualityMetric Incorporated and Medical Outcomes Trust. All Rights Reserved. SF-36® is a registered trademark of Medical Outcomes Trust. (SF-36v2 Standard, US Version 2.0)


3. The following questions are about activities you might do during a typical day. Does your health now limit you in these activities? If so, how much?

| | Yes,<br>limited<br>a lot | Yes,<br>limited<br>a little | No, not limited at all |
|---|---|---|---|
| Nigorous activities, such as running, lifting heavy objects, participating in strenuous sports | | 2 | 3 |
| Moderate activities, such as moving a table pushing a vacuum cleaner, bowling, or playing golf | | 2 | 3 |
| · Lifting or carrying groceries | 1 | 2 | 3 |
| d Climbing several flights of stairs | 1 | 2 | 3 |
| e Climbing one flight of stairs | 1 | | 3 |
| f Bending, kneeling, or stooping | 1 | 2 | 3 |
| <sub>ε</sub> Walking more than a mile | 1 | 2 | 3 |
| h Walking several hundred yards | 1 | 2 | 3 |
| Walking one hundred yards | 1 | 2 | 3 |
| Bathing or dressing yourself | | | |


4. During the <u>past 4 weeks</u>, how much of the time have you had any of the following problems with your work or other regular daily activities <u>as a result of your physical health?</u>

| | | All of the time | | Some of the time | | None of the time |
|---|---|---|---|---|---|---|
| | <sup>a</sup> Cut down on the <u>amount of time</u> you spent on work or other activities | 🔲 1 | 2 | 3 | 🔲 4 | 5 |
| | ь Accomplished less than you would like | 1 | 2 | 3 | | 5 |
| | Were limited in the <u>kind</u> of work or other activities | 🔲 1 | 2 | 3 | 🔲 4 | 5 |
| | Had <u>difficulty</u> performing the work or other activities (for example, it took extra effort) | <u> </u> | 2 | 3 | | 5 |
| 5. | During the <u>past 4 weeks</u> , how much of the following problems with your work or o result of any emotional problems (such | ther reg | gular dai | ily activi | ties <u>as</u> | <u>a</u> |
| | | All of the time | | Some of the time | A little of the time | None of the time |
| | a Cut down on the <u>amount of time</u> you spent<br>on work or other activities | 1 | 🔲 2 | 3 | 4 | 5 |
| | ь Accomplished less than you would like | 🔲 1 | 2 | 3 | []4 | 5 |
| | D'1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | | | | | |
| | Did work or other activities less carefully than usual | 1 | 2 | 3 | 4 | 5 |

 $SF-36v2 \stackrel{TM}{=} Health \ Survey © \ 1996, 2000 \ by \ Quality Metric \ Incorporated \ and \ Medical \ Outcomes \ Trust.$  All Rights Reserved.  $SF-36 @ \ is \ a \ registered \ trademark \ of \ Medical \ Outcomes \ Trust.$   $(SF-36v2 \ Standard, US \ Version \ 2.0)$ 


| 6. | During the past 4 weeks, to what extent has your physical health or |
|----|-----------------------------------------------------------------------|
| | emotional problems interfered with your normal social activities with |
| | family, friends, neighbors, or groups? |

| Not at all | Slightly | Moderately | Quite a bit | Extremely |
|------------|----------|--------------|--------------|-----------|
| | | lacktriangle | lacktriangle | • |
| 1 | 2 | 3 | 4 | 5 |

7. How much bodily pain have you had during the past 4 weeks?

| None | Very mild | Mild | Moderate | Severe | Very Severe |
|------|------------|------|------------|--------|-------------|
| • | lacksquare | | lacksquare | | lacksquare |
| 1 | 2 | 3 | 4 | 5 | 6 |

8. During the <u>past 4 weeks</u>, how much did <u>pain</u> interfere with your normal work (including both work outside the home and housework)?

| Not at all | A little bit | Moderately | Quite a bit | Extremely |
|--------------|--------------|--------------|--------------|--------------|
| lacktriangle | lacktriangle | lacktriangle | lacktriangle | lacktriangle |
| i | 2 | 3 | 4 | 5 |

 $SF-36v2 \stackrel{\mathrm{TM}}{=} Health \ Survey © \ 1996, \ 2000 \ by \ QualityMetric \ Incorporated \ and \ Medical \ Outcomes \ Trust.$  All Rights Reserved.  $SF-36@ \ is \ a \ registered \ trademark \ of \ Medical \ Outcomes \ Trust.$   $(SF-36v2 \ Standard, \ US \ Version \ 2.0)$

9. These questions are about how you feel and how things have been with you during the past 4 weeks. For each question, please give the one answer that comes closest to the way you have been feeling. How much of the time during the past 4 weeks...

| | All of<br>the time | Most of the time | Some of the time | A little of the time | None of<br>the time |
|---|---|---|---|---|---|
| a Did you feel full of life? | ı | 2 | 3 | 4 | 5 |
| ь Have you been very nervous? | ī | 2 | 3 | 4 | 5 |
| Have you felt so down in the dumps that nothing could cheer you up? | 1 | 2 | 3 | 🗖 4 | 5 |
| d Have you felt calm and peaceful? | 1 | 2 | 3 | 🗀 4 | 5 |
| e Did you have a lot of energy? | 1 | 2 | 3 | 🔲 4 | 5 |
| Have you felt downhearted and depressed? | 1 | 2 | 3 | 4 | 5 |
| ε Did you feel worn out? | <u>l</u> 1 | 2 | 3 | 🗀 4 | 5 |
| h Have you been happy? | □1 | 2 | 3 | 🔲 4 | 5 |
| Did you feel tired? | 1 | 2 | 3 | 🔲 4 | 5 |

10. During the <u>past 4 weeks</u>, how much of the time has your <u>physical health</u> <u>or emotional problems</u> interfered with your social activities (like visiting friends, relatives, etc.)?

| All of the time | Most of the time | Some of the time | A little of the time | None of the time |
|---|---|---|---|---|
| _ | lacktriangle | $\blacksquare$ | lacktriangle | • |
| 1 | 2 | 3 | 4 | 5 |

SF-36v2 TM Health Survey © 1996, 2000 by QualityMetric Incorporated and Medical Outcomes Trust. All Rights Reserved. SF-36® is a registered trademark of Medical Outcomes Trust. (SF-36v2 Standard, US Version 2.0)

| | I seem to get sick a little easier than other people |
|---|---|
| | ь I am as healthy as anybody I know |
| | $_{\circ}$ I expect my health to get worse |
| | d My health is excellent |
| | THANK YOU FOR COMPLETING THESE QUESTIONS! |
| | SF-36v2™ Health Survey © 1996, 2000 by QualityMetric Incorporated and Medical Outcomes Trust. All Rights Reserved. SF-36® is a registered trademark of Medical Outcomes Trust. (SF-36v2 Standard, US Version 2.0) |
| Today's Date: | MR#/Name: |

11. How TRUE or FALSE is each of the following statements for you?

Definitely Mostly

true

true

Don't

know

Mostly Definitely

false

false

Abbreviated Title: Pomalidomide for cGvHD


### B. CHRONIC GVHD ACTIVITY ASSESSMENT-PATIENT SELF REPORT

| Symptoms | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Please rate how severe th<br>symptoms have been in th<br>days. Please fill in the cir<br>(symptom has not been p | ne <u>last seven</u><br>cle below from 0 | Not<br>Present | : | | | | | | | | | d As You<br>Imagine |
| (the symptom was as bad imagine it could be) for ea | as you can | 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| Your <b>skin itching</b> at its \ | | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Your mouth dryness at | its WORST? | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Your <b>mouth pain</b> at its V | VORST? | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Your mouth sensitivity | at its WORST? | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
| Eyes | Please rate (not at all s | how sev | vere is thi | s eye syn | nptom, be | · | 0 1 | 2 3 | 4 5 | 6 7 | 8 9 | 10 |
| Vulvovaginal Symptom<br>(females only) | Do you hav<br>of your vag<br>OR<br>Do you hav<br>intercourse | ina, vulva<br>ve any dis | a or labia | ? | | | ( | Yes No | ıpplicable | | _ 0 | 10 |
| 1. Overall, do you think 1= mild 2=moderate 3=severe 2. Please circle the num symptoms that are not | that your chron | how sev | ere your | chronic | graft ver | sus host | disease | sympto | ms are, \ | where 0 i | s cGvHI | ) |
| 0 1 2 | 3 4 | 5 | 6 | 7 | 8 | 9 | 10 | | | | | |
| cGvHD symptoms<br>not at all severe | | | | | | sy | vere cGvHI<br>mptoms<br>oossible | ) | | | | |
| 3. Compared to a mont | <u>h ago,</u> overall w | ould you | ı say tha | t your co | SvHD sy | mptoms | are: | | | | | |
| +3= Very much better<br>+2= Moderately better<br>+1=A little better<br>0= About the same<br>-1=A little worse<br>-2=Moderately worse<br>-3=Very much worse | | | | | | | | | | | | |


# Attach copies of: Adults (persons 18 years or older): -Lee cGvHD Symptom Scale -Human Activity Profile

- -SF036
- -FACT-BMT

| Children/Adolescents | persons 17 | vears or | vounger) |
|----------------------|------------|----------|----------|

- Children/Adolescents (persons 17 years or younger):
   -Lee cGvHD Symptom Scale (persons 8-12 years old may complete with help of the health care professional)
   -ASK-p38 Activities Scale for Kids
   -VARNI-Generic and Disease Specific Inventory

| Гoday's Date: | MR#/Name: |
|---------------|-----------|
| • | |


#### C. Human Activity Profile

### **Instructions**

• Please check each activity according to these directions:

- Check Column 1 ("Still Doing This Activity") if:
- You completed the activity unassisted the last time you had the need or opportunity to do so.
- Check Column 2 ("Have Stopped Doing This Activity") if:
- You have engaged in the activity in the past, but you probably would not perform the activity today even if the opportunity should arise.
- Check Column 3 ("Never Did This Activity") if:
- You have never engaged in the specific activity.

| Human Activity Profile Test | Still doing this activity | Have stopped doing this activity | Never did<br>this activity |
|---|---|---|---|
| 1. Getting in and out of chairs | | | |
| or bed (without assistance) | | | |
| 2. Listening to the radio | | | |
| 3. Reading books, magazines or newspapers | | | |
| 4. Writing (letters, notes) | | | |
| 5. Working at a desk or table | | | |
| 6. Standing (for more than one minute) | | | |
| 7. Standing (for more than five minutes) | | | |
| 8. Dressing or undressing (without assistance) | | | |
| 9. Getting clothes from | | | |
| drawers or closets | | | |
| 10. Getting in or out of a car | | | |
| (without assistance) | | | |

| Human Activity Profile Test | Still doing this activity | Have stopped doing this activity | Never did this activity |
|---|---|---|---|
| | this activity | doing this activity | this activity |
| 11. Dining at a restaurant | | | |
| 12. Playing cards/table games | | | |
| 13. Taking a bath (no assistance needed) 14. Putting on shoes, stockings or socks (no assistance needed) 15. Attending a movie, play, church event or sports activity | | | |
| 16. Walking 30 yards (27 meters) | | | |
| 17. Walking 30 yards (non-stop) | | | |
| 18. Dressing/undressing (no rest or break needed) | | | |
| 19.Using public transportation or driving a car (100 miles or less) | | | |
| 20. Using public transportation or driving a car (99 miles or more) | | | |
| 21. Cooking your own meals | | | |
| 22. Washing or drying dishes | | | |
| 23. Putting groceries on shelves | | | |
| 24. Ironing or folding clothes | | | |
| 25. Dusting/polishing furniture or polishing cars | | | |
| 26. Showering | | | |
| 27. Climbing six steps | | | |
| 28. Climbing six steps (non-stop) | | | |
| 29. Climbing nine steps | | | |

| Human Activity Profile Test | Still doing | Have stopped | Never did |
|---|---|---|---|
| 20. Climbing 12 stone | this activity | doing this activity | this activity |
| 30. Climbing 12 steps | | | |
| 31. Walking ½ block on level ground | | | |
| 32. Walking ½ block on | | | |
| level ground (non-stop) | | | |
| 33. Making a bed (not changing sheets) | | | |
| 34. Cleaning windows | | | |
| 35. Kneeling, squatting to do light work | | | |
| 36. Carrying a light load of groceries | | | |
| 37. Climbing nine steps (non-stop) | | | |
| 38. Climbing 12 steps (non-stop) | | | |
| 39. Walking ½ block uphill | | | |
| 40. Walking ½ block uphill (non-stop) | | | |
| 41. Shopping (by yourself) | | | |
| 42. Washing clothes (by yourself) | | | |
| 43. Walking one block on level | | | |
| ground | | | |
| 44. Walking two blocks on level | | | |
| ground | | | |
| 45. Walking one block on level | | | |
| ground (non-stop) | | | |
| 46. Walking two blocks on level | | | |
| ground (non-stop) | | | |
| 47. Scrubbing (floors, walls or cars) | | | |

| Human Activity Profile Test | Still doing this activity | Have stopped doing this activity | Never did<br>this activity |
|---|---|---|---|
| 48. Making beds (changing sheets) | | | , |
| 49. Sweeping | | | |
| 50. Sweeping (five minutes non-stop) | | | |
| 51. Carrying a large suitcase or bowling (one line) | | | |
| 52. Vacuuming carpets | | | |
| 53. Vacuuming carpets (five minutes non-stop) | | | |
| 54. Painting (interior/exterior) | | | |
| 55. Walking six blocks on level ground | | | |
| 56. Walking six blocks on level ground (non-stop) | | | |
| 57. Carrying out the garbage | | | |
| 58. Carrying a heavy load of groceries | | | |
| 59. Climbing 24 steps | | | |
| 60. Climbing 36 steps | | | |
| 61. Climbing 24 steps (non-stop) | | | |
| 62. Climbing 36 steps (non-stop) | | | |
| 63. Walking one mile | | | |
| 64. Walking one mile (non-stop) | | | |

| Human Activity Profile Test | Still doing | Have stopped | Never did |
|---|---|---|---|
| | this activity | doing this activity | this activity |
| 65. Running 110 yards (100 meters) | | | |
| or playing softball/baseball | | | |
| 66. Dancing (social) | | | |
| 67. Doing calisthenics or aerobic | | | |
| dancing (5 minutes non-stop) | | | |
| 68. Mowing the lawn (power mower, | | | |
| but not a riding mower) | | | |
| 69. Walking two miles | | | |
| 70. Walking two miles (non-stop) | | | |
| 71. Climbing 50 steps | | | |
| 72. Shoveling, digging or spading | | | |
| 73. Shoveling, digging or spading | | | |
| (five minutes non-stop) | | | |
| 74. Climbing 50 steps (non-stop) | | | |
| 75. Walking three miles or golfing | | | |
| 18 holes without a riding cart | | | |
| 76. Walking three miles (non-stop) | | | |
| 77. Swimming 25 yards | | | |
| 78. Swimming 25 yards (non-stop) | | | |
| 79. Bicycling one mile | | | |
| 80. Bicycling two miles | | | |
| 81. Bicycling one mile (non-stop) | | | |
| 82. Bicycling two miles (non-stop) | | | |

| Human Activity Profile Test | Still doing this activity | Have stopped doing this activity | Never did<br>this activity |
|---|---|---|---|
| 83. Running or jogging 1/4 mile | | | |
| 84. Running or jogging ½ mile | | | |
| 85. Playing tennis or racquetball | | | |
| 86. Playing basketball (game play) | | | |
| 87. Running or jogging 1/4 mile (non-stop) | | | |
| 88. Running or jogging ½ mile (non-stop) | | | |
| 89. Running or jogging one mile | | | |
| 90. Running or jogging two miles | | | |
| 91. Running or jogging three miles | | | |
| 92. Running or jogging one mile in 12 minutes or less | | | |
| 93. Running or jogging two miles in 20 minutes or less | | | |
| 94. Running or jogging three miles in 30 minutes or less | | | |

| Todav's Date: | MR#/Name: |
|---------------|-----------|
| loday & Dale. | MR#/Name |


#### D. Disabilities of the Arm, Shoulder and Hand.




## DISABILITIES OF THE ARM, SHOULDER AND HAND

Please rate your ability to do the following activities in the last week by circling the number below the appropriate response.

| | | NO<br>DIFFICULTY | MILD<br>DIFFICULTY | MODERATE<br>DIFFICULTY | SEVERE<br>DIFFICULTY | UNABLE |
|---|---|---|---|---|---|---|
| 1. | Open a tight or new jar. | 1 | 2 | 3 | 4 | 5 |
| 2. | Write: | 1 | 2 | 3 | 4 | 5 |
| 3. | Turn a key. | 1 | 2 | 3 | 4 | 5 |
| 4. | Prepare a meal. | 1 | 2 | 3 | 4 | 5 |
| 5. | Push open a heavy door. | 1 | 2 | 3 | 4 | 5 |
| 6. | Place an object on a shelf above your head. | 1 | 2 | 3 | 4 | 5 |
| 7. | Do heavy household chores (e.g., wash walls, wash floors). | 1 | 2 | 3 | 4 | 5 |
| 8. | Garden or do yard work. | 1 | 2 | 3 | 4 | 5 |
| 9. | Make a bed. | 1 | 2 | 3 | 4 | 5 |
| 10. | Carry a shopping bag or briefcase. | 1 | 2 | 3 | 4 | 5 |
| 11. | Carry a heavy object (over 10 lbs). | 1 | 2 | 3 | 4 | 5 |
| 12. | Change a lightbulb overhead. | 1 | 2 | 3 | 4 | 5 |
| 13. | Wash or blow dry your hair. | 1 | 2 | 3 | 4 | 5 |
| 14. | Wash your back. | 1 | 2 | 3 | 4 | 5 |
| 15. | Put on a pullover sweater. | 1 | 2 | 3 | 4 | 5 |
| 16. | Use a knife to cut food. | 1 | 2 | 3 | 4 | 5 |
| 17. | Recreational activities which require little effort (e.g., cardplaying, knitting, etc.). | 1 | 2 | 3 | 4 | 5 |
| 18. | Recreational activities in which you take some force or impact through your arm, shoulder or hand (e.g., golf, hammering, tennis, etc.). | 1 | 2 | 3 | 4 | 5 |
| 19. | Recreational activities in which you move your arm freely (e.g., playing frisbee, badminton, etc.). | 1 | 2 | 3 | 4 | 5 |
| 20. | Manage transportation needs (getting from one place to another). | 1 | 2 | 3 | 4 | 5 |
| 21. | Sexual activities. | 1 | 2 | 3 | 4 | 5 |


# DISABILITIES OF THE ARM, SHOULDER AND HAND

| | | NOT AT ALL | SLIGHTLY | MODERATELY | QUITE<br>A BIT | EXTREMELY |
|---|---|---|---|---|---|---|
| 22. | During the past week, to what extent has your arm, shoulder or hand problem interfered with your normal social activities with family, friends, neighbours or groups? (circle number) | 1 | 2 | 3 | 4 | 5 |
| | • | NOT LIMITED<br>AT ALL | SLIGHTLY<br>LIMITED | MODERATELY<br>LIMITED | VERY<br>LIMITED | UNABLE |
| 23. | During the past week, were you limited in your work or other regular daily activities as a result of your arm, shoulder or hand problem? (circle number) | 1 | 2 | 3 | 4 | 5 |
| Plea | se rate the severity of the following symptoms in the last we | ek. <i>(circle num</i> | ber) | | | |
| | | NONE | MILD | MODERATE | SEVERE | EXTREME |
| 24. | Arm, shoulder or hand pain. | 1 | 2 | 3 | 4 | 5 |
| 25. | Arm, shoulder or hand pain when you performed any specific activity. | 1 | 2 | 3 | 4 | 5 |
| 26. | Tingling (pins and needles) in your arm, shoulder or hand. | 1 | 2 | 3 | 4 | 5 |
| 27. | Weakness in your arm, shoulder or hand. | 1 | 2 | 3 | 4 | 5 |
| 28. | Stiffness in your arm, shoulder or hand. | 1 | 2 | 3 | 4 | 5 |
| | | NO<br>DIFFICULTY | MILD<br>DIFFICULTY | MODERATE<br>DIFFICULTY | SEVERE<br>DIFFICULTY | SO MUCH<br>DIFFICULTY<br>THAT I<br>CAN'T SLEEP |
| 29. | During the past week, how much difficulty have you had sleeping because of the pain in your arm, shoulder or hand (circle number) | ?<br>1 | 2 | 3 | 4 | 5 |
| | | STRONGLY<br>DISAGREE | DISAGREE | NEITHER AGREE<br>NOR DISAGREE | AGREE | STRONGLY<br>AGREE |
| 30. | I feel less capable, less confident or less useful<br>because of my arm, shoulder or hand problem.<br>(circle number) | 1 | 2 | 3 | 4 | 5 |

**DASH DISABILITY/SYMPTOM SCORE** =  $[(\underbrace{\text{sum of n responses}}_{n}) - 1] \times 25$ , where n is equal to the number of completed responses.

A DASH score may not be calculated if there are greater than 3 missing items.

| <b>Abbreviated Title:</b> Pomalidomide for cGvHD <b>Version Date:</b> 4/29/2025 | |
|---|---|
| Today's Date: | MR#/Name: |


#### E. PRO-CTCAE for Pomalidomide

As individuals go through treatment for their cancer they sometimes experience different symptoms and side effects.

For each question, please check or mark an X in the one box that best describes your experiences over the past 7 days...

| FATIGUE, TIREDNESS OR LACK OF ENERGY | | | | |
|---|---|---|---|---|
| What was the SEVERITY of your FATIGUE, TIREDNESS, OR LACK OF ENERGY at its WORST? | | | | |
| O None | O None O Mild O Moderate O Severe O Very severe | | | |
| How much did FATIGUE, TIREDNESS, OR LACK OF ENERGY at its WORST INTERFERE with your usual or daily activities? | | | | |
| O Not at all | O A little bit | O Somewhat | O Quite a bit | O Very much |

| NUMBNES | NUMBNESS OR TINGLING IN YOUR HANDS OR FEET | | | |
|---|---|---|---|---|
| What was the SEVERITY of your NUMBNESS OR TINGLING IN YOUR HANDS OR FEET at its WORST? | | | | |
| O None | O None O Mild O Moderate O Severe O Very severe | | | |
| How much did NUMBNESS OR TINGLING IN YOUR HANDS OR FEET INTERFERE with your usual or daily activities? | | | | |
| O Not at all | O A little bit | O Somewhat | O Quite a bit | O Very much |

| PAIN | | | | |
|---|---|---|---|---|
| How OFTEN | N did you have | PAIN? | | |
| O Never | O Rarely | O Occasionally | O Frequently | O Almost constantly |
| What was th | e SEVERITY | of your PAIN at its V | WORST? | |
| O None | O Mild | O Moderate | O Severe | O Very severe |
| How much did PAIN INTEREFERE with your usual or daily activities? | | | | |
| O Not at | O A little | O Somewhat | O Quite a bit | O Very much |
| all | bit | | | j |

| CONSTIPATION | | | | |
|---|---|---|---|---|
| What was the SEVERITY of your CONSTIPATION at its WORST? | | | | |
| O None | O Mild | O Moderate | O Severe | O Very severe |

| PROBLEMS W | ITH CONCENT | RATION | | |
|---|---|---|---|---|
| What was the SE | VERITY of your | PROBLEMS WITH | CONCENTRATO | ON at their WORST? |
| O None | O Mild | O Moderate | O Severe | O Very severe |
| How much did PROBLEMS WITH CONCENTRATION INTERFERE with your usual or daily activities? | | | | |
| O Not at all O A little bit O Somewhat O Quite a bit O Very much | | | | O Very much |
| TREMORS | | | | |
| How OFTEN di | d you have TRE | MORS? | | |
| O Never | O Rarely | O Occasionally | O Frequently | O Almost constantly |
| What was the SEVERITY of your TREMORS at their WORST? | | | | |
| O None | O Mild | O Moderate | O Severe | O Very severe |

| OTHER SYMPTOMS | | |
|---|---|---|
| Do you have any other symptoms that | you wish | to report? |
| O Yes | | O No |
| Please list any other symptoms: | | |
| 1. | What was the severity of this symptom at its WORST? | |
| | O None O Mild O Moderate O Severe O Very Severe | |
| 2. | What was the severity of this symptom at its WORST? | |
| | O None O Mild O Moderate O Severe O Very Severe | |
| 3. | What was the severity of this symptom at its WORST? | |

| | O None O Mild O Moderate O Severe O Very Severe |
|---------------|-------------------------------------------------|
| Today's Date: | MR#/Name: |